## CLINICAL RESEARCH IN INFECTIOUS DISEASES

# STATISTICAL ANALYSIS PLAN for

DMID Protocol: 18-0018 Study Title:

A Phase 1, Open-Label, Dose-Escalation Trial to Evaluate the Safety, Reactogenicity, and Immunogenicity of the Sm-p80 + GLA-SE (SchistoShield®) Vaccine in Healthy Adults

NCT05292391

Version 4.0

**DATE: 01 FEB 2024** 

RESTRICTED

## **STUDY TITLE:**

# A Phase 1, Open-Label, Dose-Escalation Trial to Evaluate the Safety, Reactogenicity, and Immunogenicity of the Sm-p80 + GLA-SE (SchistoShield®) Vaccine in Healthy Adults

| <b>Protocol Number Code:</b> | DMID Protocol: 18-0018 |
|---|---|
| <b>Development Phase:</b> | Phase 1 |
| Products: | Sm-p80 + GLA-SE (SchistoShield®) Vaccine |
| Form/Route: | Intramuscular injections |
| Indication Studied: | Intestinal schistosomiasis |
| Sponsor: | Division of Microbiology and Infectious Diseases |
| | National Institute of Allergy and Infectious Diseases |
| | National Institutes of Health |
| Clinical Trial Initiation Date: | 28 February 2022 |
| Clinical Trial Completion Date: | Ongoing |
| Date of the Analysis Plan: | 01 FEB 2024 |
| Version Number: | Version 4.0 |

This study was performed in compliance with Good Clinical Practice.

Information contained in this publication is the property of Division of Microbiology and Infectious Diseases and is confidential. This information may not be disclosed to third parties without written authorization from Division of Microbiology and Infectious Diseases. This report may not be reproduced, stored in a retrieval system or transmitted in any form or by any means - electronic, mechanical, recording or otherwise - without the prior authorization from Division of Microbiology and Infectious Diseases. This document must be returned to Division of Microbiology and Infectious Diseases upon request.

# TABLE OF CONTENTS

| STUDY | TITLE: | 2 |
|---|---|---|
| TABLE | OF CONTENTS | 3 |
| LIST OF | F ABBREVIATIONS | 7 |
| 1. | PREFACE | 9 |
| 2. | INTRODUCTION | 10 |
| 2.1. | Purpose of the Analyses | 10 |
| 3. | STUDY OBJECTIVES AND ENDPOINTS | 12 |
| 3.1. | Study Objectives | 12 |
| 3.1.1. | Primary | 12 |
| 3.1.2. | Secondary | 12 |
| 3.1.3. | Exploratory | 12 |
| 3.2. | Study Endpoints or Outcome Measures | 12 |
| 3.2.1. | Primary | 12 |
| 3.2.2. | Secondary | 12 |
| 3.2.3. | Exploratory | 13 |
| 3.3. | Study Definitions and Derived Variables | 13 |
| 4. | INVESTIGATIONAL PLAN | 14 |
| 4.1. | Overall Study Design and Plan | 14 |
| 4.2. | Discussion of Study Design, Including the Choice of Control Groups | 14 |
| 4.3. | Selection of Study Population | 14 |
| 4.4. | Treatments | 18 |
| 4.4.1. | Treatments Administered | 18 |
| 4.4.2. | Identity of Investigational Product(s) | 18 |
| 4.4.3. | Method of Assigning Subjects to Treatment Groups (Randomization) | 18 |
| 4.4.4. | Selection of Doses in the Study | 18 |
| 4.4.5. | Selection and Timing of Dose for Each Subject | 19 |
| 4.4.6. | Blinding | 19 |
| 4.4.7. | Prior and Concomitant Therapy | 19 |
| 4.4.8. | Treatment Compliance. | 19 |
| 4.5. | Efficacy (Immunogenicity) and Safety Variables | 19 |
| 4.5.1. | Safety Variables | 20 |

#### **Table of Contents** (continued) 4.5.2. 5. SAMPLE SIZE CONSIDERATIONS ......21 6. 6.1. 6.2. Timing of Analyses 22 6.3. Analysis Populations .......24 6.3.1. 6.3.2. 6.3.3. 6.4. 6.5. Missing Data......25 6.6. 6.6.1. 6.6.2. 6.7. Multicenter Studies 26 6.8. Multiple Comparisons/Multiplicity .......26 7. 7.1. 7.2. 8. 9. 9.1. Prior and Concurrent Medical Conditions 29 9.1.1. 9.1.2. 9.2. 9.3. 9.3.1. 9.3.2. 9.4. Deaths, Serious Adverse Events and other Significant Adverse Events ......31 9.5. 9.6.

| Table of Contents (continued) | | |
|---|---|---|
| 9.7. | Vital Signs and Physical Evaluations | 31 |
| 9.8. | Concomitant Medications | 32 |
| 9.9. | Other Safety Measures | 32 |
| 10. | PHARMACOKINETICS | 33 |
| 11. | IMMUNOGENICITY | 34 |
| 11.1. | Secondary Immunogenicity Analysis | 34 |
| 11.1.1. | ELISA (anti Sm-p80 Total IgG) | 34 |
| 12. | OTHER ANALYSES | 35 |
| 13. | REPORTING CONVENTIONS | 36 |
| 14. | TECHNICAL DETAILS | 37 |
| 15. | SUMMARY OF CHANGES IN THE CONDUCT OF THE STUDY OR PLANNED ANALYSES | 38 |
| 16. | REFERENCES | 39 |
| APPENI | DICES | 41 |
| APPENI | DIX 1. TABLE MOCK-UPS | 42 |
| 9.1 | Overall Study Design and Plan Description | 48 |
| 10.2 | Protocol Deviations | 55 |
| 14.1 | Description of Study Subjects | 61 |
| 14.2 | Immunogenicity Data | 68 |
| 14.3 | Safety Data | 80 |
| 14.3.2 | Listing of Deaths, Other Serious and Significant Adverse Events | 101 |
| 14.3.3 | Narratives of Deaths, Other Serious and Significant Adverse Events | 104 |
| 14.3.4 | Abnormal Laboratory Value Listings (by Subject) | 105 |
| 14.3.5 | Displays of Laboratory Results | 107 |
| 14.3.6 | Displays of Vital Signs | 126 |
| 14.4 | Summary of Concomitant Medications | 130 |
| APPENI | DIX 2. FIGURE MOCK-UPS | 131 |
| 10.1 | Disposition of Subjects | 134 |
| 14.2 Eff | cacy/Immunogenicity Data | 135 |
| 14.2.2 | Efficacy/Immunogenicity Response Figures by Measure, Treatment/Vaccination, and Time Point | 135 |
| 14.3 Saf | ety Data | 140 |

| Table of Contents (continued) | | | |
|-------------------------------|--------|----------------------------|-----|
| 14.3.1 Adve | erse I | Events | 140 |
| 14.3.5 | Disp | lays of Laboratory Results | 147 |
| APPENDIX | 3. | LISTINGS MOCK-UPS | 149 |
| APPENDIX | ζ 4. | NCA TEMPLATE | 170 |

# LIST OF ABBREVIATIONS

| ADCC | Antibody-Dependent Cellular Cytotoxicity |
|--------|--------------------------------------------------------------|
| AE | Adverse Event |
| ALT | Alanine Aminotransferase |
| ATC | Anatomical Therapeutic Classification |
| BP | Blood Pressure |
| BMI | Body Mass Index |
| CI | Confidence Interval |
| CRF | Case Report Form |
| CSR | Clinical Study Report |
| DMID | Division of Microbiology and Infectious Diseases, NIAID, NIH |
| eCRF | Electronic Case Report Form |
| ELISA | Enzyme-linked Immunosorbent Assay |
| FDA | Food and Drug Administration |
| GLA-SE | Glucopyranosyl Lipid Adjuvant Stable oil-in-water Emulsion |
| GMFR | Geometric Mean Fold Rise |
| GMT | Geometric Mean Titers |
| HCV | Hepatitis C Virus |
| ICH | International Conference on Harmonisation |
| ICS | Intracellular Cytokine Staining |
| IM | Intramuscular |
| LLOQ | Lower Limit of Quantification |
| MAAE | Medically Attended Adverse Events |
| MedDRA | Medical Dictionary for Regulatory Activities |
| mITT | Modified Intention to Treat |
| MOP | Manual of Procedures |
| N | Number (refers to number of subjects) |
| NIH | National Institutes of Health |
| NOCMC | New Onset Chronic Medical Condition |
| PBMC | Peripheral Blood Mononuclear Cell |
| PI | Principal Investigator |
| PIMMC | Potentially Immune-Mediated Medical Condition |
| PP | Per Protocol |

# **List of Abbreviations** (continued)

| PT | Preferred Term |
|--------|----------------------------------------------------------------|
| RCD | Reverse Cumulative Distribution |
| SAE | Serious Adverse Event |
| SAP | Statistical Analysis Plan |
| SD | Standard Deviation |
| SDCC | Statistical and Data Coordinating Center |
| SMC | Safety Monitoring Committee |
| Sm-p80 | S. mansoni Caplain Protein with a mass of approximately 80 kDa |
| SOC | System Organ Class |
| ULN | Upper Limit of Normal |
| ULOQ | Upper Limit of Quantification |
| WBC | White Blood Cell |
| WFI | Water-For-Injection |
| WHO | World Health Organization |

#### 1. PREFACE

The Statistical Analysis Plan (SAP) for "A Phase 1, Open-Label, Dose-Escalation Trial to Evaluate the Safety, Reactogenicity, and Immunogenicity of Sm-p80 + GLA-SE (SchistoShield®) Vaccine in Healthy Adults" (DMID Protocol 18-0018) describes and expands upon the statistical information presented in the protocol.

This document describes all planned analyses and provides reasons and justifications for these analyses. It also includes sample tables, listings, and figures planned for the final analyses. Regarding the final analyses and Clinical Study Report (CSR), this SAP follows the International Conference on Harmonization of Technical Requirements for Registration of Pharmaceuticals for Human Use (ICH) Guidelines, as indicated in Topic E3 (Structure and Content of Clinical Study Reports), and more generally is consistent with Topic E8 (General Considerations for Clinical Trials) and Topic E9 (Statistical Principles for Clinical Trials). The structure and content of the SAP provides sufficient detail to meet the requirements identified by the FDA and ICH, while all work planned and reported for this SAP will follow internationally accepted guidelines published by the American Statistical Association and the Royal Statistical Society for statistical practice.

This document contains four sections: (1) a review of the study design, (2) general statistical considerations, (3) comprehensive statistical analysis methods for efficacy and safety outcomes, and (4) a list of proposed tables and figures. Within the table, figure, and listing mock-ups (Appendix 1, Appendix 2, and Appendix 3, respectively), references to CSR sections are included. Any deviation from this SAP will be described and justified in protocol amendments and/or in the CSR, as appropriate. The reader of this SAP is encouraged to also review the study protocol for details on conduct of the study and the operational aspects of clinical assessments.

## 2. INTRODUCTION

In preclinical and safety studies, Sm-p80-based vaccines provided comprehensive coverage against different stages of the parasite's life cycle, including its eggs, schistosomula, and adult worms. Sm-p80 is unique in that it has demonstrated desirable outcomes of Sm-p80 vaccination including: 1) prophylactic efficacy against *S. mansoni* (intestinal/hepatic schistosomiasis); [9] 2) reduction in egg-induced tissue/organ pathology; [9] 3) ost-exposure therapeutic efficacy by elimination of established adult worms in chronic disease[11] 4) cross species-protection against *S. haematobium* (urinary schistosomiasis) [12] and *S. japonicum* (Asiatic/oriental disease); [13] 5) long lived immunity as Sm-p80 specific IgG titers are present in mice for up to 60 weeks and 5-8 years in baboons; [14] and 6) maternal transfer of Sm-p80-specific antibodies in baboons. [14] Sm-p80-specific IgE has not been detected in high-risk or infected populations from Africa and South America, thus reducing the possibility of hypersensitivity following vaccination with the Sm-p80 vaccine in humans. The protective immune response to *Schistosoma* is thought to be antibody mediated with cell-mediated help to skew the antibody isotypes to IgG1 and IgG3.

The 5 µg dose of GLA-Se to be used in this trial is comfortably in the mid-range of tested doses of the adjuvant and has been shown to be safe and well tolerated in hundreds of human subjects. As reported in the GLA-SE Investigator Brochure (v5, March 2016) many preclinical and nonclinical studies in mice, guinea pigs, rats, rabbits, and non-human primates have demonstrated the immunostimulatory properties of GLA-SE with no significant safety signals. GLA-SE has also been evaluated in numerous completed and ongoing clinical trials. These trials have investigated GLA-SE formulated with antigens, including recombinant antigens, developed for vaccines against a wide variety of diseases, including leishmaniasis, [15] tuberculosis, [16, 17] influenza, [18, 19] schistosomiasis, [20] and malaria. These clinical trials have evaluated GLA-SE at 0.5, 1, 2, 2.5, 5, 10, or 20 µg dose levels. In these studies, over 1100 subjects have received at least one study injection containing GLA-SE. Safety data have not revealed any significant safety issues at any dose level tested. Reactions to vaccines varied from study to study, but were generally mild, resolved quickly, and typical of vaccinations by the IM route.

In the GLP-toxicity study of SchistoShield®, there were no findings definitively attributed to systemic toxicity of Sm-p80 with or without GLA-SE. This study indicated that the SchistoShield® vaccine is safe and well tolerated in rabbits when administered IM for up to four injections at the highest proposed human dose of Sm-p80 antigen given with GLA-SE. No significant local or systemic toxicity was found. A general safety assessment of SchistoShield® vaccine in baboons also indicated that the vaccine is safe and well tolerated for up to the highest dose of 250  $\mu$ g of Sm-p80 and 50  $\mu$ g of GLA-SE, further supporting the observation from the GLP-toxicity study in rabbits. Based on the N+1 rule, the GLP-toxicity study in rabbits supports the use of SchistoShield® vaccine in the first-in-human clinical trial for up to three injections at the high dose of 100  $\mu$ g Sm-p80.

The promising results of the preclinical evaluations and the urgent need for an effective schistosomiasis vaccine support advancement of the SchistoShield® vaccine candidate to an initial Phase 1 human trial in healthy volunteers in the United States.

# 2.1. Purpose of the Analyses

The purpose of this trial is to determine the safety, reactogenicity, and immunogenicity in 45 healthy adult subjects of the candidate investigational schistosomiasis vaccine: Sm-p80 (10 µg, 30 µg, and 100 µg) adjuvanted with 5 µg of GLA-SE adjuvant. The analyses will also assess the necessity of the adjuvant by comparison of the previous doses to 100 µg Sm-p80 only (Table 1). Subjects will receive three IM injections

of 0.5 mL of the designated study product formulation, on Days 1, 29, and 57 (28 days apart) or on a delayed booster dose schedule on Days 1, 29, and 180.

The protocol for DMID 18-0018 calls for a planned interim analysis on safety data and immunogenicity assays, including total IgG Enzyme-linked Immunosorbent Assay (ELISA), at the discretion of the study team prior to completion of follow-up of all subjects.

## 3. STUDY OBJECTIVES AND ENDPOINTS

# 3.1. Study Objectives

## **3.1.1. Primary**

- To assess the safety and reactogenicity following receipt of three doses of the following
  - Group A: 100 μg Sm-p80 (unadjuvanted)
  - Group B: 10 μg Sm-p80 + 5 μg GLA-SE
  - Group C: 30 μg Sm-p80 + 5 μg GLA-SE (delayed booster)
  - Group D: 30 μg Sm-p80 + 5 μg GLA-SE
  - Group E: 100 μg Sm-p80 + 5 μg GLA-SE

with Groups A, B, D, and E administered intramuscularly on Days 1, 29, and 57 and Group C administered on Days 1, 29, and 180.

#### 3.1.2. Secondary

• To assess anti-Sm-p80 IgG antibody responses from samples collected at specified time points.

## 3.1.3. Exploratory

• To assess innate and adaptive immune signatures from samples collected at specified time points.

## 3.2. Study Endpoints or Outcome Measures

#### **3.2.1. Primary**

- Occurrence of study vaccine-related SAEs from the time of the first study vaccination through approximately 12 months after the last study vaccination
- Occurrence of solicited injection site and systemic reactogenicity events from the time of each study vaccination through 7 days after each study vaccination
- Occurrence of clinical safety laboratory AEs form the time of each study vaccination through approximately 28 days after each study vaccination
- Occurrence of all unsolicited AEs, regardless of the assessment of seriousness or relatedness, from the time of each study vaccination through 28 days after each study vaccination
- Occurrence of SAEs, MAAEs, NOCMCs, and PIMMCs from the time of the first study vaccination through approximately 12 months after the last study vaccination

## 3.2.2. Secondary

- For Sm-p80 IgG antibodies, number of subjects achieving seroconversion, defined as fourfold rise from baseline, at approximately 28 days after the first, second, and third study vaccinations
- Geometric mean titers of serum Sm-p80 IgG antibodies from samples collected at 7 and 28 days after each vaccination, and at 124 days after the last vaccination

#### 3.2.3. Exploratory

- Identification and characterization of gene expression changes as measured using RNA-seq analysis from whole blood relative to last vaccination
  - o Days 8 and 29 vs. Day 1, and Day 36 vs. Day 29 for all study groups
  - o Day 57 vs. Day 29, Day 64 vs. Day 57 for Groups A, B, D, and E
  - o Day 187 vs. Day 180 for Group C
- Identification and characterization of gene expression changes as measured using RNA-seq relative to last vaccination that correlate with peak Sm-p80 IgG antibody levels
  - o Days 8 and 29 vs. Day 1, and Day 36 vs. Day 29 for all study groups
  - o Day 57 vs. Day 29, Day 64 vs. Day 57 for Groups A, B, D, and E
  - o Day 187 vs. Day 180 for Group C

## 3.3. Study Definitions and Derived Variables

Seroconversion is defined as a fourfold rise from baseline.

Clinical laboratory evaluations, vital signs, reactogenicity, and immunogenicity will be assessed on the day of, prior to the first study product injection (Day 1) to establish baseline. If a single ELISA result is below the lower limit of quantification (LLOQ) or above the upper limit of quantification (ULOQ) then the result will be imputed as LLOQ or ULOQ, respectively. If both ELISA results are below LLOQ, then the value will be imputed as ½\*LLOQ. If both ELISA results are above ULOQ, then ULOQ will be reported.

Any medical condition that is present at the time that the subject is screened will be considered baseline and not reported as an AE. However, if the existing severity of any pre-existing medical condition increases, it will be recorded as an AE.

#### 4. INVESTIGATIONAL PLAN

## 4.1. Overall Study Design and Plan

This is a Phase 1, open label, dose-escalation clinical trial to evaluate the safety, reactogenicity, and immunogenicity of Sm-p80 + GLA-SE candidate schistosomiasis vaccine (SchistoShield®) in healthy adults 18 through 55 years of age. The Sm-p80 antigen is a recombinant protein produced in *E. coli* and GLA-SE is an immunological adjuvant.

Five treatment groups, each including nine subjects, will receive three intramuscular (IM) injections of 0.5 mL of designated study product on either Days 1, 29, and 57 or on Days 1, 29, and 180. Group A (unadjuvanted comparator) will receive 100  $\mu$ g Sm-p80 alone on Days 1, 29, and 57; Group B (low dose standard schedule) will receive 10  $\mu$ g Sm-p80 + 5  $\mu$ g GLA-SE on Days 1, 29, and 57; Group C (mid dose delayed booster) will receive 30  $\mu$ g Sm-p80 + 5  $\mu$ g GLA-SE on Days 1, 29, and 180; Group D (mid dose standard schedule) will receive 30  $\mu$ g Sm-p80 + 5  $\mu$ g GLA-SE on Days 1, 29, and 57; Group E (high dose standard schedule) will receive 100  $\mu$ g Sm-p80 + 5  $\mu$ g GLA-SE on Days 1, 29, and 57. Dose escalation will proceed as described in the Protocol Summary (protocol v2.0).

Reactogenicity will be measured by the occurrence of solicited injection site and systemic reactions form the time of each study product injection through seven days after each study product injection. Unsolicited AEs of all severities, and concomitant medications, will be collected form the time of each study product injection through the next 28 days. During period of follow-up outside of the 28-day post-vaccination interval, only SAEs, medically attended adverse events (MAAEs), new onset chronic medical conditions (NOCMCs), and potentially immune-mediated medical conditions (PIMMCs) will be collected. Clinical laboratory evaluations for safety will be performed on venous blood collected prior to, and approximately seven days after, each study vaccination.

Immunogenicity testing will include measuring titers of total IgG against the Sm-p80 protein by ELISA. Gene expression will be evaluated using RNA Seq analysis from whole blood.

# 4.2. Discussion of Study Design, Including the Choice of Control Groups

# **4.3.** Selection of Study Population

The study population of 45 subjects will be enrolled from a population of healthy, *Schistosoma*-naïve subjects ages 18 through 55 years at a single study site in Seattle, Washington.

Subject Inclusion and Exclusion Criteria must be assessed by a study clinician licensed to make medical diagnoses and listed on the Form FDA 1572 as the site PI or sub-investigator. No exemptions are granted on Subject Inclusion/Exclusion Criteria in DMID-sponsored studies. Questions about eligibility will be directed toward the DMID Medical Officer.

## **Subject Inclusion Criteria**

Subjects must meet all the following inclusion criteria to be eligible for enrollment in this study

- 1. Male or non-pregnant female 18 through 55 years of age, inclusive, at the time of consent
- 2. Able and willing to participate for the duration of the study and able to understand and comply with planned study procedures
- 3. Able and willing to provide written (not proxy) informed consent

4. Is in good health, as judged by the investigator, and determined by medical history and physical examination\*

\*Existing medical diagnoses or conditions (except those in the Subject Exclusion Criteria) must be deemed as stable. A stable medical condition is defined as no change in prescription medication, dose, or frequency of medication in the last three months (90 days) and health outcomes of the specific disease are considered to be within acceptable limits in the last size months (180 days). Any change due to change of health care provider, insurance company, or that is done for financial reasons, as long as in the same class of medication, will nor be considered a violation of this inclusion criterion. Any change in prescription medication due to **improvement** of a disease outcome, as determined by the site PI or appropriate subinvestigator, will not be considered a violation of this inclusion criterion. Subjects may be on chronic or as needed (prn) medications if, in the opinion of the site PI or appropriate subinvestigator, they pose no additional risk to the subject safety or assessment of solicited events and immunogenicity.

Topical, nasal, and inhaled medications (with the exception of some uses of corticosteroids as outlined in the Subject Exclusion Criteria), vitamins, and contraceptives are permitted.

- 5. Women of childbearing potential\* must have a negative serum pregnancy test at screening and a negative urine pregnancy test within 24 hours prior to each study product injection
  - \*Not sterilized via bilateral tubal ligation, bilateral oophorectomy, or hysterectomy, or, if menopausal, still menstruating or < 1 year of the last menses.
- 6. Women of childbearing potential must have used an acceptable form of contraception\* in the 30 days prior to their first study product injection
  - \*Acceptable single forms of contraception include abstinence from sexual activity that could lead to pregnancy, monogamous relationship with vasectomized partner who has been vasectomized for six months or more prior to enrollment, successful Essure® placement (permanent, non-surgical, non-hormonal sterilization), intrauterine devices, and hormonal methods, including the birth control patch, shot (Depo-Provera), pills, the vaginal ring (NuvaRing), and the contraceptive implant (Nexplanon). Acceptable barrier methods include diaphragm or cervical cap with spermicide and the contraceptive sponge.
- 7. Women of childbearing potential must agree to continue use of an acceptable form of contraception through 30 days after their last study product injection
- 8. Weight  $\geq$  50 kg and body mass index (BMI)  $\leq$  35.0 kg/m<sup>2</sup>
- 9. Vital signs (oral temperature, pulse, and blood pressure) are within normal protocol-defined ranges\*
  - \*The normal protocol-defined ranges for vital signs include (a) oral temperature less than 38°C (100.4°F), (b) pulse no greater than 100 bpm, (c) systolic blood pressure 85 to 150 mmHg, inclusive, and (d) diastolic BP  $\leq$  100 mmHg.
- 10. Screening clinical lab values are all within normal protocol-defined reference ranges\*
  - \*The normal protocol-defined ranges for laboratory tests include (a) ALT of < 47 IU/L, (b) creatinine less than or equal to the laboratory upper limit of normal, (c) WBC  $\ge$  3.80x10<sup>3</sup>/UL and  $\le$  13.00x10<sup>3</sup>/UL, (d) hemoglobin 11.5 g/dL or greater for females or 12.6 g/dL or greater for males, (e) platelets between 131x10<sup>3</sup>/UL and 415x10<sup>3</sup>/UL, inclusive.

#### **Subject Exclusion Criteria**

Subjects must not meet any of the exclusion criteria at baseline to be eligible for enrollment in this study.

- 1. Has had known schistosomiasis infection or has traveled to an endemic area for schistosomiasis infection and, during that travel, was potentially exposed to a Schistosoma species
- 2. Has been treated for schistosomiasis
- 3. Has previous exposure to schistosome vaccines or experimental products containing GLA-SE
- 4. Female subjects who are breastfeeding a child, or who plan to breastfeed a child from the first study product injection through 30 days after the last study product injection
- 5. Asthma, other than mild, well-controlled asthma\*
  - \*Cold or exercise-induced asthma controlled with inhaled medications other than inhaled corticosteroids is permissible. Subjects should be excluded if they require daily bronchodilator use or have had an asthma exacerbation requiring oral/parental steroid use or have used theophylline or inhaled corticosteroids in the past year.
- 6. Known atherosclerotic cardiovascular disease or history of myocardial infarction, pericarditis, or myocarditis
- 7. Diabetes mellitus
- 8. History of psychiatric condition that may make study compliance difficult, such as schizophrenia, or poorly controlled bipolar disorder\*
  - \*Includes persons with psychoses or history of suicide attempt or gesture in the 3 years before study entry or an ongoing risk for suicide.
- 9. Chronic or active neurologic condition (including seizures\* and migraine headaches\*\*)
  - \*Seizure within the past 5 years.
  - \*\*Four or more migraine headaches in the past 12 months that interfered with normal daily activity or any migraine headache in the past 5 years that required emergency or inpatient medical care.
- 10. Autoimmune disease\*
  - \*Autoimmune hypothyroidism with or without replacement therapy, and vitiligo or mild eczema or psoriasis not requiring chronic therapy, are permissible
- 11. Known or suspected congenital or acquired immunodeficiency including anatomic or functional asplenia\* or immunosuppression as a result of underlying illness or treatment
  - \*Any splenectomy is exclusionary
- 12. Use of alcohol or drugs that, in the opinion of the investigator, may interfere with ability to comply with the protocol or increase risk to subject's health during the study period
  - \*Subjects with a history of malignancy may be included if treated by surgical excision, or by chemotherapy or radiation therapy and has been observed for a period that in the investigator's estimation provides a reasonable assurance of sustained cure (not less than 36 months). Cervical neoplasia under surveillance and non-melanoma skin cancer are not exclusionary.
- 13. Active neoplastic disease\*

\*Subjects with a history of malignancy may be included if treated by surgical excision, or by chemotherapy or radiation therapy and has been observed for a period that in the investigator's estimation provides a reasonable assurance of sustained cure (not less than 36 months). Cervical neoplasia under surveillance and non-melanoma skin cancer are not exclusionary.

14. Chronic topical or systemic corticosteroid use\*

\*Corticosteroid nasal sprays for allergic rhinitis are permissible. Persons using a topical corticosteroid for a limited duration for mild uncomplicated dermatitis such as poison ivy or contact dermatitis prior to enrollment may be enrolled the day after their therapy is completed. Oral or parenteral (intravenous, IM, subcutaneous) corticosteroids given for non-chronic conditions not expected to recur are permissible if, within the year prior to enrollment, the longest course of therapy was no more than 14 days and no oral or parenteral corticosteroids were given within 30 days prior to enrollment. Intraarticular, bursal, tendon, or epidural injections of corticosteroids are permissible if the most recent injection was at least 30 days prior to enrollment. Topical or systemic corticosteroid use for study related AEs is not exclusionary.

- 15. Known contraindication to repeated phlebotomy\*
  - \*Such as minimal venous access or recent history of anemia
- 16. Receipt or planned receipt of inactivated vaccine or allergy desensitization injection within 14 days before or after a study product injection
- 17. Receipt or planned receipt of live attenuated vaccine 28 days before or after a study product injection
- 18. Receipt of blood products or immunoglobulin within six months prior to, or donation of unit of blood within two months prior to, the first study product injection.
- 19. Receipt of any experimental agent\* within 30 days prior to screening or planned receipt prior to the last study visit\*\*
  - \*Vaccine, drug, biologic, device, blood product, or medication.
  - \*\*Receipt of experimental COVID-19 related products are not necessarily exclusionary and will be evaluated on a case-by-case basis.
- 20. Plan to undergo surgery (elective or otherwise) within six months after study enrollment
- 21. Plans to enroll in another interventional clinical trial\* at any time during the study period
  - \*Includes trials evaluating interventions such as a drug, biologic, or device.
- 22. Positive confirmatory test for HIV infection
- 23. Positive serologic test for hepatitis B surface antigen (HBsAg)
- 24. Positive confirmatory test for hepatitis C virus (HCV) infection
- 25. Acute febrile illness (oral temperature ≥ 38°C) or other acute illness within three days prior to study product injection\*

\*Note for afebrile, acute illness only: If a subject is afebrile, his/her acute illness is nearly resolved with only minor residual symptoms remaining, and, in the opinion of the site PI or appropriate sub-investigator, the residual symptoms will not interfere with the ability ro assess

safety parameters as required by the protocol, the subject may receive study product injection without further approval form the DMID Medical Officer.

- 26. Not willing to avoid donating blood during the study
- 27. Has any condition that would, in the opinion of the site investigator, place the subject at an unacceptable risk of injury or render the subject unable to meet the requirements of the protocol

#### 4.4. Treatments

#### 4.4.1. Treatments Administered

Each dose of study vaccine will be administered as a single 0.5-mL IM injection in the deltoid muscle of the participant's arm. Participants will be observed in the clinic for a minimum of 30 minutes following the study product injection. After 30 minutes, the injections site will be examined and the participant will be questioned about the presence of any localized or generalized reactogenicity symptoms. Any spontaneous AEs that occur will be assessed.

See the protocol-specific MOP for detailed information on the administration of the study product for each group. Treatment for each study group is summarized in Table 1.

#### 4.4.2. Identity of Investigational Product(s)

The vaccine product is a two-component system comprised of Sm-p80 antigen and GLA-SE adjuvant.

## Sm-p80 for injection

Sm-p80 is a recombinant protein produced in *E. coli* bacteria. The protein antigen is the largesubunit of the *S. mansoni* calcium-activated neutral protease, calpain. The Sm-p80 protein is formulated and lyophilized to yield the vaccine antigen, Sm-p80 for Injection. The final 758 amino acid protein antigen has a predicted mass of approximately 87kDa.

#### **GLA-SE Adjuvant**

GLA-SE is a synthetic Monophosphoryl Lipid A-like molecule which is a Toll-like receptor 4 agonist formulated in a SE to produce GLA-SE.

#### Sm-p80 + GLA-SE

Sm-p80 + GLA-SE contains the antigen and adjuvant. After reconstitution of the antigen with water-for-injection (WFI) and mixing with the liquid adjuvant, it is ready for administration to the study participant.

#### 4.4.3. Method of Assigning Subjects to Treatment Groups (Randomization)

This is a non-randomized trial. Approximately 9 subjects will be assigned to each treatment arm.

## 4.4.4. Selection of Doses in the Study

Subjects receive 100 µg Sm-p80 alone or 10 µg, 30 µg, or 100 µg Sm-p80 with 5 µg GLA-SE.

The adjuvant dose of 5 µg of GLA-SE is selected for this trial as this dose is in the mid-range of doses evaluated in the 1100 previous subjects, has been shown to increase antibody levels and cellular immune responses, and has been evaluated in multiple clinical trials, including administering three vaccinations, demonstrating an acceptable safety profile. The preclinical studies of SchistoShield® do not inform the

selection of antigen dose for this study, as non-human primates require much higher doses of antigen and adjuvant than humans due to the tolerizing effects of their environment. In other vaccine trials in humans, GLA-SE adjuvant administered with antigen doses suggest that lower antigen doses are best to elicit T cell responses while the higher doses tend to elicit better humoral responses. Since it appears that the primary mechanism of action of SchistoShield® is mediated by humoral responses, this study will evaluate a range of Sm-p80 doses from 10 to 100  $\mu$ g.

## 4.4.5. Selection and Timing of Dose for Each Subject

Subjects were evenly distributed between treatment arms. Each subject receives three doses of the study product on Days 1, 29, and 57 or Days 1, 29, and 180. Each dose of study vaccine will be administered as a single 0.5-mL IM injection in the deltoid muscle of the participant's arm. Detailed descriptions of study agent preparation and administration are found in the study MOP.

## 4.4.6. Blinding

This is an open-label clinical trial.

Subjects, investigators, study personnel performing any study-related assessments following study vaccine administration are not blinded to study treatment. Laboratory personnel performing immunologic assays will receive samples blinded to subject ID number and sample visit number.

#### 4.4.7. Prior and Concomitant Therapy

Administration of any medications, therapies, or vaccines will be recorded on the appropriate eCRF. Concomitant medications will include all current medications and medications taken in the 60 days prior to the first vaccination and those taken from the time of vaccination through approximately 28 days after each vaccination, as described in Section 3.1. Medications reported in the electronic case report form (eCRF) are limited to those taken within 30 days prior to the first study product injection and those taken in the 28-day post-vaccination interval. Prescriptionand over-the-counter drugs will be included as well as herbals, vitamins, and supplements. In addition, receipt of non-study vaccines will be solicited from the time of each vaccination through approximately 28 days after each vaccination and reported in the eCRF. Use of a new medication should prompt evaluation for the occurrence of any MAAE, including a NOCMC.

Medications that might interfere with the evaluation of the investigational product(s) should not be used during the trial-reporting period (approximately 12 months after the last study vaccination) unless clinically indicated as part of the subject's health care. Medications in this category include the prohibited medications per the Subject Exclusion Criteria (see Section 4.3). In addition, the site PI or appropriate sub-investigator may identify other medications that should not be used due to a risk to subject safety or assessment of reactogenicity and immunogenicity.

#### 4.4.8. Treatment Compliance

All subjects receive a total of three doses of study product delivered intramuscularly in the clinic by a qualified study personnel member according to subject treatment assignment.

# 4.5. Efficacy (Immunogenicity) and Safety Variables

As this is a Phase 1 clinical trial in healthy adult subjects, there is no assessment of drug efficacy. For a detailed schedule of activities, refer to Table 2 and Table 3. Refer to Section 3 for a list of primary and secondary objectives.

In general, multiple observations within a specific visit period will be accepted. In case of multiple observations within a specific window, the assessment value that is closest to the scheduled visit window will be used in the analyses for the post-baseline records. If observations have the same distance to the scheduled assessment, the latest one will be used. All recorded data will be listed.

#### 4.5.1. Safety Variables

Serious adverse events (SAEs) will be assessed from the time of the first study product injection through the end of the follow-up which is approximately 12 months after the last study product injection.

Solicited adverse events (AEs) will document reactogenicity events occurring from the time of each study product injection through 7 days after each study product injection. Injection site reactions of interest include pruritus, erythema, induration/swelling, pain, and tenderness. Systemic reactions of interest include fever, chills, fatigue malaise, myalgia, arthralgia, headache, nausea, and vomiting.

Unsolicited AEs will document non-serious AEs occurring from the time of each study product injection through 28 days after the study product injection.

Clinical safety laboratory AEs will be collected on the day of and prior to each study product injection, approximately 7 days after each study product injection, and approximately 28 days after each study product injection (which may also serve as the clinical safety laboratory samples for the second and/or third study product injection). Parameters to be evaluated include white blood cells (WBC), hemoglobin, platelets, alanine aminotransferase (ALT), and creatinine.

MAAEs, NOCMCs, and PIMMCs will be assessed from the time of the first study product injection through the end of the follow-up period, which is approximately 12 months after the last study product injection.

All solicited and unsolicited AEs and laboratory values are graded on a scale of 0 (absent), 1 (mild), 2 (moderate), and 3 (severe) according to toxicity grading scales (Table 6, Table 7).

#### 4.5.2. Immunogenicity Variables

Assessment of antibody responses are measured by total IgG production to Sm-p80 protein using ELISA. RNA-Seq data will be pre-processed by removing adaptors and low-quality reads, trimming low quality ends, and mapping sequences to the latest human reference genome using splice-aware alignment software such as *HISAT2* for transcriptomic exploratory analysis.

Samples for immunogenicity assays are collected prior to each vaccination on the day of vaccination, at 7 and 28 days after each vaccination, and at 124 days after the last vaccination. The 28-day post-vaccination sample will also serve as the day of vaccination sample for a subsequent vaccination given at a 28-day interval.

Additional details on RNA-Seq analysis will be described in a separate SAP, and the analyses will be presented in a CSR Addendum.

## 5. SAMPLE SIZE CONSIDERATIONS

This Phase 1 study is not designed for confirmatory testing but rather to detect AEs related to the study product. If an AE has a 20% chance of occurring after receiving one of the product formulations being tested, then there is an 87% probability that the event would be observed in one or more of the 9 subjects in that treatment group in this study. If the event has a 20% chance or higher of occurring in any of the product formulations being tested, then there is at > 99% probability that the event would be observed in one or more of the 45 subjects in any treatment group in the study. The Table 4 shows analogous probabilities for events with other frequencies.

#### 6. GENERAL STATISTICAL CONSIDERATIONS

## **6.1.** General Principles

All continuous variables will be summarized using the following descriptive statistics: n (non-missing sample size), mean, standard deviation, median, maximum, and minimum. The frequency and percentages (based on the non-missing sample size) of observed levels will be reported for all categorical measures. In general, all data will be listed, sorted by treatment and subject, and when appropriate by visit number within subject. All summary tables will be structured with a column for each treatment in the order (Group A, Group B, Group C, Group D, Group E) and will be annotated with the total population size relevant to that table/treatment, including any missing observations. If the table including all treatment groups in one table results in the table being too wide, separate tables will be made for each treatment group.

## **6.2.** Timing of Analyses

Two interim analyses of safety and immunogenicity data will be conducted prior to completion of follow-up of all subjects: 1.) after the Day 85 visit for Groups A and B and 2.) after the Day 208 visit for Group C or the Day 85 visit for Group D, whichever occurs last. The data will be cleaned but not locked. The following TFLs will be included in these interim analyses:

#### Tables:

- Table 8: Subject Disposition by Treatment Group
- Table 9: Analysis Population by Treatment Group
- Table 12: Summary of Categorical Demographic and Baseline Characteristics by Treatment Group, All Enrolled Subjects
- Table 13: Summary of Continuous Demographic and Baseline Characteristics by Treatment Group, All Enrolled Subjects
- All immunogenicity tables listed in Section 11 (Table 15, Table 16, Table 17)
- Table 18: Overall Summary of Adverse Events
- Table 19: Adverse Events Occurring in 5% of Subjects in Any Treatment MedDRA System Organ Class and Preferred Term, and Treatment Group Safety Population
- Table 20: Number and Percentage of Subjects Experiencing Solicited Events with 95% Confidence Intervals by Symptom and Treatment Group Post Dose 1
- Table 21: Number and Percentage of Subjects Experiencing Solicited Events with 95% Confidence Intervals by Symptom and Treatment Group Post Dose 2
- Table 22: Number and Percentage of Subjects Experiencing Solicited Events with 95% Confidence Intervals by Symptom and Treatment Group Post Dose 3
- Table 23: Number and Percentage of Subjects Experiencing Solicited Events with 95% Confidence Intervals by Symptom and Treatment Group Post Any Dose
- Table 48: Unsolicited Adverse Events by MedDRA System Organ Class and Preferred Term, Maximum Severity, Relationship, and Treatment Group
- Table 54: Listing of Serious Adverse Events

- Table 55: Listing of Non-Serious, Unsolicited, Moderate or Severe Adverse Events
- Table 56: Listing of Other Significant Adverse Events
- Table 57: Listing of Abnormal Laboratory Results Chemistry
- Table 58: Listing of Abnormal Laboratory Results Hematology
- Table 59: Laboratory Results by Parameter, Maximum Severity, Time Point, and Treatment Group Any Chemistry Parameter
- Table 60: Laboratory Results by Parameter, Maximum Severity, Time Point, and Treatment Group Creatinine
- Table 61: Laboratory Results by Parameter, Maximum Severity, Time Point, and Treatment Group Alanine Aminotransferase
- Table 67: Laboratory Results by Parameter, Maximum Severity, Time Point, and Treatment Group Any Hematology Parameter
- Table 68: Laboratory Results by Parameter, Maximum Severity, Time Point, and Treatment Group White Blood Cells
- Table 69: Laboratory Results by Parameter, Maximum Severity, Time Point, and Treatment Group Hemoglobin
- Table 70: Laboratory Results by Parameter, Maximum Severity, Time Point, and Treatment Group Platelets

#### Figures:

- All immunogenicity figures listed in Section 11 (Figure 2, Figure 3, Figure 4)
- Figure 8: Number and Percentage of Subjects Experiencing Solicited Systemic Events by Event, Maximum Severity, and Treatment Group Post Dose 1
- Figure 9: Number and Percentage of Subjects Experiencing Solicited Systemic Events by Event, Maximum Severity, and Treatment Group Post Dose 2
- Figure 10: Number and Percentage of Subjects Experiencing Solicited Systemic Events by Event, Maximum Severity, and Treatment Group Post Dose 3
- Figure 11: Number and Percentage of Subjects Experiencing Solicited Systemic Events by Event, Maximum Severity, and Treatment Group Post Any Dose
- Figure 15: Number and Percentage of Subjects Experiencing Solicited Injection Site Events by Event, Maximum Severity, and Treatment Group Post Dose 1
- Figure 16: Number and Percentage of Subjects Experiencing Solicited Injection Site Events by Event, Maximum Severity, and Treatment Group Post Dose 2
- Figure 17: Number and Percentage of Subjects Experiencing Solicited Injection Site Events by Event, Maximum Severity, and Treatment Group Post Dose 3
- Figure 18: Number and Percentage of Subjects Experiencing Solicited Injection Site Events by Event, Maximum Severity, and Treatment Group Post Any Dose
- Figure 19: Frequency of Related Adverse Events by MedDRA System Organ Class and Severity

## Listings:

• Listing 9: Individual Immunogenicity Response Data

The SMC will review safety at least annually. A final SMC review meeting will occur 6 to 8 months after clinical database lock. Additional interim analyses of safety and immunogenicity data may be conducted at the discretion of the SMC prior to completion of follow-up of all subjects. The final analysis will be performed after all outcome data from all subjects through the final study visit have been monitored and locked.

## 6.3. Analysis Populations

Summaries and analysis for safety data will be presented for the Safety Population. Summaries and analysis of immunogenicity data will be presented for the modified intention-to-treat population. If there are major protocol deviations, a per-protocol (PP) analysis may also be performed. Immunogenicity data from any visit that occurs substantially out of window will be reviewed by the Principal Investigator, DMID Scientific Lead, and/or DMID Medical Officer for decisions regarding inclusion or exclusion of the data. A tabular listing of all subjects, visits, and observations excluded from the analysis will be provided in the CSR (Listing 5).

## **6.3.1.** Modified Intention-to-Treat (mITT) Immunogenicity Population

The modified intention-to-treat (mITT) immunogenicity population includes all subjects who received at least one dose of study vaccine and contributed both pre- and at least one post-study vaccination venous blood sample for immunogenicity testing for which valid results were reported. For analyses using the mITT immunogenicity population, subjects will be grouped based on treatment assignments:  $100 \mu g$  Sm-p80 (unadjuvanted),  $10 \mu g$  Sm-p80 +  $5 \mu g$  GLA-SE,  $30 \mu g$  Sm-p80 +  $5 \mu g$  GLA-SE (delayed booster),  $30 \mu g$  Sm-p80 +  $5 \mu g$  GLA-SE,  $100 \mu g$  Sm-p80 +  $5 \mu g$  GLA-SE.

#### **6.3.2.** Per Protocol Population

The per protocol (PP) population includes all subjects in the mITT subset with the following exclusions:

- Data from all available visits for subjects found to be ineligible.
- Data from all visits subsequent to protocol deviations such as:
  - o Second or third study vaccine not received,
  - o Second or third vaccine received out of window,
  - o Receipt of non-study licensed live vaccine within 30 days prior to or 28 days after each study vaccination,
  - Receipt of non-study licensed inactivated vaccine within 14 days prior to or 28 days after each study vaccination,
  - Receipt of immunosuppressive therapy (e.g., systemic corticosteroids) or cytotoxic drugs within 30 days prior to or 28 days after each study vaccine.
- Data from any visit that occurs substantially out of window.

For analyses using the PP population, subjects will be grouped based on study vaccinations received.

All subject visits identified for exclusion from the PP population will be reviewed by the Principal Investigator, DMID Scientific Lead, and/or DMID Medical Officer.

#### **6.3.3.** Safety Population

The safety population will include all subjects who received at least one dose of the study product and will be summarized according to treatment received.

## 6.4. Covariates and Subgroups

The protocol does not define any formal subgroup analyses, and the study is not adequately powered to perform subgroup analyses. No analysis for this study has planned covariate adjustment.

## 6.5. Missing Data

Analyses for this Phase 1 study will be descriptive and are exploratory rather than confirmatory in nature. All attempts will be made to collect all data per protocol. As missing data are expected to be minimal, no imputation will be performed for missing values.

# 6.6. Interim Analyses and Data Monitoring

Interim analyses will be used to terminate this trial in the event that unanticipated safety events deemed to be of sufficient concern require such action by the sponsor. These assessments will not be made on the basis of testing a formal statistical hypothesis; therefore, p-value adjustment will not be made to any analyses. A SMC will be convened by DMID to review study progress and participant, clinical, safety, reactogenicity and immunogenicity data as described in Protocol v3.0 Section 8.7.

To guide protocol development of future studies of the candidate vaccine, interim analyses of safety data and immunogenicity assays, including the total IgG ELISA assay, will be performed as data is available for Groups A and B and again when data is available for Groups C and D prior to the completion of follow-up of all subjects. The interim immunogenicity analyses report(s) will include between-Group comparisons of those who received different Sm-p80 study product formulations and different schedules. The information from the reports may be used in abstracts and scientific presentations and reports.

#### 6.6.1. Interim Safety Review

An interim safety review may include enrollment and demographic information, medical history, concomitant medications, physical assessments, dosing compliance, and solicited and unsolicited AE/SAEs. Additional data may be requested by the SMC, and interim statistical reports may be generated as deemed necessary and appropriate by DMID. The SMC may receive data in aggregate and presented by treatment arm. The SMC will meet and review this data at scheduled time points or ad hoc as needed during this trial as defined in the SMC charter. As an outcome of each review/meeting, the SMC will make a recommendation as to the advisability of proceeding with study vaccinations (as applicable), and to continue, modify, or terminate this trial. Additionally, this trial will be monitored to determine if any of the halting rules described in Protocol v3.0 Section 8.6 are met.

# 6.6.2. Interim Immunogenicity or Efficacy Review

Interim immunogenicity analyses of, for example, total IgG ELISA responses will be performed for each Study Group, as the data is available for each study group. Depending on the timing of data availability, a report may cover one or more Study Groups. Immunogenicity reports will be provided by the SDCC to the DMID Scientific Lead and CPM, the IDCRC LOU representative(s), the study PI and investigators, and the SMC. Reports will include data summarized by Study Group. The data will be cleaned but not locked. These

reports along with interim safety results may be presented in publications, or public forums and used by the product developers for internal decision-making.

# 6.7. Multicenter Studies

Not applicable.

# 6.8. Multiple Comparisons/Multiplicity

This study is not designed to test any specific null hypothesis, and as such no adjustments for multiple testing are planned.

## 7. STUDY SUBJECTS

# 7.1. Disposition of Subjects

Table 11 will present a summary of the reasons that subjects were screened but not enrolled. The composition of analysis populations, including reasons for subject exclusion, by treatment arm, is presented in Table 9.

The disposition of subjects in the study will be tabulated by treatment group (Table 8). The table shows the total number of subjects screened, enrolled, received first dose, received second dose, received third dose, discontinued dosing or terminated from study follow-up, and the number completing the study. The number of subjects in each cohort who received study product by month will be summarized in Table 10.

A flowchart showing the disposition of study subjects, adapted from the Consort Statement will be included (Figure 1). This figure will present the number of subjects screened, enrolled, lost to follow-up, and analyzed by treatment arm.

A listing of subjects who discontinued dosing or terminated from study follow-up and the reason will be included in Listing 2.

## 7.2. Protocol Deviations

A summary of subject-specific protocol deviations will be presented by the reason for the deviation, the deviation category, and treatment group for all subjects (Table 5). Deviations that are considered major deviations that will be reviewed for possible subject exclusion from the per protocol population include: ineligibility and product deviations. All subject-specific protocol deviations and non-subject specific protocol deviations will be included in Appendix 3 as data listings (Listing 3 and Listing 4, respectively).

# 8. EFFICACY EVALUATION

Not applicable. No efficacy evaluations will be performed for the main study objectives.

## 9. SAFETY EVALUATION

All safety analyses will be presented using the safety population. Subjects will be grouped for summary statistics using treatment group. An additional "All Subjects" group will be included to summarize across groups for solicited and unsolicited AE exhibits.

Any medical condition that is present at the time that the subject is screened will be considered baseline and not reported as an AE, unless it worsens in severity or increases in frequency during the study.

# 9.1. Demographic and Other Baseline Characteristics

Summaries of age, sex, ethnicity, race, height, weight and BMI will be presented by treatment group and overall (Table 12 and Table 13). Ethnicity is categorized as Hispanic or Latino, or not Hispanic and not Latino. In accordance with NIH reporting policy, subjects may self-designate as belonging to more than one race or may refuse to identify a race, the latter reflected in the CRF as "No" to each racial option. Numeric variables will be summarized by mean and standard deviation; categorical variables will be tabulated.

Individual subject listings (Appendix 3) will be presented for all demographics (Listing 6); pre-existing medical conditions (Listing 7); vital signs and oral temperature (Listing 15); and concomitant medications (Listing 17).

#### 9.1.1. Prior and Concurrent Medical Conditions

All current illnesses and past pre-existing medical conditions will be Medical Dictionary for Regulatory Activities® (MedDRA) coded using MedDRA dictionary version 25.0 or higher.

Summaries of subjects' pre-existing medical conditions will be presented by treatment group (Table 14).

#### 9.1.2. Prior and Concomitant Medications

Summaries of medications that were started prior to dosing and continuing at the time of dosing will be presented by World Health Organization (WHO) Drug Terms 2 and 3 and treatment group (Table 83).

# **9.2.** Measurements of Treatment Compliance

Any subject receiving any number of doses of study product will be tabulated in Listing 8. The number of subjects who enrolled but were not vaccinated, the number who received any study product, and the number who received all scheduled treatments will be presented by treatment group as part of the subject disposition table (Table 8). Table 10 will present the time and number of subjects who received first dose by treatment arm.

#### 9.3. Adverse Events

When calculating the incidence of adverse events (i.e., on a per subject basis), each subject will only be counted once and any repetitions of adverse events within a subject will be ignored; the denominator will be the total population size. All adverse events reported will be included in the summaries and analyses. An overall summary of adverse events is presented in Table 18 along with adverse events occurring in the Safety Population (Table 19). A summary of the proportion of subjects with solicited and unsolicited AEs by treatment group with be presented in Table 24.

#### 9.3.1. Solicited Events and Symptoms

Systemic solicited adverse events were collected pre-vaccination, and systemic and injection site solicited adverse events were collected 30 minutes post-vaccination and then daily for 7 days after each vaccination and graded on a scale of 0 (absent), 1 (mild), 2 (moderate) and 3 (severe). Systemic events include: fever, chills, fatigue, malaise, myalgia, arthralgia, headache, nausea, and vomiting. Injection site events include: pruritus, erythema, induration/swelling, pain, and tenderness.

The proportion of subjects reporting at least one solicited adverse event will be summarized for each solicited adverse event, any systemic symptom, any injection site symptom, and any symptoms. The 95% CI calculated using Wilson score methodology from binomial distribution without continuity correction (Table 20, Table 21, Table 22, Table 23).

For each systemic and injection site event, any systemic event, any injection site event, and any solicited event, the maximum severity over 7 days after each vaccination will be summarized for the Safety population. The number and percentage of subjects reporting each event will be summarized by the maximum severity and treatment group, separately for each vaccination and over all vaccinations. For each event the denominator is the number of subjects with non-missing data for the specific event (Table 25, Table 26, Table 27, Table 28; and Figure 8, Figure 9, Figure 10, Figure 11, Figure 15, Figure 16, Figure 17, Figure 18).

The number of subjects reporting a solicited adverse event will be summarized for each day post vaccination for each vaccination and for all vaccinations combined both in a summary table beginning Table 29 and continuing through Table 43, and graphically in a bar chart (Figure 5, Figure 6, Figure 7, Figure 12, Figure 13, Figure 14). A comparison of the event rate for each treatment group between vaccination 1 and vaccination 2 and vaccination 1 and vaccination 3 will be presented (Table 44).

Solicited adverse events by subject will be presented in Listing 10 and Listing 11.

#### 9.3.2. Unsolicited Adverse Events

The proportion of subjects reporting at least one unsolicited adverse event will be summarized by MedDRA system organ class and preferred term for each vaccination and over all vaccinations. Denominators for percentages are the number of subjects who received the vaccination being summarized. The 95% CI will be calculated using Wilson score methodology from binomial distribution without continuity correction.

Adverse events by subject will be presented in Listing 12.

The following summaries for unsolicited adverse events will be presented by MedDRA system organ class, preferred term, vaccination, and treatment group:

- Subject incidence and total frequency of adverse events by treatment group and dose with 95% CI (Table 45, Table 46, Table 47);
- Summary of severity and relationship to study product (Table 48);
- Subject incidence and total frequency of related adverse events over time (Table 49, Table 50, Table 51, Table 52, Table 53);
- Subject listing of non-serious adverse events of moderate or greater severity (Table 55);
- Listing of other significant adverse events (Table 56);
- Bar chart of non-serious related adverse events by severity and MedDRA system organ class (Figure 19);

Bar chart of non-serious related adverse events by severity (Figure 20);

## 9.4. Deaths, Serious Adverse Events and other Significant Adverse Events

The following listings will be presented including Subject ID, Adverse Event Description, Adverse Event Onset Date/End Date, Last Dose Received/Days Post Dose, Reason Reported as an SAE, Relationship to Treatment, Alternate Etiology if not Related, Outcome, and Duration of Event (days):

- Deaths and Serious Adverse Events (Table 54);
- Adverse Events of Special Interest;
- New Onset Chronic Medical Conditions.

## 9.5. Pregnancies

For any subjects in the Safety population who became pregnant during the study, every attempt was made to follow these subjects to completion of pregnancy to document the outcome, including information regarding any complications with pregnancy and/or delivery. A listing of pregnancies and outcomes will be presented (Listing 18, Listing 19, Listing 20, Listing 21, Listing 22) if a pregnancy occurs post dosing.

# 9.6. Clinical Laboratory Evaluations

The distribution of laboratory results by severity, time point, and treatment group will be presented in Table 59, Table 60 and Table 61 for chemistry parameters and Table 67, Table 68, Table 69 and Table 70 for hematology parameters. Descriptive statistics including mean, standard deviation, median, minimum, and maximum values by time point, for each laboratory parameter, will be summarized in Table 65, Table 66, Table 75, Table 76 and Table 77. Changes in laboratory values will be presented in Figure 21, Figure 22, Figure 23, Figure 24 and Figure 25.

Subject visits with related laboratory results will be presented in Table 62, Table 63 and Table 64 for chemistry parameters and Table 71, Table 72, Table 73, and Table 74 for hematology parameters. A list of abnormal results will be presented in Table 57 and Table 58.

Listing 13 and Listing 14 will provide a complete listing of individual clinical laboratory results with applicable reference ranges.

# 9.7. Vital Signs and Physical Evaluations

Vital sign measurements included oral temperature, pulse, and blood pressure. Vital signs were assessed at screening visit, at vaccination visits, and at clinic visits scheduled within 7 days after vaccination. At other visits, vital signs were assessed if clinically indicated. Vital signs will be tabulated by visit and treatment group (Table 78, Table 89, Table 81, Table 82 and Listing 15).

Physical Examinations performed at screening visit. At subsequent clinic visits, a targeted physical examination may be performed, if indicated based on the subject's interim medical history, by a study clinician licensed to make medical diagnoses. Targeted physical examinations also include an assessment for signs suggestive of MAAE/NOCMC/PIMMC. A full listing of abnormal physical exam findings by subject is presented in Listing 16.

## 9.8. Concomitant Medications

Concomitant medications will be coded to the Anatomical Therapeutic Classification (ATC) using the WHO Drug Dictionary. The use of prior and concomitant medications taken during the study will be recorded on the CRFs. A by-subject listing of concomitant medication use will be presented. The use of concomitant medications during the study will be summarized by ATC1, ATC2 code and treatment group for the Safety population (Table 83).

# 9.9. Other Safety Measures

Not applicable.

# 10. PHARMACOKINETICS

Not applicable.

## 11. IMMUNOGENICITY

## 11.1. Secondary Immunogenicity Analysis

## 11.1.1. ELISA (anti Sm-p80 Total IgG)

Antibody responses, measured by total IgG production to the recombinant Sm-p80 protein using ELISA will be presented at baseline (Day 1) and by study day (Days 8, 29, 36, 57 for all treatment groups; additionally Days 64, 85, 181 for Groups A, B, D, and E, and Days 180, 187, 208, 304 for Group C) using descriptive statistics in Table 15 (mITT immunogenicity population). For post-baseline timepoints, geometric mean fold rise (GMFR) and the proportion of subjects with at least a 4-fold rise will be presented with 95% confidence intervals for mITT population in Table 16 (mITT immunogenicity population). The ELISA seroresponse (at least 4-fold rise) rates at 28-days post vaccination will be compared between Group A vaccine group and each treatment group using Fisher's Exact Test (Table 17). Confidence intervals for proportions are calculated using Wilson Score methodology without continuity correction. Confidence intervals calculated for GMT and GMFR follow a t-distribution.

Antibody responses will be adjusted for baseline. Reverse cumulative distributions (RCD) curves will be presented with separate panels for each timepoint for mITT population in Figure 2. Graphs of Geometric Mean Anti-Sm-p80 ELISA responses over time will be presented in Figure 3. Individual time trends for each Anti-Sm-p80 ELISA will be presented in Figure 4.

Results of individual total IgG immunogenicity responses, scheduled and unscheduled, will be presented in Listing 9.

# 12. OTHER ANALYSES

Not applicable.

## 13. REPORTING CONVENTIONS

P-values  $\geq 0.001$  and  $\leq 0.999$  will be reported to 3 decimal places; p-values less than 0.001 will be reported as "< 0.001" The mean, standard deviation, and other statistics will be reported to 1 decimal place greater than the original data. The minimum and maximum will use the same number of decimal places as the original data. Proportions will be presented as 2 decimal places; values greater than zero but < 0.01 will be presented as "< 0.01". Percentages will be reported to the nearest whole number; values greater than zero but < 1% will be presented as "< 1"; values greater than 99% but less than 100% will be reported as > 99%. Estimated parameters, not on the same scale as raw observations (e.g. regression coefficients) will be reported to 3 significant figures.
## 14. TECHNICAL DETAILS

All tables, figures, and listings will be generated using SAS version 9.4 or above or R version 3.4.2 or above.

# 15. SUMMARY OF CHANGES IN THE CONDUCT OF THE STUDY OR PLANNED ANALYSES

Version 2.0 of Statistical Analysis Plan incorporates the following updates:

- Section 11.2 added for exploratory immunogenicity analysis. Details of ELISA IgG subclasses were moved from Section 11.1 to Section 11.2. Section 11.1 only includes ELISA total IgG information. The exploratory immunogenicity analysis will be included in a CSR addendum, after the completion of the interim CSR.
- Tables and figures pertaining to ELISA IgG subclasses were removed from Section 6.2.

Version 3.0 of Statistical Analysis Plan incorporates the following updates:

- Removal of text related to ELISA IgG subclasses including Section 11.2 exploratory immunogenicity analysis. These exploratory analyses will no longer be performed.
- Tables and figures pertaining to ELISA IgG subclasses were removed from Appendix 1 and Appendix 2. Listings that included ELISA IgG subclasses were revised in Appendix 3.

Version 4.0 of Statistical Analysis Plan incorporates the following updates:

- Removal of exploratory endpoints with the exception of RNA-Seq in Section 3.1.3 and Section 3.2.3.
- Removal of text related to exploratory endpoints with the exception of RNA-Seq in Section 4.1 and Section 4.5.2.
- Clarifications added to Section 9.1, Section 9.3.2 and Section 9.6.

#### 16. REFERENCES

- 1. Gryseels B, Polman K, Clerinx J and Kestens L. Human schistosomiasis. Lancet 2006;368:1106-18.
- 2. Savioli L, Mott KE. Urinary schistosomiasis on Pemba Island: low-cost diagnosis for control in a primary health care setting. Parasitol Today **1989**;5:333-7.
- 3. De Vlas SJ, Engels D, Rabello AL, et al. Validation of a chart to estimate true Schistosoma mansoni prevalences from simple egg counts. Parasitology **1997**;114 ( Pt 2):113-21.
- 4. King CH. Parasites and poverty: the case of schistosomiasis. Acta Trop 2010;113:95-104.
- 5. Hotez PJ, Strych U, Lustigman S and Bottazzi ME. Human anthelminthic vaccines: Rationale and challenges. Vaccine **2016**;34:3549-55.
- 6. Mo AX, Colley DG. Workshop report: Schistosomiasis vaccine clinical development and product characteristics. Vaccine **2016**;34:995-1001.
- 7. Stylianou A, Hadjichrysanthou C, Truscott JE and Anderson RM. Developing a mathematical model for the evaluation of the potential impact of a partially efficacious vaccine on the transmission dynamics of Schistosoma mansoni in human communities. Parasit Vectors **2017**;10:294.
- 8. Ahmad G, Zhang W, Torben W, et al. Preclinical prophylactic efficacy testing of Sm-p80-based vaccine in a nonhuman primate model of Schistosoma mansoni infection and immunoglobulin G and E responses to Sm-p80 in human serum samples from an area where schistosomiasis is endemic. J Infect Dis **2011**;204:1437-49.
- 9. Zhang W, Molehin AJ, Rojo JU, et al. Sm-p80-based schistosomiasis vaccine: double-blind preclinical trial in baboons demonstrates comprehensive prophylactic and parasite transmission-blocking efficacy. Ann N Y Acad Sci **2018**;1425:38-51.
- 10. Siddiqui AJ, Molehin AJ, Zhang W, et al. Sm-p80-based vaccine trial in baboons: efficacy when mimicking natural conditions of chronic disease, praziquantel therapy, immunization, and Schistosoma mansoni re-encounter. Ann N Y Acad Sci **2018**
- 11. Karmakar S, Zhang W, Ahmad G, et al. Use of an Sm-p80-based therapeutic vaccine to kill established adult schistosome parasites in chronically infected baboons. J Infect Dis **2014**;209:1929-40.
- 12. Karmakar S, Zhang W, Ahmad G, et al. Cross-species protection: Schistosoma mansoni Sm-p80 vaccine confers protection against Schistosoma haematobium in hamsters and baboons. Vaccine **2014**;32:1296-303.
- 13. Molehin AJ, Sennoune SR, Zhang W, et al. Cross-species prophylactic efficacy of Sm-p80-based vaccine and intracellular localization of Sm-p80/Sm-p80 ortholog proteins during development in Schistosoma mansoni, Schistosoma japonicum, and Schistosoma haematobium. Parasitol Res **2017**;116:3175-3188.
- 14. Zhang W, Ahmad G, Le L, et al. Longevity of Sm-p80-specific antibody responses following vaccination with Sm-p80 vaccine in mice and baboons and transplacental transfer of Sm-p80-specific antibodies in a baboon. Parasitol Res **2014**;113:2239-50.
- 15. Coler RN, Duthie MS, Hofmeyer KA, et al. From mouse to man: safety, immunogenicity and efficacy of a candidate leishmaniasis vaccine LEISH-F3+GLA-SE. Clin Transl Immunology **2015**;4:e35.

- 16. Coler RN, Day TA, Ellis R, et al. The TLR-4 agonist adjuvant, GLA-SE, improves magnitude and quality of immune responses elicited by the ID93 tuberculosis vaccine: first-in-human trial. NPJ Vaccines **2018**;3:34.
- 17. Penn-Nicholson A, Tameris M, Smit E, et al. Safety and immunogenicity of the novel tuberculosis vaccine ID93 + GLA-SE in BCG-vaccinated healthy adults in South Africa: a randomised, double-blind, placebo-controlled phase 1 trial. Lancet Respir Med **2018**;6:287-298.
- 18. Pillet S, Aubin E, Trepanier S, et al. Humoral and cell-mediated immune responses to H5N1 plant-made virus-like particle vaccine are differentially impacted by alum and GLA-SE adjuvants in a Phase 2 clinical trial. NPJ Vaccines **2018**;3:3.
- 19. Treanor JJ, Essink B, Hull S, et al. Evaluation of safety and immunogenicity of recombinant influenza hemagglutinin (H5/Indonesia/05/2005) formulated with and without a stable oil-in-water emulsion containing glucopyranosyl-lipid A (SE+GLA) adjuvant. Vaccine **2013**;31:5760-5.
- 20. Santini-Oliveira M, Coler RN, Parra J, et al. Schistosomiasis vaccine candidate Sm14/GLA-SE: Phase 1 safety and immunogenicity clinical trial in healthy, male adults. Vaccine **2016**;34:586-594.
- 21. Sirima SB, Durier C, Kara L, et al. Safety and immunogenicity of a recombinant Plasmodium falciparum AMA1-DiCo malaria vaccine adjuvanted with GLA-SE or Alhydrogel(R) in European and African adults: A phase 1a/1b, randomized, double-blind multi-centre trial. Vaccine **2017**;35:6218-6227.
- 22. Belshe RB, Frey SE, Graham I, et al. Safety and immunogenicity of influenza A H5 subunit vaccines: effect of vaccine schedule and antigenic variant. J Infect Dis **2011**;203:666-73.
- 23. Marsano LS, Greenberg RN, Kirkpatrick RB, et al. Comparison of a rapid hepatitis B immunization schedule to the standard schedule for adults. Am J Gastroenterol **1996**;91:111-5.
- 24. Madan A, Segall N, Ferguson M, et al. Immunogenicity and Safety of an AS03-Adjuvanted H7N9 Pandemic Influenza Vaccine in a Randomized Trial in Healthy Adults. J Infect Dis **2016**;214:1717-1727.
- 25. Kim D, Langmead B and Salzberg SL. HISAT: a fast spliced aligner with low memory requirements. Nat Methods **2015**;12:357-60.
- 26. Liao Y, Smyth GK and Shi W. featureCounts: an efficient general purpose program for assigning sequence reads to genomic features. Bioinformatics **2014**;30:923-30.
- 27. Aken BL, Achuthan P, Akanni W, et al. Ensembl 2017. Nucleic Acids Res 2017;45:D635-D642.
- 28. Robinson MD, McCarthy DJ and Smyth GK. edgeR: a Bioconductor package for differential expression analysis of digital gene expression data. Bioinformatics **2010**;26:139-40.
- 29. Siddiqui AA, Pinkston JR, Quinlin ML, et al. Characterization of the immune response to DNA vaccination strategies for schistosomiasis candidate antigen, Sm-p80 in the baboon. Vaccine **2005**;23:1451-6.
- 30. Torben W, Ahmad G, Zhang W, et al. Role of antibody dependent cell mediated cytotoxicity (ADCC) in Sm-p80-mediated protection against Schistosoma mansoni. Vaccine **2012**;30:6753-8.

# **APPENDICES**

# APPENDIX 1. TABLE MOCK-UPS

# LIST OF TABLES

| Table 1: | Study Design | 48 |
|---|---|---|
| Table 2: | Schedule of Events and Study Procedures, Study Groups A, B, D, and E | 49 |
| Table 3: | Schedule of Events and Study Procedures, Study Group C | 52 |
| Table 4: | Sample Size/Probability Estimates | 54 |
| Table 5: | Distribution of Protocol Deviations by Category, Type, and Treatment<br>Group | 55 |
| Table 6: | Solicited Adverse Event Grading Scale | 58 |
| Table 7: | Laboratory Adverse Event Grading Scale | |
| Table 8: | Subject Disposition by Treatment Group | 61 |
| Table 9: | Analysis Populations by Treatment Group | |
| Table 10: | Dates of First Treatment by Treatment Group | |
| Table 11: | Ineligibility Summary of Screen Failures | |
| Table 12: | Summary of Categorical Demographic and Baseline Characteristics by Treatment Group, All Enrolled Subjects | |
| Table 13: | Summary of Continuous Demographic and Baseline Characteristics by Treatment Group | 66 |
| Table 14: | Summary of Subjects with Pre-Existing Medical Conditions by MedDRA System Organ Class and Treatment Group | 67 |
| Table 15: | Anti-Sm-p80 ELISA Total IgG Geometric Mean Titers (GMT) Results with 95% Confidence Intervals by Time Point and Treatment Group, mITT Immunogenicity Population | 68 |
| Table 16: | Anti-Sm-p80 ELISA Total IgG Geometric Mean Fold Rise (GMFR) and Seroconversion Results by Time Point and Treatment Group, mITT Immunogenicity Population | |
| Table 17: | Comparison of Anti-Sm-p80 ELISA Total IgG Seroresponse Rates between Group A and Each Treatment Group 28-Days Post Dose – mITT Immunogenicity Population | |
| Table 18: | Overall Summary of Adverse Events | |
| Table 19: | Adverse Events Occurring in 5% of Subjects in Any Treatment MedDRA System Organ Class and Preferred Term, and Treatment Group - Safety Population | |
| Table 20: | Number and Percentage of Subjects Experiencing Solicited Events with 95% Confidence Intervals by Symptom and Treatment Group – Post Dose 1 | |
| Table 21: | Number and Percentage of Subjects Experiencing Solicited Events with 95% Confidence Intervals by Symptom and Treatment Group – Post Dose 2 | 84 |

| Table 22: | Number and Percentage of Subjects Experiencing Solicited Events with 95% Confidence Intervals by Symptom and Treatment Group – Post Dose 3 | 84 |
|---|---|---|
| Table 23: | Number and Percentage of Subjects Experiencing Solicited Events with 95% Confidence Intervals by Symptom and Treatment Group – Post Any Dose | 84 |
| Table 24: | Comparison of the Proportion of Subjects Experiencing Solicited Events by Treatment Group. | 85 |
| Table 25: | Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Maximum Severity, and Treatment Group – Post Dose 1 | 86 |
| Table 26: | Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Maximum Severity, and Treatment Group – Post Dose 2 | 88 |
| Table 27: | Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Maximum Severity, and Treatment Group – Post Dose 3 | 88 |
| Table 28: | Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Maximum Severity, and Treatment Group – Post Any Dose | 88 |
| Table 29: | Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Severity, and Day Post Dosing – Group A: 100 µg Sm-p80 (unadjuvanted), Post Dose 1 | 89 |
| Table 30: | Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Severity, and Day Post Dosing – Group A: 100 µg Sm-p80 (unadjuvanted), Post Dose 2 | 93 |
| Table 31: | Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Severity, and Day Post Dosing – Group A: 100 µg Sm-p80 (unadjuvanted), Post Dose 3 | 93 |
| Table 32: | Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Severity, and Day Post Dosing – Group B: 10 µg Sm-p80 + 5 µg GLA-SE, Post Dose 1 | 93 |
| Table 33: | Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Severity, and Day Post Dosing – Group B: 10 µg Sm-p80 + 5 µg GLA-SE, Post Dose 2 | 93 |
| Table 34: | Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Severity, and Day Post Dosing – Group B: 10 µg Sm-p80 + 5 µg GLA-SE, Post Dose 3 | 93 |
| Table 35: | Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Severity, and Day Post Dosing – Group C: 30 µg Sm-p80 + 5 µg GLA-SE (delayed booster), Post Dose 1 | 93 |
| Table 36: | Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Severity, and Day Post Dosing – Group C: 30 µg Sm-p80 + 5 µg GLA-SE (delayed booster), Post Dose 2 | 93 |

| Table 37: | Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Severity, and Day Post Dosing – Group C: 30 µg Sm-p80 + 5 µg GLA-SE (delayed booster), Post Dose 3 | 93 |
|---|---|---|
| Table 38: | Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Severity, and Day Post Dosing – Group D: 30 $\mu$ g Sm-p80 + 5 $\mu$ g GLA-SE, Post Dose 1 | 93 |
| Table 39: | Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Severity, and Day Post Dosing – Group D: 30 $\mu$ g Sm-p80 + 5 $\mu$ g GLA-SE, Post Dose 2 | 93 |
| Table 40: | Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Severity, and Day Post Dosing – Group D: 30 µg Sm-p80 + 5 µg GLA-SE, Post Dose 3 | 93 |
| Table 41: | Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Severity, and Day Post Dosing – Group E: 100 µg Sm-p80 + 5 µg GLA-SE, Post Dose 1 | 93 |
| Table 42: | Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Severity, and Day Post Dosing – Group E: 100 µg Sm-p80 + 5 µg GLA-SE, Post Dose 2 | 93 |
| Table 43: | Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Severity, and Day Post Dosing – Group E: 100 µg Sm-p80 + 5 µg GLA-SE, Post Dose 3 | 93 |
| Table 44: | Number and Percentage of Subjects Experiencing Solicited Events for Dose 1 Compared with Dose 2 and Dose 3 by Treatment Group | 94 |
| Table 45: | Summary of Unsolicited Adverse Events by MedDRA System Organ Class and Preferred Term, and Treatment Group – Post Dose 1 | 98 |
| Table 46: | Summary of Unsolicited Adverse Events by MedDRA System Organ Class and Preferred Term, and Treatment Group – Post Dose 2 | 98 |
| Table 47: | Summary of Unsolicited Adverse Events by MedDRA System Organ Class and Preferred Term, and Treatment Group – Post Dose 3 | 98 |
| Table 48: | Unsolicited Adverse Events by MedDRA System Organ Class and Preferred Term, Maximum Severity, Relationship, and Treatment Group | 99 |
| Table 49: | Related Unsolicited Adverse Events Within 28 Days Post Dosing by MedDRA System Organ Class and Preferred Term and Dose – Group A: 100 µg Sm-p80 (unadjuvanted) (N=X) | 100 |
| Table 50: | Related Unsolicited Adverse Events Within 28 Days Post Dosing by MedDRA System Organ Class and Preferred Term, and Dose – Group B: 10 µg Sm-p80 + 5 µg GLA-SE (N=X) | 100 |
| Table 51: | Related Unsolicited Adverse Events Within 28 Days Post Dosing by MedDRA System Organ Class and Preferred Term, and Dose – Group C: 30 µg Sm-p80 + 5 µg GLA-SE (delayed booster) (N=X) | 100 |

| Table 52: | Related Unsolicited Adverse Events Within 28 Days Post Dosing by MedDRA System Organ Class and Preferred Term, and Dose – Group D: 30 µg Sm-p80 + 5 µg GLA-SE (N=X) | 100 |
|---|---|---|
| Table 53: | Related Unsolicited Adverse Events Within 28 Days Post Dosing by MedDRA System Organ Class and Preferred Term, and Dose – Group E: 100 µg Sm-p80 + 5 µg GLA-SE (N=X) | 100 |
| Table 54: | Listing of Serious Adverse Events | 101 |
| Table 55: | Listing of Non-Serious, Unsolicited, Moderate or Severe Adverse Events | 102 |
| Table 56: | Listing of Other Significant Adverse Events | 103 |
| Table 57: | Listing of Abnormal Laboratory Results - Chemistry | 105 |
| Table 58: | Listing of Abnormal Laboratory Results - Hematology | 106 |
| Table 59: | Laboratory Results by Parameter, Maximum Severity, Time Point, and Treatment Group – Any Chemistry Parameter | 107 |
| Table 60: | Laboratory Results by Parameter, Maximum Severity, Time Point, and Treatment Group – Creatinine | 109 |
| Table 61: | Laboratory Results by Parameter, Maximum Severity, Time Point, and Treatment Group Alanine Aminotransferase | 109 |
| Table 62: | Abnormal Laboratory Results Related to Study Treatment by Parameter, Maximum Severity, Time Point, and Treatment Group – Any Chemistry Parameter | 110 |
| Table 63: | Abnormal Laboratory Results Related to Study Treatment by Parameter,<br>Maximum Severity, Time Point, and Treatment Group – Creatinine | 113 |
| Table 64: | Abnormal Laboratory Results Related to Study Treatment by Parameter, Maximum Severity, Time Point, and Treatment Group – Alanine Aminotransferase | 113 |
| Table 65: | Laboratory Summary Statistics by Parameter, Time Point, and Treatment Group – Creatinine (mg/dL) | 114 |
| Table 66: | Laboratory Summary Statistics by Parameter, Time Point, and Treatment<br>Group – Alanine Aminotransferase (IU/L) | 116 |
| Table 67: | Laboratory Results by Parameter, Maximum Severity, Time Point, and Treatment Group – Any Hematology Parameter | 117 |
| Table 68: | Laboratory Results by Parameter, Maximum Severity, Time Point, and Treatment Group – White Blood Cells | 119 |
| Table 69: | Laboratory Results by Parameter, Maximum Severity, Time Point, and Treatment Group – Hemoglobin | 119 |
| Table 70: | Laboratory Results by Parameter, Maximum Severity, Time Point, and Treatment Group – Platelets | 119 |

| Table 71: | Abnormal Laboratory Results Related to Study Treatment by Parameter, Maximum Severity, Time Point, and Treatment Group – Any Hematology Parameter | 120 |
|---|---|---|
| Table 72: | Abnormal Laboratory Results Related to Study Treatment by Parameter,<br>Maximum Severity, Time Point, and Treatment Group – White Blood Cells | 122 |
| Table 73: | Abnormal Laboratory Results Related to Study Treatment by Parameter, Maximum Severity, Time Point, and Treatment Group – Hemoglobin | 122 |
| Table 74: | Abnormal Laboratory Results Related to Study Treatment by Parameter,<br>Maximum Severity, Time Point, and Treatment Group – Platelets | 122 |
| Table 75: | Laboratory Summary Statistics by Parameter, Time Point, and Treatment Group – White Blood Cells (10 <sup>9</sup> /L) | 123 |
| Table 76: | Laboratory Summary Statistics by Parameter, Time Point, and Treatment Group – Hemoglobin (g/dL) | 125 |
| Table 77: | Laboratory Summary Statistics by Parameter, Time Point, and Treatment Group – Platelets (10 <sup>9</sup> /L) | 125 |
| Table 78: | Vital Signs by Assessment, Maximum Severity, Time Point, and Treatment<br>Group – Any Assessment | 126 |
| Table 79: | Vital Signs by Assessment, Maximum Severity, Time Point, and Treatment<br>Group – Systolic Blood Pressure | 129 |
| Table 80: | Vital Signs by Assessment, Maximum Severity, Time Point, and Treatment<br>Group – Diastolic Blood Pressure | 129 |
| Table 81: | Vital Signs by Assessment, Maximum Severity, Time Point, and Treatment Group – Heart Rate | 129 |
| Table 82: | Vital Signs by Assessment, Maximum Severity, Time Point, and Treatment<br>Group – Oral Temperature | 129 |
| Table 83: | Number and Percentage of Subjects with Prior and Concurrent Medications by WHO Drug Classification and Treatment Group | 130 |

# 9.1 Overall Study Design and Plan Description

Table 1: Study Design

| Study | N | Study Product | Administration Schedule |
|-------|---|------------------------------|----------------------------------|
| Group | | | |
| A | 9 | 100 μg Sm-p80 (unadjuvanted) | Day 1, 29, 57 |
| В | 9 | 10 μg Sm-p80 + 5 μg GLA-SE | Day 1, 29, 57 |
| С | 9 | 30 μg Sm-p80 + 5 μg GLA-SE | Day 1, 29, 180 (delayed booster) |
| D | 9 | 30 μg Sm-p80 + 5 μg GLA-SE | Day 1, 29, 57 |
| E | 9 | 100 μg Sm-p80 + 5 μg GLA-SE | Day 1, 29, 57 |

### 9.5.1 Efficacy/Immunogenicity and Safety Measurements Assessed and Flow Chart

Table 2: Schedule of Events and Study Procedures, Study Groups A, B, D, and E

| | | | Study Product Injection and Follow Up Visits | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study day | | 1 | 2 | 4 | 8 | 29 | 32 | 36 | 57 | 60 | 64 | 85 | 181 | 422 |
| Days after most recent vaccination | | 0 | 1 | 3 | 7 | 28 | 3 | 7 | 28 | 3 | 7 | 28 | 124 | 365 |
| Visit Window (± number of days) | | 0 | 0 | 1 | 1 | 3 | 1 | 1 | 3 | 1 | 1 | 3 | 14 | 14 |
| Study visit | | 01 | 02P | 03 | 04 | 05 | 06 | 07 | 08 | 09 | 10 | 11 | 12 | 13P |
| Clinical Evaluations and Procedures | Tube | | | | | | | | | | | | | |
| Assessment of eligibility | | X | | | | | | | | | | | | |
| Assessment of individual halting criteria | | | | | | X | | | X | | | | | |
| Review medical history and con meds <sup>3</sup> | | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Vital signs (blood<br>pressure, pulse, and<br>oral temperature <sup>5</sup> ) | | X | | X | X | X | X | X | X | X | X | X <sup>4</sup> | X <sup>4</sup> | |
| Enrollment | | X | | | | | | | | | | | | |
| Study Product<br>Injection <sup>1</sup> | | I-1 | | | | I-2 | | | I-3 | | | | | |
| Targeted physical exam | | {X} | | {X} | {X} | {X} | {X} | {X} | {X} | {X} | {X} | {X} | {X} | |
| Pre-administration reactogenicity assessment | | X | | | | X | | | X | | | | | |
| Evaluate study product injection site | | X | | X | X | X | X | X | X | X | X | | | |

Table 2: Schedule of Events and Study Procedures, Study Groups A, B, D, and E (Continued)

| | | | | | | | | | | | | | | - |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | St | tudy Proc | luct Inje | tion and | Follow U | Jp Visits | | | | | |
| Study day | | 1 | 2 | 4 | 8 | 29 | 32 | 36 | 57 | 60 | 64 | 85 | 181 | 422 |
| Days after most recent vaccination | | 0 | 1 | 3 | 7 | 28 | 3 | 7 | 28 | 3 | 7 | 28 | 124 | 365 |
| Visit Window (± number of days) | | 0 | 0 | 1 | 1 | 3 | 1 | 1 | 3 | 1 | 1 | 3 | 14 | 14 |
| Study visit | | 01 | 02P | 03 | 04 | 05 | 06 | 07 | 08 | 09 | 10 | 11 | 12 | 13P |
| Clinical Evaluations and Procedures | Tube | | | | | | | | | | | | | |
| Provide and explain use of memory aid and thermometer | | X | | | | X | | | X | | | | | |
| Review memory aid | | | X | X | X | | X | X | | X | X | | | |
| Collection of solicited AEs | | X | X | X | X | X | X | X | X | X | X | | | |
| Collection of<br>unsolicited AEs and<br>SAEs <sup>3</sup> | | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Pregnancy test (urine) <sup>2</sup> | | X | | | | X | | | X | | | | | |
| WBC, hemoglobin, platelets (mL) | EDTA | 3 | | | 3 | 3 | | 3 | 3 | | 3 | 3 | | |
| Creatinine, ALT <sup>6</sup> | SST | 10 | | | 10 | 10 | | 10 | 10 | | 10 | 10 | | |
| Serum collection for<br>antibody assays and<br>secondary research<br>(mL) | SST | 8.5 | | | 8.5 | 8.5 | | 8.5 | 8.5 | | 8.5 | 8.5 | 8.5 | |
| PBMC isolation for<br>secondary research<br>(mL) | NaHep/ACD <sup>7</sup> | 60 | | | 60 | 60 | | 60 | 60 | | 60 | 34 | 60 | |
| Whole blood collection for gene expression assays | PAXGene | 2.5 | | | 2.5 | 2.5 | | 2.5 | 2.5 | | 2.5 | | | |

Table 2: Schedule of Events and Study Procedures, Study Groups A, B, D, and E (Continued)

| | | | | St | tudy Proc | duct Injec | ction and | Follow U | Jp Visits | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study day | | 1 | 2 | 4 | 8 | 29 | 32 | 36 | 57 | 60 | 64 | 85 | 181 | 422 |
| Days after most recent vaccination | | 0 | 1 | 3 | 7 | 28 | 3 | 7 | 28 | 3 | 7 | 28 | 124 | 365 |
| Visit Window (± number of days) | | 0 | 0 | 1 | 1 | 3 | 1 | 1 | 3 | 1 | 1 | 3 | 14 | 14 |
| Study visit | | 01 | 02P | 03 | 04 | 05 | 06 | 07 | 08 | 09 | 10 | 11 | 12 | 13P |
| Clinical Evaluations and Procedures | Tube | | | | | | | | | | | | | |
| Total volume per visit (mL) | | 84 | | | 84 | 84 | | 84 | 84 | | 84 | 55.5 | 68.5 | |
| Cumulative volume (prior 56 days) | | 113.5 | | | 197.5 | 281.5 | | 365.5 | 420 | | 420 | 391.5 | 68.5 | |

<sup>{ }</sup> required at this visit only if clinically indicated

<sup>1</sup>0.5 mL of the designated study product will be injected IM in the deltoid muscle. Prior to the injection, a pre-administration reactogenicity assessment will be performed to establish baseline. After the injection, subjects will be observed for 30 minutes. The injection site will be evaluated and vital signs obtained during that period and before the subject leaves the clinic. Subjects will be provided with a Memory Aid and thermometer for recording daily maximum oral temperature, solicited injection site and systemic reactions, unsolicited AEs, and concomitant medications, beginning on the evening of the day of study product injection and continuing daily for the next seven days. Subjects will be encouraged to take their temperature around the same time each day and also if they feel feverish. Subjects will be instructed on how to use the memory aid and how to rate any AEs. Subjects will also be instructed to notify the study center if they develop any severe reactions and/or fever ≥ 38°C (100.4°F).

<sup>2</sup>For women of childbearing potential. Must be confirmed as negative prior to injection of study product. The visit will also include review of contraceptive/menstrual history and pregnancy avoidance counseling.

<sup>3</sup>After Study Visit 11 (or Study Day 85 if Study Visit 11 is not attended), through the end of study follow-up (Day 422), only SAEs, MAAEs, NOCMCs, and PIMMCs will be collected. Other unsolicited AEs and concomitant medications will not be collected.

Subjects must not eat or drink anything hot or cold, or smoke within 10 minutes prior to taking oral temperature.

Blood collection volumes shown are the maximum that may potentially be drawn from the participant at each visit based on collection tube availability.

ACD collection tubes can be used to collect blood that will be processed for PBMC if appropriate NaHep tubes are unavailable.

P = phone assessment

<sup>&</sup>lt;sup>4</sup>Vital signs will be assessed only if clinically indicated.

 Table 3:
 Schedule of Events and Study Procedures, Study Group C

| | | Stud | y Prod | uct Inj | ection a | nd Fol | low Up | Visits | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study day | | 1 | 2 | 4 | 8 | 29 | 32 | 36 | 57 | 180 | 183 | 187 | 208 | 304 | 545 |
| Days after most recent vaccination | | 0 | 1 | 3 | 7 | 28 | 3 | 7 | 28 | 151 | 3 | 7 | 28 | 124 | 365 |
| Visit Window (± number of days) | | 0 | 0 | 1 | 1 | 3 | 1 | 1 | 3 | 7 | 1 | 1 | 3 | 14 | 14 |
| Study visit | | 01 | 02P | 03 | 04 | 05 | 06 | 07 | 08 | 09 | 10 | 11 | 12 | 13 | 14P |
| Clinical Evaluations and Procedures | Tube | | | | | | | | | | | | | | |
| Assessment of eligibility | | X | | | | | | | | | | | | | |
| Assessment of individual halting criteria | | | | | | X | | | | X | | | | | |
| Review medical history and con meds <sup>3</sup> | | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Vital signs (blood pressure, pulse, and oral temperature <sup>5</sup> ) | | X | | X | X | X | X | X | X | X | X | X | x <sup>4</sup> | X <sup>4</sup> | |
| Enrollment | | X | | | | | | | | | | | | | |
| Study Product Injection <sup>1</sup> | | I-1 | | | | I-2 | | | | I-3 | | | | | |
| Targeted physical exam | | {X} | | {X} | {X} | {X} | {X} | {X} | {X} | {X} | {X} | {X} | {X} | {X} | |
| Pre-administration reactogenicity assessment | | X | | | | X | | | | X | | | | | |
| Evaluate study product injection site | | X | | X | X | X | X | X | | X | X | X | | | |
| Provide and explain use of memory aid andthermometer | | X | | | | Х | | | | X | | | | | |
| Review memory aid | | | X | X | X | | X | X | | | X | X | | | |
| Collection of solicited AEs | | X | X | X | X | X | X | X | | X | X | X | | | |
| Collection of unsolicited AEs and SAEs <sup>3</sup> | | X | X | X | X | X | X | X | $X^3$ | X | X | X | X | X | X |
| Pregnancy test (urine) <sup>2</sup> | | X | | | | X | | | | X | | | | | |
| WBC, hemoglobin, platelets (mL) | EDTA | 3 | | | 3 | 3 | | 3 | 3 | 3 | | 3 | 3 | | |
| Creatinine, ALT <sup>6</sup> | SST | 10 | | | 10 | 10 | | 10 | 10 | 10 | | 10 | 10 | | |
| Serum collection for antibody assays and secondary research (mL) | SST | 8.5 | | | 8.5 | 8.5 | | 8.5 | 8.5 | 8.5 | | 8.5 | 8.5 | 8.5 | |
| PBMC isolation for secondary research (mL) | NaHep/ACD <sup>7</sup> | 60 | | | 60 | 60 | | 60 | 60 | 60 | | 60 | 34 | 60 | |

Table 3: Schedule of Events and Study Procedures, Study Group C (Continued)

| | | Stud | y Prod | uct Inj | ection a | nd Fol | low Up | Visits | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study day | | 1 | 2 | 4 | 8 | 29 | 32 | 36 | 57 | 180 | 183 | 187 | 208 | 304 | 545 |
| Days after most recent vaccination | | 0 | 1 | 3 | 7 | 28 | 3 | 7 | 28 | 151 | 3 | 7 | 28 | 124 | 365 |
| Visit Window (± number of days) | | 0 | 0 | 1 | 1 | 3 | 1 | 1 | 3 | 7 | 1 | 1 | 3 | 14 | 14 |
| Study visit | | 01 | 02P | 03 | 04 | 05 | 06 | 07 | 08 | 09 | 10 | 11 | 12 | 13 | 14P |
| Clinical Evaluations and Procedures | Tube | | | | | | | | | | | | | | |
| Whole blood collection for gene expression assays | PAXGene | 2.5 | | | 2.5 | 2.5 | | 2.5 | | 2.5 | | 2.5 | | | |
| Total volume per visit (mL) | | 84 | | | 84 | 84 | | 84 | 84 | 84 | | 84 | 55.5 | 68.5 | |
| Cumulative volume (prior 56 days) | | 113.5 | | | 197.5 | 281.5 | | 365.5 | 420 | 84 | | 168 | 223.5 | 68.5 | |

<sup>{ }</sup> required at this visit only if clinically indicated

<sup>1</sup>0.5 mL of the designated study product will be injected IM in the deltoid muscle. Prior to the injection, a pre-administration reactogenicity assessment will be performed to establish baseline. After the injection, subjects will be observed for 30 minutes. The injection site will be evaluated and vital signs obtained during that period and before the subject leaves the clinic. Subjects will be provided with a Memory Aid and thermometer for recording daily maximum oral temperature, solicited injection site and systemic reactions, unsolicited AEs, and concomitant medications, beginning on the evening of the day of study product injection and continuing daily for the next seven days. Subjects will be encouraged to take their temperature around the same time each day and also if they feel feverish. Subjects will be instructed on how to use the memory aid and how to rate any AEs. Subjects will also be instructed to notify the study center if they develop any severe reactions and/or fever ≥ 38°C (100.4°F).

<sup>2</sup>For women of childbearing potential. Must be confirmed as negative prior to injection of study product. The visit will also include review of contraceptive/menstrual history and pregnancy avoidance counseling.

After Study Visit 8 (or Study Day 57 if Study Visit 8 is not attended), through the time of the third study vaccination at Study Visit 09, only SAEs, MAAEs, NOCMCs, and PIMMCs will be collected. Other unsolicited AEs and concomitant medications will not be collected during this period. Collection of unsolicited AEs and concomitant medications will then resume at the time of the third vaccination and continue through Study Visit 12 (or Study Day 208 if Study Visit 12 is not attended), after which only SAEs, MAAEs, NOCMCs, and PIMMCs will be collected.

<sup>4</sup>Vital signs will be assessed only if clinically indicated.

Subjects must not eat or drink anything hot or cold, or smoke within 10 minutes prior to taking oral temperature.

<sup>6</sup>Blood collection volumes shown are the maximum that may potentially be drawn from the participant at each visit based on collection tube availability.

ACD collection tubes can be used to collect blood that will be processed for PBMC if appropriate NaHep tubes are unavailable.

P = phone assessment

## 9.7.1 Sample Size

**Table 4:** Sample Size/Probability Estimates

| Probability of event after receiving studyproduct | Probability of observing event among 9 subjects | Probability of observing event among 45 subjects |
|---|---|---|
| 0.01 | 0.086 | 0.364 |
| 0.05 | 0.370 | 0.901 |
| 0.10 | 0.613 | 0.991 |
| 0.15 | 0.768 | 0.999 |
| 0.20 | 0.866 | >0.99 |
| 0.25 | 0.925 | >0.99 |

#### 10.2 Protocol Deviations

#### Table 5: Distribution of Protocol Deviations by Category, Type, and Treatment Group

[Implementation Note: Only deviation types with at least one deviation observed in any treatment group will be shown. If none observed, that deviation type will not be shown.]

| | | Group A:<br>100 μg Sm-p80<br>(unadjuvanted)<br>(N=X) | | Group B:<br>10 µg Sm-p80 + 5<br>µg GLA-SE<br>(N=X) | | Group C:<br>30 µg Sm-p80 + 5<br>µg GLA-SE<br>(delayed booster)<br>(N=X) | | 30 μg Sm-p80 + 5<br>μg GLA-SE<br>(N=X) | | Group E:<br>100 μg Sm-p80 +<br>5 μg GLA-SE<br>(N=X) | | All Subjects<br>(N=X) | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Category | Deviation Type | No. of<br>Subj. | No. of<br>Dev. | No. of<br>Subj. | No. of<br>Dev. | No. of<br>Subj. | No. of<br>Dev. | No. of<br>Subj. | No. of<br>Dev. | No. of<br>Subj. | No. of<br>Dev. | No. of<br>Subj. | No. of<br>Dev. |
| Eligibility/enrollment | Any type | | | | | | | | | | | | |
| | Did not meet inclusion criterion | x | X | x | x | x | x | x | X | x | X | X | X |
| | Met exclusion criterion | | | | | | | | | | | | |
| | ICF not signed prior to study procedures | | | | | | | | | | | | |
| | Other | | | | | | | | | | | | |
| Treatment administration schedule | Any type | | | | | | | | | | | | |
| | Out of window visit | | | | | | | | | | | | |
| | Missed visit/visit not conducted | | | | | | | | | | | | |
| | Missed treatment administration | | | | | | | | | | | | |
| | Delayed treatment administration | | | | | | | | | | | | |
| | Other | | | | | | | | | | | | |
| Follow-up visit schedule | Any type | | | | | | | | | | | | |

 Table 5: Distribution of Protocol Deviations by Category, Type, and Treatment Group (Continued)

| | | Group A:<br>100 μg Sm-p80<br>(unadjuvanted)<br>(N=X) | | Group B:<br>10 µg Sm-p80 + 5<br>µg GLA-SE<br>(N=X) | | Group C:<br>30 µg Sm-p80 + 5<br>µg GLA-SE<br>(delayed booster)<br>(N=X) | | 30 μg Sm-p80 + 5 | | Group E:<br>100 μg Sm-p80 +<br>5 μg GLA-SE<br>(N=X) | | All Subjects<br>(N=X) | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Category | Deviation Type | No. of<br>Subj. | No. of<br>Dev. | No. of<br>Subj. | No. of<br>Dev. | No. of<br>Subj. | No. of<br>Dev. | No. of<br>Subj. | No. of<br>Dev. | No. of<br>Subj. | No. of<br>Dev. | No. of<br>Subj. | No. of<br>Dev. |
| | Out of window visit | | | | | | | | | | | | |
| | Missed visit/visit not conducted | | | | | | | | | | | | |
| | Other | | | | | | | | | | | | |
| Protocol procedure/assessment | Any type | | | | | | | | | | | | |
| | Incorrect version of ICF signed | | | | | | | | | | | | |
| | Blood not collected | | | | | | | | | | | | |
| | Urine not collected | | | | | | | | | | | | |
| | Stool not collected | | | | | | | | | | | | |
| | Other specimen not collected | | | | | | | | | | | | |
| | Too few aliquots obtained | | | | | | | | | | | | |
| | Specimen result not obtained | | | | | | | | | | | | |
| | Required procedure not conducted | | | | | | | | | | | | |
| | Required procedure done incorrectly | | | | | | | | | | | | |
| | Study product temperature excursion | | | | | | | | | | | | |

Table 5: Distribution of Protocol Deviations by Category, Type, and Treatment Group (Continued)

| | Deviation Type | Group A:<br>100 μg Sm-p80<br>(unadjuvanted)<br>(N=X) | | Group B:<br>10 μg Sm-p80 + 5<br>μg GLA-SE<br>(N=X) | | Group C:<br>30 µg Sm-p80 + 5<br>µg GLA-SE<br>(delayed booster)<br>(N=X) | | Group D:<br>30 µg Sm-p80 + 5<br>µg GLA-SE<br>(N=X) | | Group E:<br>100 μg Sm-p80 +<br>5 μg GLA-SE<br>(N=X) | | All Subjects<br>(N=X) | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Category | | No. of<br>Subj. | No. of<br>Dev. | No. of<br>Subj. | No. of<br>Dev. | No. of<br>Subj. | No. of<br>Dev. | No. of<br>Subj. | No. of<br>Dev. | No. of<br>Subj. | No. of<br>Dev. | No. of<br>Subj. | No. of<br>Dev. |
| | Specimen temperature excursion | | | | | | | | | | | | |
| | Other | | | | | | | | | | | | |
| Treatment administration | Any type | | | | | | | | | | | | |
| | Required procedure done incorrectly | | | | | | | | | | | | |
| | Study product temperature excursion | | | | | | | | | | | | |
| Note: N - Number of cubic | Other | | | | | | | | | | | | |

#### 12.2.2 Displays of Adverse Events

#### **Table 6:** Solicited Adverse Event Grading Scale

Pulse and Blood Pressure

| | Mild<br>(Grade 1) | Moderate<br>(Grade 2) | Severe<br>(Grade 3) |
|---|---|---|---|
| Physiologic Parameter | | | |
| Tachycardia - beats per minute | 101 – 115 | 116 – 130 | > 130 |
| Hypotension (systolic) mm Hg <sup>1</sup> | 85 – 89 | 80 - 84 | < 80 |
| Hypertension (systolic) mm Hg <sup>2</sup> | 141 - 150 | 151 – 155 | > 155 |
| Hypertension (diastolic) mm Hg <sup>3</sup> | 96 – 100 | 101 – 105 | >105 |

The inclusion criteria for systolic blood pressure includes values from 85 through 150, inclusive and for diastolic blood pressure includes values  $\leq 100$ .

<sup>1</sup>Subjects with baseline (prior to first vaccination) Grade 1 values of 85-89 mm Hg are defined with a hypotension (systolic) AE only due to post-vaccination values ≤ 84 mm Hg and the AE isDefined as Grade 1 based on values of 80 through 84 and Grade 2 based on values less than 80.

<sup>2</sup>Subjects with baseline (prior to first vaccination) Grade 1 values of 141-150 mm Hg are defined with a hypertension (systolic) AE only due to post-vaccination values over 150 mm Hg and the AE is Defined as Grade 1 based on values of 151 through 155 mm Hg and Grade 2 based on values over 155.

<sup>3</sup>Subjects with baseline (prior to first vaccination) Grade 1 values of 96-100 mm Hg are defined with a hypertension (diastolic) AE only due to post-vaccination values ≥ 101 mm Hg and the AEis Defined as Grade 1 based on values of 101 through 105 mm Hg and Grade 2 based on values over 105.

 Table 6:
 Solicited Adverse Event Grading Scale (Continued)

Clinical Adverse Events

| | Mild<br>(Grade 1) | Moderate<br>(Grade 2) | Severe<br>(Grade 3) |
|---|---|---|---|
| Cardiovascular | , | , | , |
| Arrhythmia | | Asymptomatic, transient signs, no Rx required | Recurrent/persistent;<br>symptomatic Rx required |
| Hemorrhage, Blood Loss | Estimated blood loss ≤ 100 mL | Estimated blood loss > 100 mL, no transfusion required | Transfusionrequired |
| Respiratory | | | |
| Cough | Transient- notreatment | Persistent cough; | Interferes withdaily activities |
| Bronchospasm, Acute | Transient; no treatment; 71% – 80% FEV1 of peak flow | Requires treatment;<br>normalizes with<br>bronchodilator; FEV1<br>60% – 70% (of peak<br>flow) | No normalizationwith<br>bronchodilator; FEV1 <<br>60% of peak flow |
| Dyspnea | Does not interfere with usual and social activities | Interferes with usual and social activities, no treatment | Prevents daily and usual social activityor requires treatment |
| Gastrointestinal | | | |
| Vomiting | No interference with activity or 1 - 2 episodes/24hours | Some interference with activity or > 2 episodes/24hours | Prevents daily activity or requiresIV hydration |
| Diarrhea | 2 - 3 loose or watery<br>stools or < 400 gms/24<br>hours | 4 - 5 loose or watery<br>stools or 400 - 800<br>gms/24hours | 6 or more loose or watery<br>stools or > 800gms/24<br>hours orrequires IV<br>hydration |
| Systemic Reactions | | | |
| Allergic Reaction | Pruritus without rash | Localized urticaria | Generalized urticaria;<br>angioedema or<br>anaphylaxis |
| All Other conditions | | | |
| Illness or clinical adverse<br>event (as defined according<br>to applicable regulations) | No interference with activity | Some interference with activity not requiring medical intervention | Prevents daily activity and requires medical intervention |

## 12.4.1 Individual Laboratory Measurements and Abnormal Laboratory Values

 Table 7:
 Laboratory Adverse Event Grading Scale

| | Mild<br>(Grade 1) | Moderate<br>(Grade 2) | Severe<br>(Grade 3) |
|---|---|---|---|
| Hematology | | | |
| WBC 10 <sup>3</sup> /UL (Decrease) | 2.50 - 3.50 | 1.50 - 2.49 | < 1.50 |
| WBC 10 <sup>3</sup> /UL (Increase) | 13.01 – 15.00 | 15.01 - 20.00 | > 20.00 |
| HgB g/dL (Decrease) (Female) | 11.0 – 11.49 | 9.5 - 10.9 | < 9.5 |
| HgB g/dL (Decrease) (Male) | 12.0 – 12.5 | 10.0 – 11.9 | < 10.0 |
| Platelets 10 <sup>3</sup> /UL (Decrease) | 120 – 130 | 100 – 119 | < 100 |
| Platelets 10 <sup>3</sup> /UL (Increase) | 416 – 550 | 551-750 | > 750 |
| Chemistry | | | |
| ALT IU/L (Increase) | 47 – 105 | 106 - 175 | > 175 |
| Creatinine mg/dL (Increase) | > ULN – 1.7 | 1.8 - 2.0 | > 2.0 |
| ULN = upper limit of normal range | | | |

## 14.1 Description of Study Subjects

### 14.1.1 Disposition of Subjects

#### **Table 8:** Subject Disposition by Treatment Group

[Implementation Note: Percentages are calculated using the denominators displayed in the header. Listings should be referenced by title for clarity.]

| Subject | Group A:<br>100 μg Sm-p80<br>(unadjuvanted)<br>(N=X) | | 10 μg Sm<br>GL | Group B:<br>10 μg Sm-p80 + 5 μg<br>GLA-SE<br>(N=X) | | Group C:<br>30 μg Sm-p80 + 5 μg<br>GLA-SE<br>(delayed booster)<br>(N=X) | | Group D:<br>30 μg Sm-p80 + 5 μg<br>GLA-SE<br>(N=X) | | Group E:<br>10 μg Sm-p80 + 5 μg<br>GLA-SE<br>(N=X) | | All Subjects<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Disposition | n | % | n | % | n | % | n | % | n | % | n | % |
| Screened | | | | | | | | | | | X | |
| Enrolled/Randomized | X | 100 | X | 100 | х | 100 | X | 100 | X | 100 | X | 100 |
| Received One Scheduled Treatment | X | xx | X | XX | х | xx | X | xx | X | xx | X | XX |
| Received Two Scheduled Treatments | X | xx | X | XX | х | XX | х | xx | х | xx | Х | XX |
| Received All Scheduled Treatments <sup>a</sup> | X | XX | X | xx | х | xx | х | xx | X | xx | X | XX |
| Completed All Safety Blood Draws Groups A, B, D, E [Days 1, 8, 29, 36, 57, 64, 85] Group C [Days 1, 8, 29, 36, 57, 180, 187, 208] | | | | | | | | | | | | |
| Completed All Immunogenicity Blood<br>Draws for Antibody Assays | | | | | | | | | | | | |
| Groups A, B, D, E [Days 1, 8, 29, 36, 57, 64, 85, 181] | | | | | | | | | | | | |
| Group C [Days 1, 8, 29, 36, 57, 180, 187, 208, 304] | | | | | | | | | | | | |
| Completed Follow-up <sup>a</sup> Groups A, B, D, E (Study Day 422) | | | | | | | | | | | | |
| Group C (Study Day 545) | | | | | | | | | | | | |
| Completed Per Protocol <sup>b</sup> | | | | | | | | | | | | |

Note: N = Number of subjects enrolled to the specified treatment group.

<sup>&</sup>lt;sup>a</sup> Refer to Listing 16.2.1 for reasons subjects discontinued or terminated early.

<sup>&</sup>lt;sup>b</sup> Refer to Listing 16.2.3 for reasons subjects are excluded from the Analysis populations .

**Table 9:** Analysis Populations by Treatment Group

| | | Group A:<br>100 µg Sm-p80<br>(unadjuvanted)<br>(N=X) | | Group B:<br>10 μg Sm-p80 +<br>5 μg GLA-SE<br>(N=X) | | Group C:<br>30 µg Sm-p80 + 5<br>µg GLA-SE<br>(delayed booster)<br>(N=X) | | 30 μg Sm-p80 + 5 | | Group E:<br>100 μg Sm-p80 +<br>5 μg GLA-SE<br>(N=X) | | | ıbjects<br>=X) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Analysis Populations | Reason Subjects Excluded | n | % | n | % | n | % | n | % | n | % | % | n |
| Safety Population | Any Reason | X | xx | X | XX | X | XX | X | XX | X | xx | X | XX |
| | Did not receive study product | | | | | | | | | | | | |
| | [Reason 2] | | | | | | | | | | | | |
| nITT Immunogenicity<br>Population | Any Reason | | | | | | | | | | | | |
| | Did not have post-baseline immunogenicity assay | | | | | | | | | | | | |
| | [Reason 2] | | | | | | | | | | | | |
| Per Protocol Population | Any Reason | | | | | | | | | | | | |
| | Did not have post-baseline immunogenicity assay | | | | | | | | | | | | |
| | Found to be ineligible at baseline after the enrollment | | | | | | | | | | | | |
| | [Reason 3] | | | | | | | | | | | | |

Note: N = Number of subjects enrolled to the specified treatment group. Subjects may be counted for more than one reason but will only be counted up to one time for "Any Reason" per population.

**Table 10:** Dates of First Treatment by Treatment Group

| Dates of Dosing | Group A:<br>100 μg Sm-p80<br>(unadjuvanted)<br>(N=X) | Group B:<br>10 μg Sm-p80 + 5<br>μg GLA-SE<br>(N=X) | Group C:<br>30 µg Sm-p80 + 5<br>µg GLA-SE<br>(delayed booster)<br>(N=X) | Group D:<br>30 μg Sm-p80 + 5<br>μg GLA-SE<br>(N=X) | Group E:<br>10 μg Sm-p80 + 5<br>μg GLA-SE<br>(N=X) | All Subjects<br>(N=X) |
|---|---|---|---|---|---|---|
| Total (Entire period of enrollment) | | | | | | |
| DDMMMYYYY-DDMMMYYYY [categorize based on length of enrollment period] | X | x | x | x | x | x |

Note: N = Number of subjects enrolled to the specified treatment group.

Table 11: **Ineligibility Summary of Screen Failures** 

[Implementation Note: Inclusion and exclusion criteria are listed in Section 4.3.]

| Inclusion/Exclusion<br>Category | Inclusion/Exclusion Criterion | n <sup>a</sup> | % b |
|---|---|---|---|
| Inclusion and Exclusion | Number of subjects failing any eligibility criterion | X | 100 |
| Inclusion | Any inclusion criterion | Х | XX |
| | [inclusion criterion 1] | X | XX |
| | [inclusion criterion 2] | X | XX |
| | [inclusion criterion 3] | X | XX |
| Exclusion | Any exclusion criterion | X | XX |
| | [exclusion criterion 1] | X | XX |
| | [exclusion criterion 2] | Х | XX |
| | [exclusion criterion 3] | X | XX |
| Eligible but not | [Reason 1] | Х | XX |
| enrolled | [Reason 2] | X | XX |
| <sup>a</sup> More than one criterion | may be marked per subject. | | |

b Denominator for percentages is the total number of screen failures.

#### 14.1.2 Demographic Data by Study Group

Table 12: Summary of Categorical Demographic and Baseline Characteristics by Treatment Group, All Enrolled Subjects

| | | 100 μg<br>(unadju | Group A:<br>100 μg Sm-p80<br>(unadjuvanted)<br>(N=X) | | Group B:<br>10 µg Sm-p80 + 5<br>µg GLA-SE<br>(N=X) | | Group C:<br>30 µg Sm-p80 + 5<br>µg GLA-SE<br>(delayed booster)<br>(N=X) | | Group D:<br>30 µg Sm-p80 + 5<br>µg GLA-SE<br>(N=X) | | Group E:<br>100 µg Sm-p80 + 5<br>µg GLA-SE<br>(N=X) | | ıbjects<br>=X) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Variable | Characteristic | n | % | n | % | n | % | n | % | n | % | n | % |
| Sex | Male | X | xx | X | xx | Х | XX | X | XX | х | xx | X | XX |
| | Female | | | | | | | | | | | | |
| Ethnicity | Not Hispanic or Latino | X | xx | x | xx | х | xx | X | xx | х | xx | X | xx |
| | Hispanic or Latino | | | | | | | | | | | | |
| | Not Reported | ] | | | | | | | | | | | |
| | Unknown | | | | | | | | | | | | |
| Race | American Indian or Alaska<br>Native | х | xx | X | xx | Х | XX | х | xx | х | xx | X | XX |
| | Asian | | | | | | | | | | | | |
| | Native Hawaiian or Other<br>Pacific Islander | | | | | | | | | | | | |
| | Black or African American | | | | | | | | | | | | |
| | White | | | | | | | | | | | | |
| | Multi-Racial | | | | | | | | | | | | |
| | Unknown | | | | | | | | | | | | |

 Table 13:
 Summary of Continuous Demographic and Baseline Characteristics by Treatment Group

| Variable | Statistic | Group A:<br>100 μg Sm-p80<br>(unadjuvanted)<br>(N=X) | Group B:<br>10 µg Sm-p80 + 5<br>µg GLA-SE<br>(N=X) | Group C:<br>30 µg Sm-p80 + 5<br>µg GLA-SE<br>(delayed booster)<br>(N=X) | Group D:<br>30 µg Sm-p80 + 5<br>µg GLA-SE<br>(N=X) | Group E:<br>100 μg Sm-p80 + 5<br>μg GLA-SE<br>(N=X) | All Subjects<br>(N=X) |
|---|---|---|---|---|---|---|---|
| Age (years) | Mean | xx | XX | XX | XX | XX | XX |
| | Standard Deviation | xx | XX | xx | xx | XX | XX |
| | Median | х | х | X | х | Х | X |
| | Minimum | х | х | X | х | Х | X |
| | Maximum | х | х | X | х | Х | X |
| Height (cm) | Mean | | | | | | |
| | Standard Deviation | | | | | | |
| | Median | | | | | | |
| | Minimum | | | | | | |
| | Maximum | | | | | | |
| Weight (kg) | Mean | | | | | | |
| | Standard Deviation | | | | | | |
| | Median | | | | | | |
| | Minimum | | | | | | |
| | Maximum | | | | | | |
| BMI (kg/m²) | Mean | | | | | | |
| | Standard Deviation | | | | | | |
| | Median | | | | | | |
| | Minimum | | | | | | |
| | Maximum | | | | | | |

#### 14.1.3 Prior and Concurrent Medical Conditions

Table 14: Summary of Subjects with Pre-Existing Medical Conditions by MedDRA System Organ Class and Treatment Group

| Group A:<br>100 μg Sm-p80<br>(unadjuvanted)<br>(N=X) | | Group B:<br>10 μg Sm-p80 + 5<br>μg GLA-SE<br>(N=X) | | Group C:<br>30 µg Sm-p80 + 5<br>µg GLA-SE<br>(delayed booster)<br>(N=X) | | Group D:<br>30 µg Sm-p80 + 5<br>µg GLA-SE<br>(N=X) | | Group E:<br>100 μg Sm-p80 + 5<br>μg GLA-SE<br>(N=X) | | All Subjects<br>(N=X) | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| n | % | n | % | n | % | n | % | n | % | n | % |
| X | xx | х | xx | X | xx | х | xx | х | XX | X | xx |
| | 100 μg<br>(unadju<br>(N= | 100 µg Sm-p80<br>(unadjuvanted)<br>(N=X)<br>n % | 100 μg Sm-p80 (unadjuvanted) μg Gl (N=X) (N=X) n | 100 μg Sm-p80 (unadjuvanted) (N=X) 10 μg Sm-p80 + 5 μg GLA-SE (N=X) n % | Group A: 100 μg Sm-p80 (unadjuvanted) (N=X) π % π % π % π % π 30 μg Sn μg GI μg GLA-SE (N=X) (N=X) σ η π γ η η η η η η η η η η η η η η η η η | Group A: 100 μg Sm-p80 (unadjuvanted) (N=X) Group B: 10 μg Sm-p80 + 5 μg GLA-SE (delayed booster) (N=X) n % n % n % n % | Group A: Group B: 30 μg Sm-p80 + 5 μg GLA-SE (delayed booster) Group Sm-p80 + 5 μg GLA-SE (delayed booster) Group B: (N=X) (N=X) (N=X) (N=X) (N=X) (N=X) (N=X) (N=X) (N=X) (N=X) (N=X) (N=X) (N=X) (N=X) (N=X) (N=X) (N=X) (N=X) (N=X) (N=X) (N=X) (N=X) (N=X) (N=X) (N=X) (N=X) (N=X) (N=X) (N=X) (N=X) (N=X) (N=X) (N=X) (N=X) (N=X) (N=X) (N=X) (N=X) (N=X) (N=X) (N=X) (N=X) (N=X) (N=X) (N=X) (N=X) (N=X) (N=X) (N=X) (N=X) (N=X) (N=X) (N=X) (N=X) (N=X) (N=X) (N=X) (N=X) (N=X) (N=X) (N=X) (N=X) (N=X) (N=X) (N=X) (N=X) (N=X) (N=X) (N=X) (N=X) (N=X) (N=X) (N=X) (N=X) (N=X) (N=X) (N=X) (N=X) (N=X) </td <td>Group A: Group B: 30 μg Sm-p80 + 5 μg GLA-SE (delayed booster) Group D: 30 μg Sm-p80 + 5 μg GLA-SE (delayed booster) Group D: 30 μg Sm-p80 + 5 μg GLA-SE (delayed booster) μg GLA-SE (N=X) μg GLA-SE (N=X) μg GLA-SE (N=X) κα γω κα γω κα γω κα γω κα γω κα γω κα γω κα γω κα γω κα γω κα γω κα γω κα γω κα γω κα γω κα γω κα γω κα γω κα γω κα γω κα γω κα γω κα γω κα γω κα γω κα γω κα γω κα γω κα γω κα γω κα γω κα γω κα γω κα γω κα γω κα γω κα γω κα γω κα γω κα γω κα γω κα γω κα γω κα γω κα γω κα γω κα γω κα γω κα γω κα γω κα γω κα γω κα γω κα γω κα γω κα γω κα γω κα γω κα γω κα γω κα γω κα γω κα γω κα γω κα γω κα γω κα γω κα γω κα γω κα γω κα γω</td> <td>Group A: Group B: 30 μg Sm-p80 + 5 μg GLA-SE (next) Group D: Group D: Group D: Group D: Group D: Group D: Group D: Group D: Group D: Group D: Group D: Group D: Group D: Group D: Group D: Group D: Group D: Group D: Group D: Group D: Group D: Group D: Group D: Group D: Group D: Group D: Group D: Group D: Group D: Group D: Group D: Group D: Group D: Group D: Group D: Group D: Group D: Group D: Group D: Group D: Group D: Group D: Group D: Group D: Group D: Group D: Group D: Group D: Group D: Group D: Group D: Group D: Group D: Group D: Group D: Group D: Group D: Group D: Group D: Group D: Group D: Group D: Group D: Group D: Group D: Group D: Group D: Group D: Group D: Group D: Group D: Group D: Group D: Group D:</td> <td> Group A: 100 μg Sm-p80 (unadjuvanted) (N=X) The state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the stat</td> <td> Group A: 100 μg Sm-p80 (unadjuvanted) (N=X) The standard of the standard of the standard of the standard of the standard of the standard of the standard of the standard of the standard of the standard of the standard of the standard of the standard of the standard of the standard of the standard of the standard of the standard of the standard of the standard of the standard of the standard of the standard of the standard of the standard of the standard of the standard of the standard of the standard of the standard of the standard of the standard of the standard of the standard of the standard of the standard of the standard of the standard of the standard of the standard of the standard of the standard of the standard of the standard of the standard of the standard of the standard of the standard of the standard of the standard of the standard of the standard of the standard of the standard of the standard of the standard of the standard of the standard of the standard of the standard of the standard of the standard of the standard of the standard of the standard of the standard of the standard of the standard of the standard of the standard of the standard of the standard of the standard of the standard of the standard of the standard of the standard of the standard of the standard of the standard of the standard of the standard of the standard of the standard of the standard of the standard of the standard of the standard of the standard of the standard of the standard of the standard of the standard of the standard of the standard of the standard of the standard of the standard of the standard of the standard of the standard of the standard of the standard of the standard of the standard of the standard of the standard of the standard of the standard of the standard of the standard of the standard of the standard of the standard of the standard of the standard of the standard of the standard of the standard of the standard of the standard of the standard of the standard of the standard of the standard</td> | Group A: Group B: 30 μg Sm-p80 + 5 μg GLA-SE (delayed booster) Group D: 30 μg Sm-p80 + 5 μg GLA-SE (delayed booster) Group D: 30 μg Sm-p80 + 5 μg GLA-SE (delayed booster) μg GLA-SE (N=X) μg GLA-SE (N=X) μg GLA-SE (N=X) κα γω κα γω | Group A: Group B: 30 μg Sm-p80 + 5 μg GLA-SE (next) Group D: Group D: | Group A: 100 μg Sm-p80 (unadjuvanted) (N=X) The state of the stat | Group A: 100 μg Sm-p80 (unadjuvanted) (N=X) The standard of the standard |

Note: N = Number of subjects in the Safety Population; n = Number of subjects reporting medical history within the specified SOC. A subject is only counted once per SOC.

## 14.2 Immunogenicity Data

Table 15: Anti-Sm-p80 ELISA Total IgG Geometric Mean Titers (GMT) Results with 95% Confidence Intervals by Time Point and Treatment Group, mITT Immunogenicity Population

| Time Point | Statistic | Group A:<br>100 μg Sm-p80<br>(unadjuvanted)<br>(N=X) | Group B:<br>10 μg Sm-p80 + 5<br>μg GLA-SE<br>(N=X) | Group C:<br>30 μg Sm-p80 + 5 μg GLA-SE<br>(delayed booster)<br>(N=X) | Group D:<br>30 μg Sm-p80 + 5 μg GLA-<br>SE<br>(N=X) | Group E:<br>100 μg Sm-p80 + 5<br>μg GLA-SE<br>(N=X) |
|---|---|---|---|---|---|---|
| Study Day 1 | n | | | | | |
| (Pre-Dose 1) | | | | | | |
| (Baseline) | | X | Х | X | X | Х |
| | GMT (95% CI) | x.x(x.x, x.x) | x.x (x.x, x.x) | x.x(x.x, x.x) | x.x (x.x, x.x) | x.x (x.x, x.x) |
| | Mean | x.x | x.x | X.X | X.X | x.x |
| | Std. Dev. | x.x | x.x | X.X | X.X | x.x |
| | Median | X.X | x.x | X.X | X.X | x.x |
| | (Minimum,<br>Maximum) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| Study Day 8<br>(7 Days Post Dose 1) | n | | | | | |
| | GMT (95% CI) | | | | | |
| | Mean | | | | | |
| | Std. Dev. | | | | | |
| | Median | | | | | |
| | (Minimum,<br>Maximum) | | | | | |
| Study Day 29 | n | | | | | |
| (28 Days Post Dose 1; Pre-Dose 2) | | | | | | |
| | GMT (95% CI) | | | | | |
| | Mean | | | | | |

Table 15: Anti-Sm-p80 ELISA Total IgG Geometric Mean Titers (GMT) Results with 95% Confidence Intervals by Time Point and Treatment Group, mITT Immunogenicity Population (Continued)

| Time Point | Statistic | Group A:<br>100 μg Sm-p80<br>(unadjuvanted)<br>(N=X) | Group B:<br>10 μg Sm-p80 + 5<br>μg GLA-SE<br>(N=X) | Group C:<br>30 μg Sm-p80 + 5 μg GLA-SE<br>(delayed booster)<br>(N=X) | Group D:<br>30 μg Sm-p80 + 5 μg GLA-<br>SE<br>(N=X) | Group E:<br>100 μg Sm-p80 + 5<br>μg GLA-SE<br>(N=X) |
|---|---|---|---|---|---|---|
| | Std. Dev. | | | | | |
| | Median | | | | | |
| | (Minimum,<br>Maximum) | | | | | |
| Study Day 36 | n | | | | | |
| (7 Days Post Dose 2) | | | | | | |
| | GMT (95% CI) | | | | | |
| | Mean | | | | | |
| | Std. Dev. | | | | | |
| | Median | | | | | |
| | (Minimum,<br>Maximum) | | | | | |
| Study Day 57 | n | | | | | |
| (Groups A, B, D, E: 28 Days Post Dose 2; Pre-Dose 3) | | | | | | |
| (Group C: 28 Days Post Dose 2) | | | | | | |
| | GMT (95% CI) | | | | | |
| | Mean | | | | | |
| | Std. Dev. | | | | | |
| | Median | | | | | |
| | (Minimum,<br>Maximum) | | | | | |
| Study Day 64 | n | | | | | |
| (Groups A, B, D, E: 7 Days Post Dose 3) | | | | | N/A | |

Table 15: Anti-Sm-p80 ELISA Total IgG Geometric Mean Titers (GMT) Results with 95% Confidence Intervals by Time Point and Treatment Group, mITT Immunogenicity Population (Continued)

| Time Point | Statistic | Group A:<br>100 µg Sm-p80<br>(unadjuvanted)<br>(N=X) | Group B:<br>10 μg Sm-p80 + 5<br>μg GLA-SE<br>(N=X) | Group C:<br>30 µg Sm-p80 + 5 µg GLA-SE<br>(delayed booster)<br>(N=X) | Group D:<br>30 μg Sm-p80 + 5 μg GLA-<br>SE<br>(N=X) | Group E:<br>100 μg Sm-p80 + 5<br>μg GLA-SE<br>(N=X) |
|---|---|---|---|---|---|---|
| | GMT (95% | | | N/A | | |
| | CI) | | | | | |
| | Mean | | | N/A | | |
| | Std. Dev. | | | N/A | | |
| | Median | | | N/A | | |
| | (Minimum,<br>Maximum) | | | N/A | | |
| Study Day 85 | n | | | N/A | | |
| (Groups A, B, D, E: 28 Days<br>Post Dose 3) | | | | | | |
| , | GMT (95%<br>CI) | | | N/A | | |
| | Mean | | | N/A | | |
| | Std. Dev. | | | N/A | | |
| | Median | | | N/A | | |
| | (Minimum,<br>Maximum) | | | N/A | | |
| Study Day 180<br>(Group C: Pre-Dose 3) | n | N/A | N/A | | N/A | N/A |
| | GMT (95%<br>CI) | N/A | N/A | | N/A | N/A |
| | Mean | N/A | N/A | | N/A | N/A |
| | Std. Dev. | N/A | N/A | | N/A | N/A |
| | Median | N/A | N/A | | N/A | N/A |
| | (Minimum,<br>Maximum) | N/A | N/A | | N/A | N/A |

Table 15: Anti-Sm-p80 ELISA Total IgG Geometric Mean Titers (GMT) Results with 95% Confidence Intervals by Time Point and Treatment Group, mITT Immunogenicity Population (Continued)

| Time Point | Statistic | Group A:<br>100 μg Sm-p80<br>(unadjuvanted)<br>(N=X) | Group B:<br>10 μg Sm-p80 + 5<br>μg GLA-SE<br>(N=X) | Group C:<br>30 μg Sm-p80 + 5 μg GLA-SE<br>(delayed booster)<br>(N=X) | Group D:<br>30 μg Sm-p80 + 5 μg GLA-<br>SE<br>(N=X) | Group E:<br>100 μg Sm-p80 + 5<br>μg GLA-SE<br>(N=X) |
|---|---|---|---|---|---|---|
| Study Day 187 | n | N/A | N/A | | N/A | N/A |
| (Group C: 7 Days Post Dose 3) | | | | | | |
| | GMT (95%<br>CI) | N/A | N/A | | N/A | N/A |
| | Mean | N/A | N/A | | N/A | N/A |
| | Std. Dev. | N/A | N/A | | N/A | N/A |
| | Median | N/A | N/A | | N/A | N/A |
| | (Minimum,<br>Maximum) | N/A | N/A | | N/A | N/A |
| Study Day 181<br>(Groups A, B, D, E: 124 Days<br>Post Dose 3) | n | | | N/A | | |
| , | GMT (95%<br>CI) | | | N/A | | |
| | Mean | | | N/A | | |
| | Std. Dev. | | | N/A | | |
| | Median | | | N/A | | |
| | (Minimum,<br>Maximum) | | | N/A | | |
| Study Day 208<br>(Group C: 28 Days Post Dose<br>3) | n | N/A | N/A | | N/A | N/A |
| | GMT (95%<br>CI) | N/A | N/A | | N/A | N/A |
| | Mean | N/A | N/A | | N/A | N/A |

Table 15: Anti-Sm-p80 ELISA Total IgG Geometric Mean Titers (GMT) Results with 95% Confidence Intervals by Time Point and Treatment Group, mITT Immunogenicity Population (Continued)

| Time Point | Statistic | Group A:<br>100 µg Sm-p80<br>(unadjuvanted)<br>(N=X) | Group B:<br>10 μg Sm-p80 + 5<br>μg GLA-SE<br>(N=X) | Group C:<br>30 μg Sm-p80 + 5 μg GLA-SE<br>(delayed booster)<br>(N=X) | Group D:<br>30 μg Sm-p80 + 5 μg GLA-<br>SE<br>(N=X) | Group E:<br>100 μg Sm-p80 + 5<br>μg GLA-SE<br>(N=X) |
|---|---|---|---|---|---|---|
| | Std. Dev. | N/A | N/A | | N/A | N/A |
| | Median | N/A | N/A | | N/A | N/A |
| | (Minimum,<br>Maximum) | N/A | N/A | | N/A | N/A |
| Study Day 304<br>(Group C: 124 Days Post Dose<br>3) | n | N/A | N/A | | N/A | N/A |
| | GMT (95%<br>CI) | N/A | N/A | | N/A | N/A |
| | Mean | N/A | N/A | | N/A | N/A |
| | Std. Dev. | N/A | N/A | | N/A | N/A |
| | Median | N/A | N/A | | N/A | N/A |
| Note: N = Number of subjects in the m | (Minimum,<br>Maximum) | N/A | N/A | | N/A | N/A |
#### Pseudo Code:

```
/*Geometric Mean Titers*/
data dsn2;
set dsn1;
     log aval = log(aval);
proc means data=dsn2 n mean clm noprint;
by stdy trta;
var log aval;
output out= gmt0(drop=_type__freq_)
            n=n
            mean= mean
            std= sd
            median= med
            max= max
            min= min
           lclm=lclm
            uclm=uclm;
data qmt;
 set gmt0;
                                                                         /*geometric mean titer*/
     gmt = put(exp(mean), 8.1);
     gmt l = put(exp(lclm), 8.1);
                                                                         /*lower bound*/
                                                                         /*upper bound*/
      gmt u = put(exp(uclm), 8.1);
      gmt ci = strip(gmt)||' ('||strip(gmt 1)||', '||strip(gmt u)||')'; /*GMT(95% CI)*/
      gmt_mm = '('||strip(min)||', '||strip(max)||')';
                                                                        /*(Min, Max)*/
run;
```

Table 16: Anti-Sm-p80 ELISA Total IgG Geometric Mean Fold Rise (GMFR) and Seroconversion Results by Time Point and Treatment Group, mITT Immunogenicity Population

| | | | | Group C: | | |
|---|---|---|---|---|---|---|
| | | Group A:<br>100 μg Sm-p80<br>(unadjuvanted) | Group B:<br>10 μg Sm-p80 + 5<br>μg GLA-SE | 30 µg Sm-p80 + 5<br>µg GLA-SE<br>(delayed booster) | Group D:<br>30 µg Sm-p80 + 5<br>µg GLA-SE | Group E:<br>100 µg Sm-p80 + 5<br>µg GLA-SE |
| Time Point | Statistic | (N=X) | (N=X) | (N=X) | (N=X) | (N=X) |
| Study Day 8<br>(7 Days Post Dose 1) | n | X | X | X | X | X |
| | GMFR <sup>a</sup> (95% CI) | x.x(x.x, x.x) | x.x (x.x, x.x) | x.x (x.x, x.x) | x.x (x.x, x.x) | x.x (x.x, x.x) |
| | Number (%) of Responders <sup>b</sup> | x (xx) | x (xx) | x (xx) | x (xx) | x (xx) |
| | 95% CI | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x |
| Study Day 29<br>(28 Days Post Dose 1; Pre-Dose 2) | n | Х | X | x | X | х |
| | GMFR <sup>a</sup> (95% CI) | x.x (x.x, x.x) | x.x (x.x, x.x) | x.x (x.x, x.x) | x.x (x.x, x.x) | x.x (x.x, x.x) |
| | Number (%) of Responders <sup>b</sup> | x (xx) | x (xx) | x (xx) | x (xx) | x (xx) |
| | 95% CI | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x |
| Study Day 36<br>(7 Days Post Dose 2) | n | X | X | х | х | X |
| | GMFR <sup>a</sup> (95% CI) | x.x (x.x, x.x) | x.x (x.x, x.x) | x.x (x.x, x.x) | x.x (x.x, x.x) | x.x (x.x, x.x) |
| | Number (%) of Responders <sup>b</sup> | x (xx) | x (xx) | x (xx) | x (xx) | x (xx) |
| | 95% CI | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x |
| Study Day 57<br>(Groups A, B, D, E: 28 Days Post Dose 2; Pre-<br>Dose 3) | n | Х | X | X | X | х |
| (Group C: 28 Days Post Dose 2) | | | | | | |
| | GMFR <sup>a</sup> (95% CI) | x.x (x.x, x.x) | x.x (x.x, x.x) | x.x (x.x, x.x) | x.x (x.x, x.x) | x.x (x.x, x.x) |
| | Number (%) of Responders <sup>b</sup> | x (xx) | x (xx) | x (xx) | x (xx) | x (xx) |
| | 95% CI | X.X, X.X | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x |

Table 16: Anti-Sm-p80 ELISA Total IgG Geometric Mean Fold Rise (GMFR) and Seroconversion Results by Time Point and Treatment Group, mITT Immunogenicity Population (Continued)

| | | Group A: | Group B: | Group C:<br>30 µg Sm-p80 + 5 | Group D: | Group E: |
|---|---|---|---|---|---|---|
| | | 100 μg Sm-p80<br>(unadjuvanted) | 10 μg Sm-p80 + 5<br>μg GLA-SE | μg GLA-SE<br>(delayed booster) | 30 μg Sm-p80 + 5<br>μg GLA-SE | 100 μg Sm-p80 + 5<br>μg GLA-SE |
| Time Point | Statistic | (N=X) | (N=X) | (N=X) | (N=X) | (N=X) |
| Study Day 64<br>(Groups A, B, D, E: 7 Days Post Dose 3) | n | X | X | N/A | X | X |
| | GMFR <sup>a</sup> (95% CI) | x.x(x.x, x.x) | x.x(x.x, x.x) | N/A | x.x(x.x, x.x) | x.x(x.x, x.x) |
| | Number (%) of Responders <sup>b</sup> | x (xx) | x (xx) | N/A | x (xx) | x (xx) |
| | 95% CI | x.x, x.x | x.x, x.x | N/A | x.x, x.x | x.x, x.x |
| Study Day 85<br>(Groups A, B, D, E: 28 Days Post Dose 3) | n | X | х | N/A | х | X |
| | GMFR <sup>a</sup> (95% CI) | x.x (x.x, x.x) | x.x (x.x, x.x) | N/A | x.x (x.x, x.x) | x.x (x.x, x.x) |
| | Number (%) of Responders <sup>b</sup> | x (xx) | x (xx) | N/A | x (xx) | x (xx) |
| | 95% CI | x.x, x.x | x.x, x.x | N/A | x.x, x.x | x.x, x.x |
| Study Day 180<br>(Group C: Pre-Dose 3) | n | N/A | N/A | х | N/A | N/A |
| | GMFR <sup>a</sup> (95% CI) | N/A | N/A | x.x (x.x, x.x) | N/A | N/A |
| | Number (%) of Responders <sup>b</sup> | N/A | N/A | x (xx) | N/A | N/A |
| | 95% CI | N/A | N/A | x.x, x.x | N/A | N/A |
| Study Day 187<br>(Group C: 7 Days Post Dose 3) | n | N/A | N/A | x | N/A | N/A |
| | GMFR <sup>a</sup> (95% CI) | N/A | N/A | x.x (x.x, x.x) | N/A | N/A |
| | Number (%) of Responders <sup>b</sup> | N/A | N/A | x (xx) | N/A | N/A |
| | 95% CI | N/A | N/A | x.x, x.x | N/A | N/A |
| Study Day 181<br>(Groups A, B, D, E: 124 Days Post Dose 3) | n | X | Х | N/A | х | X |

Table 16: Anti-Sm-p80 ELISA Total IgG Geometric Mean Fold Rise (GMFR) and Seroconversion Results by Time Point and Treatment Group, mITT Immunogenicity Population (Continued)

| Time Point | Statistic | Group A:<br>100 μg Sm-p80<br>(unadjuvanted)<br>(N=X) | Group B:<br>10 µg Sm-p80 + 5<br>µg GLA-SE<br>(N=X) | Group C:<br>30 µg Sm-p80 + 5<br>µg GLA-SE<br>(delayed booster)<br>(N=X) | Group D:<br>30 μg Sm-p80 + 5<br>μg GLA-SE<br>(N=X) | Group E:<br>100 μg Sm-p80 + 5<br>μg GLA-SE<br>(N=X) |
|---|---|---|---|---|---|---|
| | GMFR <sup>a</sup> (95% CI) | x.x (x.x, x.x) | x.x (x.x, x.x) | N/A | x.x (x.x, x.x) | x.x (x.x, x.x) |
| | Number (%) of Responders <sup>b</sup> | x (xx) | x (xx) | N/A | x (xx) | x (xx) |
| | 95% CI | x.x, x.x | x.x, x.x | N/A | x.x, x.x | x.x, x.x |
| Study Day 208<br>(Group C: 28 Days Post Dose 3) | n | N/A | N/A | X | N/A | N/A |
| | GMFR <sup>a</sup> (95% CI) | N/A | N/A | x.x (x.x, x.x) | N/A | N/A |
| | Number (%) of Responders <sup>b</sup> | N/A | N/A | x (xx) | N/A | N/A |
| | 95% CI | N/A | N/A | x.x, x.x | N/A | N/A |
| Study Day 304<br>(Group C: 124 Days Post Dose 3) | n | N/A | N/A | X | N/A | N/A |
| | GMFR <sup>a</sup> (95% CI) | N/A | N/A | x.x (x.x, x.x) | N/A | N/A |
| | Number (%) of Responders <sup>b</sup> | N/A | N/A | x (xx) | N/A | N/A |
| | 95% CI | N/A | N/A | x.x, x.x | N/A | N/A |

Note: N = Number of subjects in the mITT Immunogenicity Population; n = Number of subjects with results at the given timepoint.

<sup>&</sup>lt;sup>a</sup> GMFR represents the geometric mean fold rise in antibody compared to pre-dose 1.

<sup>&</sup>lt;sup>b</sup> Number of responders represents the percentage of subjects with at least a 4-Fold Rise in antibody compared to Day 1, pre-dose 1.

#### Pseudo Code:

```
/*Geometric Mean Fold Rise*/
data dsn2;
 set dsn1;
      log fold = log(mchg);
proc means data= dsn2 n mean clm noprint;
 by stdy trta;
var log fold;
 output out= gmfr0(drop= type freq )
            n= n2
            mean= mean
            lclm= lclm
            uclm= uclm;
data qmfr;
 set gmfr0;
      gmfr = put(exp(mean),8.1);
                                                                              /*geometric mean fold rise*/
                                                                              /*lower bound*/
      gmfr l = put(exp(lclm), 8.1);
      gmfr u = put(exp(uclm), 8.1);
                                                                              /*upper bound*/
      gmfr_ci = strip(gmfr)||' ('||strip(gmfr_l)||', '||strip(gmfr_u)||')'; /*GMFR(95%CI)*/
run:
/*Seroresponders*/
proc freq data= dsn1 noprint;
 table stdy*trta / out= totcnt(keep= stdy trta count rename= count=totcnt);
proc freq data= dsn1 noprint;
 where crit1fl ^= ''; /*seroconversion flag = Y*/
  table stdy*trta / out= cnt(keep= stdy trta count);
```

#### Pseudo Code (continued):

```
data cntp;
merge cnt totcnt;
by stdy trta;
     if count=. then count=0;
     scn = put(count/totcnt*100, 5.1);
data cntci;
set cntp;
     sym = 1; /*seroconversion*/
output;
     sym = 0;  /*no seroconversion*/
     count = totcnt - count;
output;
proc freq data= cntci;
by stdy trta;
tables sym / nocum norow binomial(cl= wilson);
weight count; /*zeros: for CI of zero*/
 *exact binomial;
ods output binomial= binany (keep=stdy trta name1 nvalue1 where=(name1 in ('XL_BIN','XU_BIN')));
run;
```

Table 17: Comparison of Anti-Sm-p80 ELISA Total IgG Seroresponse Rates between Group A and Each Treatment Group 28-Days Post Dose – mITT Immunogenicity Population

| Analysis Population | Dose | Statistic | Group A:<br>100 μg Sm-p80<br>(unadjuvanted)<br>(N=X) | Group B:<br>10 μg Sm-p80 + 5<br>μg GLA-SE<br>(N=X) | Group C:<br>30 µg Sm-p80 + 5<br>µg GLA-SE<br>(delayed booster)<br>(N=X) | Group D:<br>30 µg Sm-p80 + 5<br>µg GLA-SE<br>(N=X) | Group E:<br>100 µg Sm-p80 +<br>5 µg GLA-SE<br>(N=X) |
|---|---|---|---|---|---|---|---|
| mITT Immunogenicity Population | 1 | Fraction Responders, na | x | X | X | X | X |
| | | Responders, Rate | XX% | xx% | XX% | XX% | XX% |
| | | 95% CI <sup>b</sup> | x.xxx, x.xxx | x.xxx, x.xxx | x.xxx, x.xxx | x.xxx, x.xxx | x.xxx, x.xxx |
| | | Difference in Proportion | | x.xxx | x.xxx | X.XX | x.xxxx |
| | | p-value <sup>c</sup> | | 0.xxxx | 0.xxxx | 0.xxxx | 0.xxxx |
| | 2 | | | | | | |
| | 3 | | | | | | |
| Per Protocol Population | | | | | | | |

<sup>&</sup>lt;sup>a</sup> Responder is defined as subjects with at least a 4-fold rise in antibody compared to pre-dose 1.

<sup>&</sup>lt;sup>b</sup> 95% confidence intervals are from the Wilson score method without continuity correction.

<sup>°</sup> P-values were calculated using Fisher's Exact Test.

# 14.3 Safety Data

## 14.3.1 Displays of Adverse Events

 Table 18:
 Overall Summary of Adverse Events

| | 100 μg<br>(unadji | up A:<br>Sm-p80<br>uvanted)<br>= X) | 10 μg S<br>5 μg G | up B:<br>5m-p80 +<br>GLA-SE<br>= X) | 30 μg Si<br>5 μg G<br>(dela<br>boos | up C:<br>m-p80 +<br>LA-SE<br>ayed<br>ster)<br>= X) | 30 μg S<br>5 μg G | up D:<br>m-p80 +<br>LA-SE<br>= X) | 100 μg<br>+ 5 μg ( | up E:<br>Sm-p80<br>GLA-SE<br>= X) | | ıbjects<br>= X) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Subjects <sup>a</sup> with | n | % | n | % | n | % | n | % | n | % | n | % |
| At least one local solicited adverse event | X | X | X | X | X | X | X | X | X | X | X | X |
| At least one systemic solicited adverse event | X | Х | Х | Х | X | X | X | X | X | х | X | X |
| At least one unsolicited adverse event | X | X | X | X | X | X | X | X | X | X | X | X |
| At least one related unsolicited adverse event | X | X | X | X | X | X | X | X | X | X | X | X |
| Mild (Grade 1) | X | X | X | X | X | X | X | X | X | X | X | X |
| Moderate (Grade 2) | X | X | X | X | X | X | X | X | X | X | X | X |
| Severe (Grade 3) | X | X | X | X | X | X | X | X | X | X | X | X |
| Not yet assessed | | | | | | | | | | | | |
| At least one severe (Grade 3) unsolicited adverse event | X | X | X | X | X | X | X | X | X | X | X | X |
| Related | X | х | Х | Х | X | х | Х | X | X | Х | X | X |
| Unrelated | Х | х | Х | Х | X | Х | X | X | X | Х | Х | Х |
| At least one serious adverse event <sup>b</sup> | X | Х | х | X | X | X | X | X | X | Х | Х | X |
| At least one related, serious adverse event | X | х | х | Х | X | х | х | X | х | Х | X | X |
| At least one adverse event leading to early termination <sup>c</sup> | Х | X | X | X | X | X | X | X | Х | X | X | X |
| At least one medically attended adverse event | X | X | X | X | X | X | X | X | X | х | X | X |

**Overall Summary of Adverse Events** (Continued) **Table 18:** 

| | 100 μg<br>(unadju | up A:<br>Sm-p80<br>ivanted)<br>= X) | 10 μg Si<br>5 μg G | up B:<br>m-p80 +<br>LA-SE<br>= X) | 30 μg Si<br>5 μg G<br>(dela<br>boos | - | 30 μg Si<br>5 μg G | up D:<br>m-p80 +<br>LA-SE<br>= X) | 100 μg<br>+ 5 μg ( | ıp E:<br>Sm-p80<br>GLA-SE<br>= X) | | bjects<br>= X) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Subjects <sup>a</sup> with | n | % | n | % | n | % | n | % | n | % | n | % |
| At least one new onset chronic medical condition | х | y y | | X | х | X | X | Х | X | X | X | Х |
| At least one potentially immune mediated medical condition | х | X | X | X | Х | X | X | Х | X | X | X | X |

Note: N = Number of subjects in the Safety Population

a Subjects are counted once for each category regardless of the number of events.

b A listing of Serious Adverse Events is included in the Serious Adverse Event Listing.

<sup>&</sup>lt;sup>c</sup> As reported on the Adverse Event eCRF.

Table 19: Adverse Events Occurring in 5% of Subjects in Any Treatment MedDRA System Organ Class and Preferred Term, and Treatment Group - Safety Population

| Preferred Term | MedDRA<br>System Organ<br>Class | 100 | Group A<br>0 μg Sm-<br>adjuvan<br>(N=X) | -p80<br>ited) | 10 μg | Group B<br>Sm-p80<br>GLA-SF<br>(N=X) | + 5 μg | 30 μg | Group C<br>Sm-p80<br>GLA-SF<br>ayed boo<br>(N=X) | + 5 μg | 30 μg | Group D<br>Sm-p80<br>GLA-SH<br>(N=X) | + 5 μg | 100 μg | Group I<br>g Sm-p80<br>GLA-SI<br>(N=X) | ) + 5 μg<br>Ε | A | ll Subje<br>(N=X) | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | n | % | Events | n | n % | | n | % | Events | n | % | Events | n | % | Events | n | % | Events |
| Serious Adverse Events | | | • | ' | | | | | | | | | | | • | ' | | | |
| All | All | X | X | X | X | х | X | X | х | X | X | х | X | X | х | х | X | X | X |
| PT1 | SOC1 | X | X | х | X | х | х | X | х | х | X | х | х | X | х | х | X | х | X |
| Etc. | Etc. | | | | | | | | | | | | | | | | | | |
| Other (Non-serious) Adve | rse Events | | | | | | | | | | | | | | • | | | | |
| All | All | X | X | X | X | х | X | X | х | X | X | х | X | X | х | х | X | X | X |
| PT1 | SOC1 | X | X | х | х | х | х | X | х | х | X | х | х | X | х | х | X | х | х |
| Etc. | Etc. | | | | | | | | | | | | | | | | | | |

#### 14.3.1.1 Solicited Adverse Events

# Table 20: Number and Percentage of Subjects Experiencing Solicited Events with 95% Confidence Intervals by Symptom and Treatment Group – Post Dose 1

[Implementation Note: Confidence intervals will be computed via the Wilson Score method.]

| | 100 | Group A<br>0 μg Sm-<br>nadjuvan<br>(N=X) | -p80 | 10 μ <u>գ</u> | Group B<br>g Sm-p80<br>GLA-SF<br>(N=X) | + 5 μg | 30 µg | Group C<br>Sm-p80<br>GLA-SE<br>ayed boo<br>(N=X) | + 5 μg | 30 µg | Group D<br>g Sm-p80<br>GLA-SI<br>layed boo<br>(N=X) | + 5 μg | | Group E<br>g Sm-p80<br>GLA-SE<br>(N=X) | ) + 5 μg<br>E |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Symptom | n | n % CI <sup>a</sup> x xx x.x, x.x | | n | % | 95%<br>CI <sup>a</sup> | n | % | 95%<br>CI <sup>a</sup> | n | % | 95%<br>CI <sup>a</sup> | n | % | 95%<br>CI <sup>a</sup> |
| Any Symptom | X | | | X | XX | x.x, x.x | X | XX | x.x, x.x | X | XX | x.x, x.x | X | XX | X.X, X.X |
| Any Systemic Symptom | | | | | | | | | | | | | | | |
| [Systemic Symptom 1] | | | | | | | | | | | | | | | |
| [Systemic Symptom 2] | | | | | | | | | | | | | | | |
| Any Injection Site Symptom | | | | | | | | | | | | | | | |
| [Injection Site Symptom 1] | | | | | | | | | | | | | | | |
| [Injection Site Symptom 2] | | | | 1.1 | | | 1 0 | | | • • | | | | | |

Note: N = Number of subjects in the Safety Population who received the specified dose; n = number of subjects reporting the specified event.

<sup>a</sup>95% confidence intervals are from the Wilson score method without continuity correction.

#### Tables with similar format to Table 20:

- Table 21: Number and Percentage of Subjects Experiencing Solicited Events with 95% Confidence Intervals by Symptom and Treatment Group Post Dose 2
- Table 22: Number and Percentage of Subjects Experiencing Solicited Events with 95% Confidence Intervals by Symptom and Treatment Group Post Dose 3
- Table 23: Number and Percentage of Subjects Experiencing Solicited Events with 95% Confidence Intervals by Symptom and Treatment Group Post Any Dose

## Table 24: Comparison of the Proportion of Subjects Experiencing Solicited Events by Treatment Group

[Implementation Note: Confidence intervals will be computed via the Wilson Score method.]

| Symptom | Statistic | Group A:<br>100 μg Sm-p80<br>(unadjuvanted)<br>(N=X) | Group B:<br>10 μg Sm-p80 + 5 μg<br>GLA-SE<br>(N=X) | Group C:<br>30 μg Sm-p80 + 5 μg<br>GLA-SE<br>(delayed booster)<br>(N=X) | Group D:<br>30 μg Sm-p80 + 5 μg<br>GLA-SE<br>(N=X) | Group E:<br>100 μg Sm-p80 + 5<br>μg GLA-SE<br>(N=X) |
|---|---|---|---|---|---|---|
| Any Symptom | Proportion | X.XX | x.xx | X.XX | X.XX | X.XX |
| | 95% CI <sup>a</sup> (for proportion) | x.xx, x.xx | x.xx, x.xx | x.xx, x.xx | x.xx, x.xx | x.xx, x.xx |
| | Difference | | X.XX | X.XX | X.XX | X.XX |
| | 95% CI <sup>a</sup> (for difference) | | x.xx, x.xx | x.xx, x.xx | x.xx, x.xx | x.xx, x.xx |
| Any Systemic Symptom | Proportion | | | | | |
| | 95% CI <sup>a</sup> (for proportion) | | | | | |
| | Difference | | | | | |
| | 95% CI <sup>a</sup> (for difference) | | | | | |
| [Systemic Symptom 1] | | | | | | |
| Any Injection Site<br>Symptom | | | | | | |
| [Injection Site Symptom 1] | | | | | | |

Note: N = Number of subjects in the Safety Population who received at least one dose.

<sup>a</sup>95% confidence intervals are from the Wilson score method without continuity correction.

Table 25: Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Maximum Severity, and Treatment Group – Post Dose 1

[Implementation Note: Rows for Mild, Moderate, and Severe will only be shown if there is at least one non-zero count in that row. Confidence intervals will be computed via the Wilson Score method.]

| | | 100 | Group A<br>D μg Sm-<br>ladjuvar<br>(N=X) | -p80<br>ited) | 10 μg | Group F<br>Sm-p80<br>GLA-Sl<br>(N=X) | + <b>5 μg</b><br>Ε | 30 μg | Group (<br>Sm-p80<br>GLA-Sl<br>ayed boo<br>(N=X) | +5 μg<br>E<br>oster) | 30 μg | Group I<br>Sm-p80<br>GLA-SI<br>(N=X) | + <b>5 μg</b><br>Ε | 100 μg | Group F<br>3 Sm-p80<br>GLA-Sl<br>(N=X) | ) + 5 μg<br>Ξ | A | ll Subje<br>(N = X) | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Symptom | Severity | n | % | 95%<br>CI <sup>a</sup> | n | % | 95%<br>CI <sup>a</sup> | n | % | 95%<br>CI <sup>a</sup> | n | % | 95%<br>CI <sup>a</sup> | n | % | 95%<br>CI <sup>a</sup> | n | % | 95%<br>CI <sup>a</sup> |
| Any Symptom | None | X | xx | x.x,<br>x.x | х | XX | X.X,<br>X.X | х | XX | X.X,<br>X.X | х | xx | x.x,<br>x.x | х | XX | x.x,<br>x.x | X | XX | X.X,<br>X.X |
| | Mild | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | |
| Systemic Symptoms | | | | | | | | | | | | | | | • | | | | |
| Any Systemic<br>Symptom | None | Х | XX | x.x,<br>x.x | х | XX | x.x,<br>x.x | х | XX | x.x,<br>x.x | Х | XX | X.X,<br>X.X | Х | XX | X.X,<br>X.X | Х | XX | x.x,<br>x.x |
| | Mild | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | |
| [Systemic Symptom 1] | None | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | |
| [Systemic Symptom 2] | None | | | | | | | | | | | | | | | | | | |

Table 25: Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Maximum Severity and Treatment Group – Post Dose 1 (Continued)

| | | 100 | Group A<br>) μg Sma<br>adjuvar<br>(N=X) | -p80<br>ited) | 10 µg | Group I<br>Sm-p80<br>GLA-S<br>(N=X) | + 5 μg<br>Ε | 30 µg | Group (<br>Sm-p80<br>GLA-Sl<br>ayed boo<br>(N=X) | + <b>5 μg</b><br>Ε | 30 μg | Group I<br>Sm-p80<br>GLA-Sl<br>(N=X) | + <b>5 μg</b><br>Ε | 100 μg | Group F<br>Sm-p80<br>GLA-SI<br>(N=X) | ) + 5 μg<br>E | A | ll Subje | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Symptom | Severity | n | % | 95%<br>CI <sup>a</sup> | n | % | 95%<br>CI <sup>a</sup> | n | % | 95%<br>CI <sup>a</sup> | n | % | 95%<br>CI <sup>a</sup> | n | % | 95%<br>CI <sup>a</sup> | n | % | 95%<br>CI <sup>a</sup> |
| | Mild | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | |
| Injection Site Symp | otoms | | | | | | | | | | | | | | | | | | |
| Any Injection Site<br>Symptom | None | x | xx | x.x,<br>x.x | X | xx | x.x,<br>x.x | X | xx | x.x,<br>x.x | х | xx | x.x,<br>x.x | х | xx | x.x,<br>x.x | X | xx | x.x,<br>x.x |
| | Mild | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | |
| [Injection Site<br>Symptom 1] | None | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | |
| [Injection Site<br>Symptom 2] | None | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | |

Table 25: Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Maximum Severity and Treatment Group – Post Dose 1 (Continued)

| | | 100 | Group A) µg Sm-<br>adjuvan<br>(N=X) | -p80 | 10 μg | Group B<br>Sm-p80<br>GLA-SI<br>(N=X) | + 5 μg | 30 µg | Group C<br>Sm-p80<br>GLA-SI<br>yed boo<br>(N=X) | + 5 μg | 30 μg | Group E<br>Sm-p80<br>GLA-SI<br>(N=X) | +5 μg<br>Ε | 100 μg | Group E<br>Sm-p80<br>GLA-SF<br>(N=X) | + 5 μg | Al | l Subjec<br>(N = X) | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Symptom | Severity | n | % | 95%<br>CI <sup>a</sup> | n | % | 95%<br>CI <sup>a</sup> | n | % | 95%<br>CI <sup>a</sup> | n | % | 95%<br>CI <sup>a</sup> | n | % | 95%<br>CI <sup>a</sup> | n | % | 95%<br>CI <sup>a</sup> |

Note: N = Number of subjects in the Safety Population who received the specified dose. Severity is the maximum severity reported over all solicited symptoms post dosing for each subject.

<sup>a</sup>95% confidence intervals are from the Wilson score method without continuity correction.

#### Tables with similar format to Table 25:

- Table 26: Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Maximum Severity, and Treatment Group Post Dose 2
- Table 27: Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Maximum Severity, and Treatment Group Post Dose 3
- Table 28: Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Maximum Severity, and Treatment Group Post Any Dose

Table 29: Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Severity, and Day Post Dosing – Group A: 100 µg Sm-p80 (unadjuvanted), Post Dose 1

| | | Pre- | -Dose | Post | -Dose | Da | ıy 1 | Da | ıy 2 | Da | ıy 3 | Da | ıy 4 | Da | ıy 5 | Da | ıy 6 | Da | y 7+ |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Symptom | Severity | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| Any<br>Symptom | None | х | xx | х | xx | x | xx | х | xx | х | xx | х | xx | х | xx | х | xx | х | XX |
| | Mild | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | |
| | Not Reported | | | | | | | | | | | | | | | | | | |
| Systemic Sy | mptoms | | | | | | | | | | | | | | | | | | |
| Any<br>Systemic<br>Symptom | None | x | xx | х | xx | x | xx | x | xx | x | xx | x | xx | x | xx | x | xx | x | xx |
| | Mild | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | |
| | Not Reported | | | | | | | | | | | | | | | | | | |
| [Systemic<br>Symptom 1] | None | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | |
| | Not Reported | | | | | | | | | | | | | | | | | | |
| [Systemic<br>Symptom 2] | None | | | | | | | | | | | | | | | | | | |

Table 29: Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Severity, and Day Post Dosing – Group A: 100 μg Sm-p80 (unadjuvanted), Post Dose 1 (Continued)

| | | Pre- | -Dose | Post | -Dose | Da | y 1 | Da | y 2 | Da | y 3 | Da | y 4 | Da | ıy 5 | Da | ıy 6 | Day | y 7+ |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Symptom | Severity | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| | Mild | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | |
| | Not Reported | | | | | | | | | | | | | | | | | | |
| Injection Sit | e Symptoms | | | | | | | | | | | | | | | | | | |
| Any<br>Injection<br>Site<br>Symptom | None | х | xx | х | XX | x | xx | X | xx | X | xx | X | xx | х | XX | х | xx | X | xx |
| | Mild | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | |
| | Not Reported | | | | | | | | | | | | | | | | | | |
| [Injection<br>Site<br>Symptom 1] | None | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | |
| | Not Reported | | | | | | | | | | | | | | | | | | |
| [Injection<br>Site<br>Symptom 2] | None | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | |

Table 29: Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Severity, and Day Post Dosing – Group A: 100 μg Sm-p80 (unadjuvanted), Post Dose 1 (Continued)

| 100 μg Sm-p | 80 (unadjuvanted | ), Post I | Dose 1 (N | N=X) | | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Pre- | Dose | Post- | -Dose | Da | y 1 | Da | y 2 | Da | y 3 | Da | y 4 | Da | ıy 5 | Da | y 6 | Day | y 7+ |
| Symptom | Severity | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| | Moderate | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | |
| | Not Reported | | | | | | | | | | | | | | | | | | |

Note: N = Number of subjects in the Safety Population who received the specified dose. Severity is the maximum severity reported post dosing for each subject for each day.

Tables with similar format to Table 29:

[Implementation Note: Replace header with appropriate treatment and dose.]

- Table 30: Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Severity, and Day Post Dosing Group A: 100 µg Sm-p80 (unadjuvanted), Post Dose 2
- Table 31: Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Severity, and Day Post Dosing Group A: 100 µg Sm-p80 (unadjuvanted), Post Dose 3
- Table 32: Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Severity, and Day Post Dosing Group B: 10 μg Sm-p80 + 5 μg GLA-SE, Post Dose 1
- Table 33: Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Severity, and Day Post Dosing Group B: 10 μg Sm-p80 + 5 μg GLA-SE, Post Dose 2
- Table 34: Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Severity, and Day Post Dosing Group B: 10 μg Sm-p80 + 5 μg GLA-SE, Post Dose 3
- Table 35: Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Severity, and Day Post Dosing Group C: 30 μg Sm-p80 + 5 μg GLA-SE (delayed booster), Post Dose 1
- Table 36: Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Severity, and Day Post Dosing Group C: 30 μg Sm-p80 + 5 μg GLA-SE (delayed booster), Post Dose 2
- Table 37: Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Severity, and Day Post Dosing Group C: 30 μg Sm-p80 + 5 μg GLA-SE (delayed booster), Post Dose 3
- Table 38: Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Severity, and Day Post Dosing Group D: 30 μg Sm-p80 + 5 μg GLA-SE, Post Dose 1
- Table 39: Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Severity, and Day Post Dosing Group D: 30 μg Sm-p80 + 5 μg GLA-SE, Post Dose 2
- Table 40: Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Severity, and Day Post Dosing Group D: 30 μg Sm-p80 + 5 μg GLA-SE, Post Dose 3
- Table 41: Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Severity, and Day Post Dosing Group E: 100 µg Sm-p80 + 5 µg GLA-SE, Post Dose 1
- Table 42: Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Severity, and Day Post Dosing Group E: 100 µg Sm-p80 + 5 µg GLA-SE, Post Dose 2
- Table 43: Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Severity, and Day Post Dosing Group E: 100 µg Sm-p80 + 5 µg GLA-SE, Post Dose 3

Table 44: Number and Percentage of Subjects Experiencing Solicited Events for Dose 1 Compared with Dose 2 and Dose 3 by Treatment Group

[Implementation Note: Add group name to treatment, e.g. "Group A: 100 µg Sm-p80 (unadjuvanted)".]

| Treatment<br>Group | | Dose 2 – Subjects<br>with No Symptoms | Dose 2 – Subjects<br>with Moderate or<br>Greater Symptoms | Dose 2 – Total<br>Number of<br>Subjects | Dose 3 – Subjects<br>with No Symptoms | Dose 3 – Subjects<br>with Moderate or<br>Greater Symptoms | Dose 3 – Total<br>Number of<br>Subjects |
|---|---|---|---|---|---|---|---|
| Systemic Sympton | ns | | | | | | |
| 100 μg Sm-p80<br>(unadjuvanted) | Dose 1 Subject<br>with No Symptoms | x (%) | x (%) | x (%) | x (%) | x (%) | x (%) |
| | Dose 1 Subjects<br>with Moderate or<br>Greater Symptoms | x (%) | x (%) | x (%) | x (%) | x (%) | x (%) |
| | Dose 1 Total<br>Number of Subjects | x (%) | x (%) | x (100%) | x (%) | x (%) | x (100%) |
| 10 μg Sm-p80 + 5<br>μg GLA-SE | Dose 1 Subject<br>with No Symptoms | | | | | | |
| | Dose 1 Subjects<br>with Moderate or<br>Greater Symptoms | | | | | | |
| | Dose 1 Total<br>Number of Subjects | | | | | | |
| 30 μg Sm-p80 + 5<br>μg GLA-SE | Dose 1 Subject<br>with No Symptoms | | | | | | |
| | Dose 1 Subjects<br>with Moderate or<br>Greater Symptoms | | | | | | |
| | Dose 1 Total<br>Number of Subjects | | | | | | |
| 30 μg Sm-p80 + 5<br>μg GLA-SE<br>(delayed booster) | Dose 1 Subject<br>with No Symptoms | | | | | | |

Table 44: Number and Percentage of Subjects Experiencing Solicited Events for Dose 1 Compared with Dose 2 and Dose 3 by Treatment Group (Continued)

| | | | | 1 |
|---|---|---|---|---|
| | Dose 1 Subjects<br>with Moderate or<br>Greater Symptoms | | | |
| | Dose 1 Total<br>Number of Subjects | | | |
| 100 μg Sm-p80 +<br>5 μg GLA-SE | Dose 1 Subject with No Symptoms | | | |
| | Dose 1 Subjects<br>with Moderate or<br>Greater Symptoms | | | |
| | Dose 1 Total<br>Number of Subjects | | | |
| <b>Local Symptoms</b> | | | | |
| 100 μg Sm-p80<br>(unadjuvanted) | Dose 1 Subjects with No Symptoms | x (%) | x (%) | x (%) |
| | Dose 1 Subjects<br>with Moderate or<br>Greater Symptoms | x (%) | x (%) | x (%) |
| | Dose 1Total<br>Number of Subjects | x (%) | x (%) | x (100%) |
| 10 μg Sm-p80 + 5<br>μg GLA-SE | Dose 1 Subject<br>with No Symptoms | | | |
| | Dose 1 Subjects<br>with Moderate or<br>Greater Symptoms | | | |
| | Dose 1 Total<br>Number of Subjects | | | |
| 30 μg Sm-p80 + 5<br>μg GLA-SE | Dose 1 Subject<br>with No Symptoms | | | |

Table 44: Number and Percentage of Subjects Experiencing Solicited Events for Dose 1 Compared with Dose 2 and Dose 3 by Treatment Group (Continued)

| | Dose 1 Subjects<br>with Moderate or<br>Greater Symptoms | |
|---|---|---|
| | Dose 1 Total<br>Number of Subjects | |
| 30 μg Sm-p80 + 5<br>μg GLA-SE<br>(delayed booster) | Dose 1 Subject<br>with No Symptoms | |
| | Dose 1 Subjects<br>with Moderate or<br>Greater Symptoms | |
| | Dose 1 Total<br>Number of Subjects | |
| 100 μg Sm-p80 +<br>5 μg GLA-SE | Dose 1 Subject<br>with No Symptoms | |
| | Dose 1 Subjects<br>with Moderate or<br>Greater Symptoms | |
| | Dose 1 Total<br>Number of Subjects | who received both dose |

Note: Denominators for percentages are the number of subjects in the Safety Population who received both doses being compared.

#### Pseudo Code:

```
/*Data Format*/
ID
        Dose1 Dose2 Dose3
            0
                 1
            1
                    1
 В
           0
                    0
С
            1 1
                           0
Where 0 = No Symptoms and 1 = Moderate or Greater at the given dose
proc freq data= t56;
tables Dose1*Dose2 / out= dose12; /*counts for dose 1 vs. dose 2*/
tables Dose1*Dose3 / out= _dose13; /*counts for dose 1 vs. dose 3*/
run;
```

#### 14.3.1.2 Unsolicited Adverse Events

Table 45: Summary of Unsolicited Adverse Events by MedDRA System Organ Class and Preferred Term, and Treatment Group – Post Dose 1

| MedDRA System Organ | 100 | Group A<br>) µg Sm-<br>adjuvan<br>(N=X) | -p80<br>ited) | 10 μg | Group B<br>Sm-p80<br>GLA-SF<br>(N=X) | + 5 μg | 30 µg | Group C<br>Sm-p80<br>GLA-SE<br>yed boo<br>(N=X) | + 5 μg | 30 μg | Group D<br>Sm-p80<br>GLA-SI<br>(N=X) | + 5 μg | 100 μg | Group E<br>Sm-p80<br>GLA-SI<br>(N=X) | ) + 5 μg | Al | ll Subjec<br>(N=X) | ets |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Class/<br>Preferred Term | n | % | 95%<br>CI <sup>a</sup> | n | % | 95%<br>CI <sup>a</sup> | n | % | 95%<br>CI <sup>a</sup> | n | % | 95%<br>CI <sup>a</sup> | n | % | 95%<br>CI <sup>a</sup> | n | % | 95%<br>CI <sup>a</sup> |
| Any SOC | X | XX | xx, xx | X | XX | xx, xx | X | XX | xx, xx | X | XX | xx, xx | X | XX | xx, xx | X | XX | xx, xx |
| [SOC 1] | | | | | | | | | | | | | | | | | | |
| [PT 1] | | | | | | | | | | | | | | | | | | |
| [PT 2] | | | | | | | | | | | | | | | | | | |
| [SOC 2] | | | | | | | | | | | | | | | | | | |
| [PT 1] | | | | | | | | | | | | | | | | | | |
| [PT 2] | | | | | | | | | | | | | | | | | | |

Note: N = number of subjects in the Safety Population who received the specified dose. This table presents number and percentage of subjects. A subject is only counted once per PT/time point.

## <u>Tables with similar format to Table 45:</u>

- Table 46: Summary of Unsolicited Adverse Events by MedDRA System Organ Class and Preferred Term, and Treatment Group Post Dose 2
- Table 47: Summary of Unsolicited Adverse Events by MedDRA System Organ Class and Preferred Term, and Treatment Group Post Dose 3

<sup>&</sup>lt;sup>a</sup>95% confidence intervals are from the Wilson score method without continuity correction.

Table 48: Unsolicited Adverse Events by MedDRA System Organ Class and Preferred Term, Maximum Severity, Relationship, and Treatment Group

| MedDRA<br>System | Preferred | Severity | | 00 μg<br>nadju | | 80 | | μg Sn<br>μg GI | | + 5 | | Grou<br>µg Sn<br>µg GI<br>layed<br>(N= | 1-p80<br>LA-SI | + <b>5</b> | 30 | Grou<br>µg Sn<br>µg GI<br>(N = | ı-p80 | + 5 | 100 | Grou<br>μg Sr<br>μg GI<br>(N = | n-p8( | ) + <b>5</b> | 1 | All Su<br>(N = | | s |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Organ<br>Class | Term | | Rel | ated | | ot<br>ated | Rel | ated | | ot<br>ated | Rela | ated | | ot<br>ated | | ot<br>ated | | ot<br>ated | Rel | ated | | ot<br>ated | Rel | ated | | ot<br>ated |
| | | | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| Any SOC | Any PT | Any<br>Severity | Х | XX | Х | XX | х | XX | х | XX | Х | XX | х | XX | Х | XX | х | XX | Х | XX | Х | XX | Х | XX | х | xx |
| | | Mild | | | | | | | | | | | | | | | | | | | | | | | | |
| | | Moderate | | | | | | | | | | | | | | | | | | | | | | | | |
| | | Severe | | | | | | | | | | | | | | | | | | | | | | | | |
| SOC 1 | PT 1 | Any<br>Severity | | | | | | | | | | | | | | | | | | | | | | | | |
| | | Mild | | | | | | | | | | | | | | | | | | | | | | | | |
| | | Moderate | | | | | | | | | | | | | | | | | | | | | | | | |
| | | Severe | | | | | | | | | | | | | | | | | | | | | | | | |
| | PT 2 | Any<br>Severity | | | | | | | | | | | | | | | | | | | | | | | | |
| | | Mild | | | | | | | | | | | | | | | | | | | | | | | | |
| | | Moderate | | | | | | | | | | | | | | | | | | | | | | | | |
| | | Severe | | | | | | | | | | | | | | | | | | | | | | | | |

Table 49: Related Unsolicited Adverse Events Within 28 Days Post Dosing by MedDRA System Organ Class and Preferred Term and Dose – Group A: 100 μg Sm-p80 (unadjuvanted) (N=X)

| | | ] | Post Dose | 1 | | Post Dose | 2 | ] | Post Dose | 3 | Po | st Any D | ose |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| MedDRA System Organ<br>Class | MedDRA Preferred<br>Term | n | % | Events | n | % | Events | n | % | Events | n | % | Events |
| Any SOC | Any PT | Х | XX | х | Х | XX | х | X | XX | х | X | XX | x |
| [SOC 1] | Any PT | | | | | | | | | | | | |
| | [PT 1] | | | | | | | | | | | | |
| | [PT 2] | | | | | | | | | | | | |
| [SOC 2] | Any PT | | | | | | | | | | | | |
| | [PT 1] | | | | | | | | | | | | |
| | [PT 2] | | | | | | | | | | | | |
| Note: N = Number of subjects | in the Safety Population. Th | is table pr | esents nun | nber and pe | ercentage | of subjects | For each t | time point | a subject | is only cou | inted once | per PT. | |

Tables with similar format to Table 49:

- Table 50: Related Unsolicited Adverse Events Within 28 Days Post Dosing by MedDRA System Organ Class and Preferred Term, and Dose Group B: 10 µg Sm-p80 + 5 µg GLA-SE (N=X)
- Table 51: Related Unsolicited Adverse Events Within 28 Days Post Dosing by MedDRA System Organ Class and Preferred Term, and Dose Group C: 30 µg Sm-p80 + 5 µg GLA-SE (delayed booster) (N=X)
- Table 52: Related Unsolicited Adverse Events Within 28 Days Post Dosing by MedDRA System Organ Class and Preferred Term, and Dose Group D: 30 µg Sm-p80 + 5 µg GLA-SE (N=X)
- Table 53: Related Unsolicited Adverse Events Within 28 Days Post Dosing by MedDRA System Organ Class and Preferred Term, and Dose Group Ε: 100 μg Sm-p80 + 5 μg GLA-SE (N=X)

## 14.3.2 Listing of Deaths, Other Serious and Significant Adverse Events

**Table 54:** Listing of Serious Adverse Events

| Adverse<br>Event | Associated<br>with Dose<br>No. | No. of<br>Days Post<br>Associated<br>Dose<br>(Duration) | No. of<br>Days Post<br>Dose the<br>Event<br>Became<br>Serious | Reason<br>Reported<br>as an SAE | Severity | Relationship<br>to Study<br>Treatment | If Not<br>Related,<br>Alternative<br>Etiology | Action<br>Taken<br>with<br>Study<br>Treatment | Subject<br>Discontinued<br>Due to AE | Outcome | MedDRA<br>System<br>Organ<br>Class | MedDRA<br>Preferred<br>Term |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject II | D: , Treatmen | t Group: , AE | Number: | | | | | | | | | |
| Comments | S: | | | | | | | | | | | |
| Subject II | D: , Treatmen | t Group: , AE | Number: | | | | | | | | | |
| Comments | s: | | | | | | | | | 1 | | |

Table 55: Listing of Non-Serious, Unsolicited, Moderate or Severe Adverse Events

| Adverse<br>Event | Associated with Dose No. | No. of Days<br>Post<br>Associated<br>Dose<br>(Duration) | Severity | Relationship<br>to Study<br>Treatment | If Not<br>Related,<br>Alternative<br>Etiology | Action Taken<br>with Study<br>Treatment | Subject<br>Discontinued<br>Due to AE | Outcome | MedDRA<br>System Organ<br>Class | MedDRA<br>Preferred<br>Term |
|---|---|---|---|---|---|---|---|---|---|---|
| Subject ID: , Tr | eatment Group: , | AE Number: | | | | | | | | |
| | | | | | T | | | | ı | |
| Comments: | | | | | | | | | | |
| Subject ID: , Tr | eatment Group: , | AE Number: | | | | | | | | |
| Comments: | | | | | l | | | | | |

 Table 56:
 Listing of Other Significant Adverse Events

| Adverse<br>Event | Number of<br>Doses<br>Received at<br>Time of<br>Event | No. of Days<br>Post<br>Associated<br>Dose | Duration of<br>Event | Severity | MedDRA<br>System<br>Organ Class | MAAE? | PIMMC/AESI? | NOCMC? | Relationship | Outcome |
|---|---|---|---|---|---|---|---|---|---|---|
| Subject ID: , | Freatment Grou | ip: , AE Numbe | r: | | | | | | | |
| | Comments: | | | | | | | | | |
| Subject ID: , | Treatment Grou | ıp: , AE Numbe | r: | | | | | | | |
| | Comments: | 1 | ı | | 1 | | 1 | | 1 | |

## 14.3.3 Narratives of Deaths, Other Serious and Significant Adverse Events

(not included in SAP, but this is a placeholder for the CSR)

## 14.3.4 Abnormal Laboratory Value Listings (by Subject)

 Table 57:
 Listing of Abnormal Laboratory Results - Chemistry

| Subject<br>ID | Treatment<br>Group | Sex | Age<br>(years) | Planned<br>Time Point | Actual<br>Study Day | Laboratory<br>Parameter<br>(Units) | Result<br>(Severity) | Relationship to<br>Treatment | If Not Related,<br>Alternate<br>Etiology | Action Taken<br>with Study<br>Treatment | Subject Discontinued Due to Result? |
|---|---|---|---|---|---|---|---|---|---|---|---|

 Table 58:
 Listing of Abnormal Laboratory Results - Hematology

| Subject<br>ID | Treatment<br>Group | Sex | Age<br>(years) | Planned<br>Time Point | Actual<br>Study Day | Laboratory<br>Parameter<br>(Units) | Result<br>(Severity) | Relationship to<br>Treatment | If Not Related,<br>Alternate<br>Etiology | Action Taken<br>with Study<br>Treatment | Subject Discontinued Due to Result? |
|---|---|---|---|---|---|---|---|---|---|---|---|

## 14.3.5 Displays of Laboratory Results

## 14.3.5.1 Chemistry Results

Table 59: Laboratory Results by Parameter, Maximum Severity, Time Point, and Treatment Group – Any Chemistry Parameter

[Implementation Note: Add group name to treatment, e.g. "Group A: 100 µg Sm-p80 (unadjuvanted)".]

| Time Point | Treatment Group | | N | one | Mild /<br>Grade 1 | | Moderate/<br>Grade 2 | | Severe/<br>Grade 3 | | Missing | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | N | n | % | n | % | n | % | n | % | n | % |
| Study Day 1<br>(Baseline) | 100 μg Sm-p80 (unadjuvanted) | х | Х | XX | X | XX | Х | xx | X | XX | х | XX |
| | 10 μg Sm-p80 + 5 μg GLA-SE | | | | | | | | | | | |
| | 30 μg Sm-p80 + 5 μg GLA-SE (delayed booster) | | | | | | | | | | | |
| | 30 μg Sm-p80 + 5 μg GLA-SE | | | | | | | | | | | |
| | 100 μg Sm-p80 + 5 μg GLA-SE | | | | | | | | | | | |
| Study Day 8 | 100 μg Sm-p80 (unadjuvanted) | | | | | | | | | | | |
| | 10 μg Sm-p80 + 5 μg GLA-SE | | | | | | | | | | | |
| | 30 μg Sm-p80 + 5 μg GLA-SE (delayed booster) | | | | | | | | | | | |
| | 30 μg Sm-p80 + 5 μg GLA-SE | | | | | | | | | | | |
| | 100 μg Sm-p80 + 5 μg GLA-SE | | | | | | | | | | | |
| Study Day 29 | 100 μg Sm-p80 (unadjuvanted) | | | | | | | | | | | |
| | 10 μg Sm-p80 + 5 μg GLA-SE | | | | | | | | | | | |
| | 30 μg Sm-p80 + 5 μg GLA-SE (delayed booster) | | | | | | | | | | | |
| | 30 μg Sm-p80 + 5 μg GLA-SE | | | | | | | | | | | |
| | 100 μg Sm-p80 + 5 μg GLA-SE | | | | | | | | | | | |
| Study Day 36 | 100 μg Sm-p80 (unadjuvanted) | | | | | | | | | | | |

Table 59: Laboratory Results by Parameter, Maximum Severity, Time Point, and Treatment Group – Any Chemistry Parameter (Continued)

| | Continued) | | None | | Mild /<br>Grade 1 | | | erate/<br>ide 2 | Severe/<br>Grade 3 | | Missing | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time Point | Treatment Group | N | n | % | n | % | n | % | n | % | n | % |
| | 10 μg Sm-p80 + 5 μg GLA-SE | | | | | | | | | | | |
| | 30 μg Sm-p80 + 5 μg GLA-SE (delayed booster) | | | | | | | | | | | |
| | 30 μg Sm-p80 + 5 μg GLA-SE | | | | | | | | | | | |
| | 100 μg Sm-p80 + 5 μg GLA-SE | | | | | | | | | | | |
| Study Day 57 | 100 μg Sm-p80 (unadjuvanted) | | | | | | | | | | | |
| | 10 μg Sm-p80 + 5 μg GLA-SE | | | | | | | | | | | |
| | 30 μg Sm-p80 + 5 μg GLA-SE (delayed booster) | | | | | | | | | | | |
| | 30 μg Sm-p80 + 5 μg GLA-SE | | | | | | | | | | | |
| | 100 μg Sm-p80 + 5 μg GLA-SE | | | | | | | | | | | |
| Study Day 64 | 100 μg Sm-p80 (unadjuvanted) | | | | | | | | | | | |
| | 10 μg Sm-p80 + 5 μg GLA-SE | | | | | | | | | | | |
| | 30 μg Sm-p80 + 5 μg GLA-SE | | | | | | | | | | | |
| | 100 μg Sm-p80 + 5 μg GLA-SE | | | | | | | | | | | |
| Study Day 85 | 100 μg Sm-p80 (unadjuvanted) | | | | | | | | | | | |
| | 10 μg Sm-p80 + 5 μg GLA-SE | | | | | | | | | | | |
| | 30 μg Sm-p80 + 5 μg GLA-SE | | | | | | | | | | | |
| | 100 μg Sm-p80 + 5 μg GLA-SE | | | | | | | | | | | |
| Study Day 180 | 30 μg Sm-p80 + 5 μg GLA-SE (delayed booster) | | | | | | | | | | | |
| Study Day 187 | 30 μg Sm-p80 + 5 μg GLA-SE (delayed booster) | | | | | | | | | | | |
Table 59: Laboratory Results by Parameter, Maximum Severity, Time Point, and Treatment Group – Any Chemistry Parameter (Continued)

| | | | None | | Mild /<br>Grade 1 | | Moderate/<br>Grade 2 | | Severe/<br>Grade 3 | | Missing | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time Point | Treatment Group | N | n | % | n | % | n | % | n | % | n | % |
| Study Day 208 | 30 μg Sm-p80 + 5 μg GLA-SE (delayed booster) | | | | | | | | | | | |
| Max Severity Post<br>Baseline | 100 μg Sm-p80 (unadjuvanted) | | | | | | | | | | | |
| | 10 μg Sm-p80 + 5 μg GLA-SE | | | | | | | | | | | |
| | 30 μg Sm-p80 + 5 μg GLA-SE (delayed booster) | | | | | | | | | | | |
| | 30 μg Sm-p80 + 5 μg GLA-SE | | | | | | | | | | | |
| | 100 μg Sm-p80 + 5 μg GLA-SE | | | | | | | | | | | |

Note: The "Max Post Baseline" rows indicate the maximum severity experienced by each subject at any time point post baseline, including unscheduled assessments. Note: N = Number of subjects in the Safety Population with lab results at the specified visit.

#### Tables with similar format to Table 59:

Table 60: Laboratory Results by Parameter, Maximum Severity, Time Point, and Treatment Group – Creatinine

Table 61: Laboratory Results by Parameter, Maximum Severity, Time Point, and Treatment Group -- Alanine Aminotransferase

Table 62: Abnormal Laboratory Results Related to Study Treatment by Parameter, Maximum Severity, Time Point, and Treatment Group – Any Chemistry Parameter

[Implementation Note: Only scheduled time points at which at least one related abnormal lab result is observed in any treatment group will be shown. Add group name to treatment, e.g. "Group A: 100 µg Sm-p80 (unadjuvanted)".]

| | | | N | one | | ild /<br>ade 1 | | erate/<br>ide 2 | | evere/<br>rade 3 |
|---|---|---|---|---|---|---|---|---|---|---|
| Time Point | Treatment Group | N | n | % | n | % | n | % | n | % |
| Study Day 1 (Baseline) | 100 μg Sm-p80 (unadjuvanted) | X | х | х | х | х | х | х | Х | X |
| | 10 μg Sm-p80 + 5 μg GLA-SE | | | | | | | | | |
| | 30 μg Sm-p80 + 5 μg GLA-SE (delayed booster) | | | | | | | | | |
| | 30 μg Sm-p80 + 5 μg GLA-SE | | | | | | | | | |
| | 100 μg Sm-p80 + 5 μg GLA-SE | | | | | | | | | |
| Study Day 8 | 100 μg Sm-p80 (unadjuvanted) | | | | | | | | | |
| | 10 μg Sm-p80 + 5 μg GLA-SE | | | | | | | | | |
| | 30 μg Sm-p80 + 5 μg GLA-SE (delayed booster) | | | | | | | | | |
| | 30 μg Sm-p80 + 5 μg GLA-SE | | | | | | | | | |
| | 100 μg Sm-p80 + 5 μg GLA-SE | | | | | | | | | |
| Study Day 29 | 100 μg Sm-p80 (unadjuvanted) | | | | | | | | | |
| | 10 μg Sm-p80 + 5 μg GLA-SE | | | | | | | | | |
| | 30 μg Sm-p80 + 5 μg GLA-SE (delayed booster) | | | | | | | | | |
| | 30 μg Sm-p80 + 5 μg GLA-SE | | | | | | | | | |
| | 100 μg Sm-p80 + 5 μg GLA-SE | | | | | | | | | |
| Study Day 36 | 100 μg Sm-p80 (unadjuvanted) | | | | | | | | | |
| | 10 μg Sm-p80 + 5 μg GLA-SE | | | | | | | | | |
| | 30 μg Sm-p80 + 5 μg GLA-SE (delayed booster) | | | | | | | | | |
| | 30 μg Sm-p80 + 5 μg GLA-SE | | | | | | | | | |
| | 100 μg Sm-p80 + 5 μg GLA-SE | | | | | | | | | |

Table 62: Abnormal Laboratory Results Related to Study Treatment by Parameter, Maximum Severity, Time Point, and Treatment Group

- Any Chemistry Parameter (Continued)

| | | | N | one | | ild /<br>ade 1 | | erate/<br>ide 2 | | evere/<br>rade 3 |
|---|---|---|---|---|---|---|---|---|---|---|
| Time Point | Treatment Group | N | n | % | n | % | n | % | n | % |
| Study Day 57 | 100 μg Sm-p80 (unadjuvanted) | | | | | | | | | |
| | 10 μg Sm-p80 + 5 μg GLA-SE | | | | | | | | | |
| | 30 μg Sm-p80 + 5 μg GLA-SE (delayed booster) | | | | | | | | | |
| | 30 μg Sm-p80 + 5 μg GLA-SE | | | | | | | | | |
| | 100 μg Sm-p80 + 5 μg GLA-SE | | | | | | | | | |
| Study Day 64 | 100 μg Sm-p80 (unadjuvanted) | | | | | | | | | |
| | 10 μg Sm-p80 + 5 μg GLA-SE | | | | | | | | | |
| | 30 μg Sm-p80 + 5 μg GLA-SE | | | | | | | | | |
| | 100 μg Sm-p80 + 5 μg GLA-SE | | | | | | | | | |
| Study Day 85 | 100 μg Sm-p80 (unadjuvanted) | | | | | | | | | |
| | 10 μg Sm-p80 + 5 μg GLA-SE | | | | | | | | | |
| | 30 μg Sm-p80 + 5 μg GLA-SE | | | | | | | | | |
| | 100 μg Sm-p80 + 5 μg GLA-SE | | | | | | | | | |
| Study Day 180 | 30 μg Sm-p80 + 5 μg GLA-SE (delayed booster) | | | | | | | | | |
| Study Day 187 | 30 μg Sm-p80 + 5 μg GLA-SE (delayed booster) | | | | | | | | | |
| Study Day 208 | 30 μg Sm-p80 + 5 μg GLA-SE (delayed booster) | | | | | | | | | |
| Max Severity Post<br>Baseline | 100 μg Sm-p80 (unadjuvanted) | | | | | | | | | |
| | 10 μg Sm-p80 + 5 μg GLA-SE | | | | | | | | | |
| | 30 μg Sm-p80 + 5 μg GLA-SE (delayed booster) | | | | | | | | | |
| | 30 μg Sm-p80 + 5 μg GLA-SE | | | | | | | | | |
| | 100 μg Sm-p80 + 5 μg GLA-SE | | | | | | | | | |

Table 62: Abnormal Laboratory Results Related to Study Treatment by Parameter, Maximum Severity, Time Point, and Treatment Group

- Any Chemistry Parameter (Continued)

| • | | | No | ne | Mi<br>Gra | | Mode | erate/<br>de 2 | | evere/<br>rade 3 |
|---|---|---|---|---|---|---|---|---|---|---|
| | | | 110 | | Gia | | Gia | | 0. | |
| Time Point | Treatment Group | N | n | % | n | % | n | % | n | % |

Note: The "Max Post Baseline" rows indicate the maximum severity experienced by each subject at any time point post baseline.

Note: N = Number of subjects in the Safety Population with lab results at the specified visit.

#### Tables with similar format to Table 62:

- Table 63: Abnormal Laboratory Results Related to Study Treatment by Parameter, Maximum Severity, Time Point, and Treatment Group
  - Creatinine
- Table 64: Abnormal Laboratory Results Related to Study Treatment by Parameter, Maximum Severity, Time Point, and Treatment Group
  - Alanine Aminotransferase

# Table 65: Laboratory Summary Statistics by Parameter, Time Point, and Treatment Group – Creatinine (mg/dL)

[Implementation Note: Add group name to treatment, e.g. "Group A: 100 µg Sm-p80 (unadjuvanted)".]

| Time Point | Treatment Group | N | Mean | Standard Deviation | Median | Min, Max |
|---|---|---|---|---|---|---|
| Study Day 1 (Baseline) | 100 μg Sm-p80 (unadjuvanted) | х | xx.x | XX.X | XX.X | xx, xx |
| | 10 μg Sm-p80 + 5 μg GLA-SE | | | | | |
| | 30 μg Sm-p80 + 5 μg GLA-SE<br>(delayed booster) | | | | | |
| | 30 μg Sm-p80 + 5 μg GLA-SE | | | | | |
| | 100 μg Sm-p80 + 5 μg GLA-SE | | | | | |
| Study Day 8 | 100 μg Sm-p80 (unadjuvanted) | | | | | |
| | 10 μg Sm-p80 + 5 μg GLA-SE | | | | | |
| | 30 μg Sm-p80 + 5 μg GLA-SE (delayed booster) | | | | | |
| | 30 μg Sm-p80 + 5 μg GLA-SE | | | | | |
| | 100 μg Sm-p80 + 5 μg GLA-SE | | | | | |
| Study Day 8, Change from Baseline | 100 μg Sm-p80 (unadjuvanted) | | | | | |
| Study Day 29 | 100 μg Sm-p80 (unadjuvanted) | | | | | |
| | 10 μg Sm-p80 + 5 μg GLA-SE | | | | | |
| | 30 μg Sm-p80 + 5 μg GLA-SE (delayed booster) | | | | | |
| | 30 μg Sm-p80 + 5 μg GLA-SE | | | | | |
| | 100 μg Sm-p80 + 5 μg GLA-SE | | | | | |
| Study Day 29, Change from Baseline | 100 μg Sm-p80 (unadjuvanted) | | | | | |
| Study Day 36 | 100 μg Sm-p80 (unadjuvanted) | | | | | |
| | 10 μg Sm-p80 + 5 μg GLA-SE | | | | | |
| | 30 μg Sm-p80 + 5 μg GLA-SE<br>(delayed booster) | | | | | |

Table 65: Laboratory Summary Statistics by Parameter, Time Point, and Treatment Group – Creatinine (mg/dL) (Continued)

| Time Point | Treatment Group | N | Mean | Standard Deviation | Median | Min, Max |
|---|---|---|---|---|---|---|
| | 30 μg Sm-p80 + 5 μg GLA-SE | | | | | |
| | 100 μg Sm-p80 + 5 μg GLA-SE | | | | | |
| Study Day 36, Change from Baseline | 100 μg Sm-p80 (unadjuvanted) | | | | | |
| Study Day 57 | 100 μg Sm-p80 (unadjuvanted) | | | | | |
| | 10 μg Sm-p80 + 5 μg GLA-SE | | | | | |
| | 30 μg Sm-p80 + 5 μg GLA-SE (delayed booster) | | | | | |
| | 30 μg Sm-p80 + 5 μg GLA-SE | | | | | |
| | 100 μg Sm-p80 + 5 μg GLA-SE | | | | | |
| Study Day 57, Change from Baseline | 100 μg Sm-p80 (unadjuvanted) | | | | | |
| Study Day 64 | 100 μg Sm-p80 (unadjuvanted) | | | | | |
| | 10 μg Sm-p80 + 5 μg GLA-SE | | | | | |
| | 30 μg Sm-p80 + 5 μg GLA-SE | | | | | |
| | 100 μg Sm-p80 + 5 μg GLA-SE | | | | | |
| Study Day 64, Change from Baseline | 100 μg Sm-p80 (unadjuvanted) | | | | | |
| Study Day 85 | 100 μg Sm-p80 (unadjuvanted) | | | | | |
| | 10 μg Sm-p80 + 5 μg GLA-SE | | | | | |
| | 30 μg Sm-p80 + 5 μg GLA-SE | | | | | |
| | 100 μg Sm-p80 + 5 μg GLA-SE | | | | | |
| Study Day 85, Change from Baseline | 100 μg Sm-p80 (unadjuvanted) | | | | | |
| Study Day 180 | 30 μg Sm-p80 + 5 μg GLA-SE<br>(delayed booster) | | | | | |

Table 65: Laboratory Summary Statistics by Parameter, Time Point, and Treatment Group – Creatinine (mg/dL) (Continued)

| Treatment Group | N | Mean | Standard Deviation | Median | Min, Max |
|---|---|---|---|---|---|
| 30 μg Sm-p80 + 5 μg GLA-SE<br>(delayed booster) | | | | | |
| 30 μg Sm-p80 + 5 μg GLA-SE (delayed booster) | | | | | |
| 30 μg Sm-p80 + 5 μg GLA-SE (delayed booster) | | | | | |
| 30 μg Sm-p80 + 5 μg GLA-SE<br>(delayed booster) | | | | | |
| 30 μg Sm-p80 + 5 μg GLA-SE<br>(delayed booster) | | | | | |
| | 30 μg Sm-p80 + 5 μg GLA-SE (delayed booster) 30 μg Sm-p80 + 5 μg GLA-SE (delayed booster) 30 μg Sm-p80 + 5 μg GLA-SE (delayed booster) 30 μg Sm-p80 + 5 μg GLA-SE (delayed booster) 30 μg Sm-p80 + 5 μg GLA-SE (delayed booster) | 30 μg Sm-p80 + 5 μg GLA-SE (delayed booster) 30 μg Sm-p80 + 5 μg GLA-SE (delayed booster) 30 μg Sm-p80 + 5 μg GLA-SE (delayed booster) 30 μg Sm-p80 + 5 μg GLA-SE (delayed booster) 30 μg Sm-p80 + 5 μg GLA-SE (delayed booster) 30 μg Sm-p80 + 5 μg GLA-SE | 30 μg Sm-p80 + 5 μg GLA-SE (delayed booster) 30 μg Sm-p80 + 5 μg GLA-SE (delayed booster) 30 μg Sm-p80 + 5 μg GLA-SE (delayed booster) 30 μg Sm-p80 + 5 μg GLA-SE (delayed booster) 30 μg Sm-p80 + 5 μg GLA-SE (delayed booster) 30 μg Sm-p80 + 5 μg GLA-SE | 30 μg Sm-p80 + 5 μg GLA-SE (delayed booster) 30 μg Sm-p80 + 5 μg GLA-SE (delayed booster) 30 μg Sm-p80 + 5 μg GLA-SE (delayed booster) 30 μg Sm-p80 + 5 μg GLA-SE (delayed booster) 30 μg Sm-p80 + 5 μg GLA-SE (delayed booster) | 30 μg Sm-p80 + 5 μg GLA-SE (delayed booster) 30 μg Sm-p80 + 5 μg GLA-SE (delayed booster) 30 μg Sm-p80 + 5 μg GLA-SE (delayed booster) 30 μg Sm-p80 + 5 μg GLA-SE (delayed booster) 30 μg Sm-p80 + 5 μg GLA-SE (delayed booster) |

Tables with similar format to Table 65:

Table 66: Laboratory Summary Statistics by Parameter, Time Point, and Treatment Group – Alanine Aminotransferase (IU/L)

# 14.3.5.2 Hematology Results

# Table 67: Laboratory Results by Parameter, Maximum Severity, Time Point, and Treatment Group – Any Hematology Parameter

[Implementation Note: Add group name to treatment, e.g. "Group A: 100 µg Sm-p80 (unadjuvanted)".]

| | | | N | one | | ild /<br>ide 1 | | erate/<br>ide 2 | | vere/<br>ade 3 | Mis | ssing |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time Point | Treatment Group | N | n | % | n | % | n | % | n | % | n | % |
| Study Day 1<br>(Baseline) | 100 μg Sm-p80 (unadjuvanted) | Х | х | XX | х | XX | Х | xx | Х | xx | х | XX |
| | 10 μg Sm-p80 + 5 μg GLA-SE | | | | | | | | | | | |
| | 30 μg Sm-p80 + 5 μg GLA-SE (delayed booster) | | | | | | | | | | | |
| | 30 μg Sm-p80 + 5 μg GLA-SE | | | | | | | | | | | |
| | 100 μg Sm-p80 + 5 μg GLA-SE | | | | | | | | | | | |
| Study Day 8 | 100 μg Sm-p80 (unadjuvanted) | | | | | | | | | | | |
| | 10 μg Sm-p80 + 5 μg GLA-SE | | | | | | | | | | | |
| | 30 μg Sm-p80 + 5 μg GLA-SE (delayed booster) | | | | | | | | | | | |
| | 30 μg Sm-p80 + 5 μg GLA-SE | | | | | | | | | | | |
| | 100 μg Sm-p80 + 5 μg GLA-SE | | | | | | | | | | | |
| Study Day 29 | 100 μg Sm-p80 (unadjuvanted) | | | | | | | | | | | |
| | 10 μg Sm-p80 + 5 μg GLA-SE | | | | | | | | | | | |
| | 30 μg Sm-p80 + 5 μg GLA-SE (delayed booster) | | | | | | | | | | | |
| | 30 μg Sm-p80 + 5 μg GLA-SE | | | | | | | | | | | |
| | 100 μg Sm-p80 + 5 μg GLA-SE | | | | | | | | | | | |
| Study Day 36 | 100 μg Sm-p80 (unadjuvanted) | | | | | | | | | | | |
| | 10 μg Sm-p80 + 5 μg GLA-SE | | | | | | | | | | | |
| | 30 μg Sm-p80 + 5 μg GLA-SE (delayed booster) | | | | | | | | | | | |
| | 30 μg Sm-p80 + 5 μg GLA-SE | | | | | | | | | | | |
| | 100 μg Sm-p80 + 5 μg GLA-SE | | | | | | | | | | | |
| Study Day 57 | 100 μg Sm-p80 (unadjuvanted) | | | | | | | | | | | |

Table 67: Laboratory Results by Parameter, Maximum Severity, Time Point, and Treatment Group – Any Hematology Parameter (Continued)

| | | | N | one | | ild /<br>ide 1 | | erate/<br>de 2 | | vere/<br>ade 3 | Mis | ssing |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time Point | Treatment Group | N | n | % | n | % | n | % | n | % | n | % |
| | 10 μg Sm-p80 + 5 μg GLA-SE | | | | | | | | | | | |
| | 30 μg Sm-p $80 + 5$ μg GLA-SE (delayed booster) | | | | | | | | | | | |
| | 30 μg Sm-p $80 + 5$ μg GLA-SE | | | | | | | | | | | |
| | 100 μg Sm-p80 + 5 μg GLA-SE | | | | | | | | | | | |
| Study Day 64 | 100 μg Sm-p80 (unadjuvanted) | | | | | | | | | | | |
| | 10 μg Sm-p80 + 5 μg GLA-SE | | | | | | | | | | | |
| | 30 μg Sm-p80 + 5 μg GLA-SE | | | | | | | | | | | |
| | 100 μg Sm-p80 + 5 μg GLA-SE | | | | | | | | | | | |
| Study Day 85 | 100 μg Sm-p80 (unadjuvanted) | | | | | | | | | | | |
| | 10 μg Sm-p80 + 5 μg GLA-SE | | | | | | | | | | | |
| | 30 μg Sm-p80 + 5 μg GLA-SE | | | | | | | | | | | |
| | 100 μg Sm-p80 + 5 μg GLA-SE | | | | | | | | | | | |
| Study Day 180 | 30 μg Sm-p80 + 5 μg GLA-SE (delayed booster) | | | | | | | | | | | |
| Study Day 187 | 30 μg Sm-p80 + 5 μg GLA-SE (delayed booster) | | | | | | | | | | | |
| Study Day 208 | 30 μg Sm-p80 + 5 μg GLA-SE (delayed booster) | | | | | | | | | | | |
| Max Severity Post<br>Baseline | 100 μg Sm-p80 (unadjuvanted) | | | | | | | | | | | |
| | 10 μg Sm-p80 + 5 μg GLA-SE | | | | | | | | | | | |
| | 30 μg Sm-p80 + 5 μg GLA-SE (delayed booster) | | | | | | | | | | | |
| | 30 μg Sm-p80 + 5 μg GLA-SE | | | | | | | | | | | |
| | 100 μg Sm-p80 + 5 μg GLA-SE | | | | | | | | | | | |

Note: The "Max Post Baseline" rows indicate the maximum severity experienced by each subject at any time point post baseline, including unscheduled assessments. Note: N = Number of subjects in the Safety Population with lab results at the specified visit.

#### Tables with similar format to Table 67:

[Implementation Note: For white blood cells and hemoglobin, columns will be separated into increase and decrease severity. For example, "Mild/Grade 1" will be "Mild/Grade 1 Decrease" and "Mild/Grade 1 Increase".]

Table 68: Laboratory Results by Parameter, Maximum Severity, Time Point, and Treatment Group – White Blood Cells

Table 69: Laboratory Results by Parameter, Maximum Severity, Time Point, and Treatment Group – Hemoglobin

Table 70: Laboratory Results by Parameter, Maximum Severity, Time Point, and Treatment Group – Platelets

# Table 71: Abnormal Laboratory Results Related to Study Treatment by Parameter, Maximum Severity, Time Point, and Treatment Group – Any Hematology Parameter

[Implementation Note: Only scheduled time points at which at least one related abnormal lab result is observed in any treatment group will be shown. Add group name to treatment, e.g. "Group A: 100 µg Sm-p80 (unadjuvanted)".]

| | | | N | one | | ild /<br>ade 1 | | erate/<br>ade 2 | | rere/<br>ide 3 |
|---|---|---|---|---|---|---|---|---|---|---|
| Time Point | Treatment Group | N | n | % | n | % | n | % | n | % |
| Study Day 1 (Baseline) | 100 μg Sm-p80 (unadjuvanted) | | | | | | | | | |
| | 10 μg Sm-p80 + 5 μg GLA-SE | | | | | | | | | |
| | 30 μg Sm-p80 + 5 μg GLA-SE (delayed booster) | | | | | | | | | |
| | 30 μg Sm-p80 + 5 μg GLA-SE | | | | | | | | | |
| | 100 μg Sm-p80 + 5 μg GLA-SE | | | | | | | | | |
| Study Day 8 | 100 μg Sm-p80 (unadjuvanted) | | | | | | | | | |
| | 10 μg Sm-p80 + 5 μg GLA-SE | | | | | | | | | |
| | 30 μg Sm-p80 + 5 μg GLA-SE (delayed booster) | | | | | | | | | |
| | 30 μg Sm-p80 + 5 μg GLA-SE | | | | | | | | | |
| | 100 μg Sm-p80 + 5 μg GLA-SE | | | | | | | | | |
| Study Day 29 | 100 μg Sm-p80 (unadjuvanted) | | | | | | | | | |
| | 10 μg Sm-p80 + 5 μg GLA-SE | | | | | | | | | |
| | 30 μg Sm-p80 + 5 μg GLA-SE (delayed booster) | | | | | | | | | |
| | 30 μg Sm-p80 + 5 μg GLA-SE | | | | | | | | | |
| | 100 μg Sm-p80 + 5 μg GLA-SE | | | | | | | | | |
| Study Day 36 | 100 μg Sm-p80 (unadjuvanted) | | | | | | | | | |
| | 10 μg Sm-p80 + 5 μg GLA-SE | | | | | | | | | |
| | 30 μg Sm-p80 + 5 μg GLA-SE (delayed booster) | | | | | | | | | |
| | 30 μg Sm-p80 + 5 μg GLA-SE | | | | | | | | | |
| | 100 μg Sm-p80 + 5 μg GLA-SE | | | | | | | | | |
| Study Day 57 | 100 μg Sm-p80 (unadjuvanted) | | | | | | | | | |

Table 71: Abnormal Laboratory Results Related to Study Treatment by Parameter, Maximum Severity, Time Point, and Treatment Group

- Any Hematology Parameter (Continued)

| | | | N | one | | ild /<br>ade 1 | Mod<br>Gra | erate/<br>de 2 | Sev<br>Gra | |
|---|---|---|---|---|---|---|---|---|---|---|
| Time Point | Treatment Group | N | n | % | n | % | n | % | n | % |
| | 10 μg Sm-p80 + 5 μg GLA-SE | | | | | | | | | |
| | 30 μg Sm-p80 + 5 μg GLA-SE (delayed booster) | | | | | | | | | |
| | 30 μg Sm-p80 + 5 μg GLA-SE | | | | | | | | | |
| | 100 μg Sm-p80 + 5 μg GLA-SE | | | | | | | | | |
| Study Day 64 | 100 μg Sm-p80 (unadjuvanted) | | | | | | | | | |
| | 10 μg Sm-p80 + 5 μg GLA-SE | | | | | | | | | |
| | 30 μg Sm-p80 + 5 μg GLA-SE | | | | | | | | | |
| | 100 μg Sm-p80 + 5 μg GLA-SE | | | | | | | | | |
| Study Day 85 | 100 μg Sm-p80 (unadjuvanted) | | | | | | | | | |
| | 10 μg Sm-p80 + 5 μg GLA-SE | | | | | | | | | |
| | 30 μg Sm-p80 + 5 μg GLA-SE | | | | | | | | | |
| | 100 μg Sm-p80 + 5 μg GLA-SE | | | | | | | | | |
| Study Day 180 | 30 μg Sm-p80 + 5 μg GLA-SE (delayed booster) | | | | | | | | | |
| Study Day 187 | 30 μg Sm-p80 + 5 μg GLA-SE (delayed booster) | | | | | | | | | |
| Study Day 208 | 30 μg Sm-p80 + 5 μg GLA-SE (delayed booster) | | | | | | | | | |
| Max Severity Post<br>Baseline | 100 μg Sm-p80 (unadjuvanted) | | | | | | | | | |
| | 10 μg Sm-p80 + 5 μg GLA-SE | | | | | | | | | |
| | 30 μg Sm-p80 + 5 μg GLA-SE (delayed booster) | | | | | | | | | |
| | 30 μg Sm-p80 + 5 μg GLA-SE | | | | | | | | | |
| | 100 μg Sm-p80 + 5 μg GLA-SE | | | | | | | | | |

Note: The "Max Post Baseline" rows indicate the maximum severity experienced by each subject at any time point post baseline, including unscheduled assessments.

Note: N = Number of subjects in the Safety Population with lab results at the specified visit.

#### Tables with similar format to Table 71:

[Implementation Note: For white blood cells and hemoglobin, columns will be separated into increase and decrease severity. For example, "Mild/Grade 1" will be "Mild/Grade 1 Decrease" and "Mild/Grade 1 Increase".]

- Table 72: Abnormal Laboratory Results Related to Study Treatment by Parameter, Maximum Severity, Time Point, and Treatment Group White Blood Cells
- Table 73: Abnormal Laboratory Results Related to Study Treatment by Parameter, Maximum Severity, Time Point, and Treatment Group Hemoglobin
- Table 74: Abnormal Laboratory Results Related to Study Treatment by Parameter, Maximum Severity, Time Point, and Treatment Group Platelets

Table 75: Laboratory Summary Statistics by Parameter, Time Point, and Treatment Group – White Blood Cells (109/L)

[Implementation Note: Add group name to treatment, e.g. "Group A: 100 µg Sm-p80 (unadjuvanted)".]

| Time Point | Treatment Group | N | Mean | Standard Deviation | Median | Min, Max |
|---|---|---|---|---|---|---|
| Study Day 1 (Baseline) | 100 μg Sm-p80 (unadjuvanted) | Х | XX.X | xx.x | XX.X | xx.x, xx.x |
| | 10 μg Sm-p80 + 5 μg GLA-SE | | | | | |
| | 30 μg Sm-p80 + 5 μg GLA-SE<br>(delayed booster) | | | | | |
| | 30 μg Sm-p80 + 5 μg GLA-SE | | | | | |
| | 100 μg Sm-p80 + 5 μg GLA-SE | | | | | |
| Study Day 8 | 100 μg Sm-p80 (unadjuvanted) | | | | | |
| | 10 μg Sm-p80 + 5 μg GLA-SE | | | | | |
| | 30 μg Sm-p80 + 5 μg GLA-SE<br>(delayed booster) | | | | | |
| | 30 μg Sm-p80 + 5 μg GLA-SE | | | | | |
| | 100 μg Sm-p80 + 5 μg GLA-SE | | | | | |
| Study Day 8, Change from Baseline | 100 μg Sm-p80 (unadjuvanted) | | | | | |
| Study Day 29 | 100 μg Sm-p80 (unadjuvanted) | | | | | |
| | 10 μg Sm-p80 + 5 μg GLA-SE | | | | | |
| | 30 μg Sm-p80 + 5 μg GLA-SE (delayed booster) | | | | | |
| | 30 μg Sm-p80 + 5 μg GLA-SE | | | | | |
| | 100 μg Sm-p80 + 5 μg GLA-SE | | | | | |
| Study Day 29, Change from Baseline | 100 μg Sm-p80 (unadjuvanted) | | | | | |
| Study Day 36 | 100 μg Sm-p80 (unadjuvanted) | | | | | |
| | 10 μg Sm-p80 + 5 μg GLA-SE | | | | | |
| | 30 μg Sm-p80 + 5 μg GLA-SE<br>(delayed booster) | | | | | |

Table 75: Laboratory Summary Statistics by Parameter, Time Point, and Treatment Group – White Blood Cells (109/L) (Continued)

| Time Point | Treatment Group | N | Mean | Standard Deviation | Median | Min, Max |
|---|---|---|---|---|---|---|
| | 30 μg Sm-p80 + 5 μg GLA-SE | | | | | |
| | 100 μg Sm-p80 + 5 μg GLA-SE | | | | | |
| Study Day 36, Change from Baseline | 100 μg Sm-p80 (unadjuvanted) | | | | | |
| Study Day 57 | 100 μg Sm-p80 (unadjuvanted) | | | | | |
| | 10 μg Sm-p80 + 5 μg GLA-SE | | | | | |
| | 30 μg Sm-p80 + 5 μg GLA-SE<br>(delayed booster) | | | | | |
| | 30 μg Sm-p80 + 5 μg GLA-SE | | | | | |
| | 100 μg Sm-p80 + 5 μg GLA-SE | | | | | |
| Study Day 57, Change from Baseline | 100 μg Sm-p80 (unadjuvanted) | | | | | |
| Study Day 64 | 100 μg Sm-p80 (unadjuvanted) | | | | | |
| | 10 μg Sm-p80 + 5 μg GLA-SE | | | | | |
| | 30 μg Sm-p80 + 5 μg GLA-SE | | | | | |
| | 100 μg Sm-p80 + 5 μg GLA-SE | | | | | |
| Study Day 64, Change from Baseline | 100 μg Sm-p80 (unadjuvanted) | | | | | |
| Study Day 85 | 100 μg Sm-p80 (unadjuvanted) | | | | | |
| | 10 μg Sm-p80 + 5 μg GLA-SE | | | | | |
| | 30 μg Sm-p80 + 5 μg GLA-SE | | | | | |
| | 100 μg Sm-p80 + 5 μg GLA-SE | | | | | |
| Study Day 85, Change from Baseline | 100 μg Sm-p80 (unadjuvanted) | | | | | |
| Study Day 180 | 30 μg Sm-p80 + 5 μg GLA-SE<br>(delayed booster) | | | | | |

Table 75: Laboratory Summary Statistics by Parameter, Time Point, and Treatment Group – White Blood Cells (109/L) (Continued)

| Time Point | Treatment Group | N | Mean | Standard Deviation | Median | Min, Max |
|---|---|---|---|---|---|---|
| Study Day 180, Change from Baseline | 30 μg Sm-p80 + 5 μg GLA-SE<br>(delayed booster) | | | | | |
| Study Day 187 | 30 μg Sm-p80 + 5 μg GLA-SE<br>(delayed booster) | | | | | |
| Study Day 187, Change from Baseline | 30 μg Sm-p80 + 5 μg GLA-SE (delayed booster) | | | | | |
| Study Day 208 | 30 μg Sm-p80 + 5 μg GLA-SE<br>(delayed booster) | | | | | |
| Study Day 208, Change from Baseline | 30 μg Sm-p80 + 5 μg GLA-SE<br>(delayed booster) | | | | | |

### <u>Tables with similar format to Table 75:</u>

Table 76: Laboratory Summary Statistics by Parameter, Time Point, and Treatment Group – Hemoglobin (g/dL)

Table 77: Laboratory Summary Statistics by Parameter, Time Point, and Treatment Group – Platelets (109/L)

#### 14.3.6 Displays of Vital Signs

#### Table 78: Vital Signs by Assessment, Maximum Severity, Time Point, and Treatment Group – Any Assessment

[Implementation Note: For Groups A, B, D, and E, vital signs will be assessed if clinically indicated for study days 85 and 181. For Group C, vital signs will be assessed if clinically indicated for study days 208 and 304. Only include these days if at least one subject assessed on the given day. Add group name to treatment, e.g. "Group A: 100 µg Sm-p80 (unadjuvanted)".]

| | | | None | | Mild /<br>Grade 1 | | Moderate/<br>Grade 2 | | Severe/<br>Grade 3 | | Missing | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time Point | Treatment Group | N | n | % | n | % | n | % | n | % | n | % |
| Study Day 1<br>(Baseline) | 100 μg Sm-p80 (unadjuvanted) | Х | Х | XX | X | XX | Х | XX | X | XX | х | XX |
| | 10 μg Sm-p80 + 5 μg GLA-SE | | | | | | | | | | | |
| | 30 μg Sm-p80 + 5 μg GLA-SE (delayed booster) | | | | | | | | | | | |
| | 30 μg Sm-p80 + 5 μg GLA-SE | | | | | | | | | | | |
| | 100 μg Sm-p80 + 5 μg GLA-SE | | | | | | | | | | | |
| Study Day 4 | 100 μg Sm-p80 (unadjuvanted) | | | | | | | | | | | |
| | 10 μg Sm-p80 + 5 μg GLA-SE | | | | | | | | | | | |
| | 30 μg Sm-p80 + 5 μg GLA-SE (delayed booster) | | | | | | | | | | | |
| | 30 μg Sm-p80 + 5 μg GLA-SE | | | | | | | | | | | |
| | 100 μg Sm-p80 + 5 μg GLA-SE | | | | | | | | | | | |
| Study Day 8 | 100 μg Sm-p80 (unadjuvanted) | | | | | | | | | | | |
| | 10 μg Sm-p80 + 5 μg GLA-SE | | | | | | | | | | | |
| | 30 μg Sm-p80 + 5 μg GLA-SE (delayed booster) | | | | | | | | | | | |
| | 30 μg Sm-p80 + 5 μg GLA-SE | | | | | | | | | | | |
| | 100 μg Sm-p80 + 5 μg GLA-SE | | | | | | | | | | | |
| Study Day 29 | 100 μg Sm-p80 (unadjuvanted) | | | | | | | | | | | |

Table 78: Vital Signs by Assessment, Maximum Severity, Time Point, and Treatment Group – Any Assessment (Continued)

| | | | None | | Mild /<br>Grade 1 | | Moderate/<br>Grade 2 | | Severe/<br>Grade 3 | | Missing | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time Point | Treatment Group | N | n | % | n | % | n | % | n | % | n | % |
| | 10 μg Sm-p80 + 5 μg GLA-SE | | | | | | | | | | | |
| | 30 μg Sm-p80 + 5 μg GLA-SE (delayed booster) | | | | | | | | | | | |
| | 30 μg Sm-p80 + 5 μg GLA-SE | | | | | | | | | | | |
| | 100 μg Sm-p80 + 5 μg GLA-SE | | | | | | | | | | | |
| Study Day 32 | 100 μg Sm-p80 (unadjuvanted) | | | | | | | | | | | |
| | 10 μg Sm-p80 + 5 μg GLA-SE | | | | | | | | | | | |
| | 30 μg Sm-p80 + 5 μg GLA-SE (delayed booster) | | | | | | | | | | | |
| | 30 μg Sm-p80 + 5 μg GLA-SE | | | | | | | | | | | |
| | 100 μg Sm-p80 + 5 μg GLA-SE | | | | | | | | | | | |
| Study Day 36 | 100 μg Sm-p80 (unadjuvanted) | | | | | | | | | | | |
| | 10 μg Sm-p80 + 5 μg GLA-SE | | | | | | | | | | | |
| | 30 μg Sm-p80 + 5 μg GLA-SE (delayed booster) | | | | | | | | | | | |
| | 30 μg Sm-p80 + 5 μg GLA-SE | | | | | | | | | | | |
| | 100 μg Sm-p80 + 5 μg GLA-SE | | | | | | | | | | | |
| Study Day 57 | 100 μg Sm-p80 (unadjuvanted) | | | | | | | | | | | |
| | 10 μg Sm-p80 + 5 μg GLA-SE | | | | | | | | | | | |
| | 30 μg Sm-p80 + 5 μg GLA-SE (delayed booster) | | | | | | | | | | | |
| | 30 μg Sm-p80 + 5 μg GLA-SE | | | | | | | | | | | |
| | 100 μg Sm-p80 + 5 μg GLA-SE | | | | | | | | | | | |
| Study Day 60 | 100 μg Sm-p80 (unadjuvanted) | | | | | | | | | | | |

Table 78: Vital Signs by Assessment, Maximum Severity, Time Point, and Treatment Group – Any Assessment (Continued)

| | | | None | | Mild /<br>Grade 1 | | Moderate/<br>Grade 2 | | Severe/<br>Grade 3 | | Missing | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time Point | Treatment Group | N | n | % | n | % | n | % | n | % | n | % |
| | 10 μg Sm-p80 + 5 μg GLA-SE | | | | | | | | | | | |
| | 30 μg Sm-p80 + 5 μg GLA-SE | | | | | | | | | | | |
| | 100 μg Sm-p80 + 5 μg GLA-SE | | | | | | | | | | | |
| Study Day 64 | 100 μg Sm-p80 (unadjuvanted) | | | | | | | | | | | |
| | 10 μg Sm-p80 + 5 μg GLA-SE | | | | | | | | | | | |
| | 30 μg Sm-p80 + 5 μg GLA-SE | | | | | | | | | | | |
| | 100 μg Sm-p80 + 5 μg GLA-SE | | | | | | | | | | | |
| Study Day 180 | 30 μg Sm-p80 + 5 μg GLA-SE (delayed booster) | | | | | | | | | | | |
| Study Day 183 | 30 μg Sm-p80 + 5 μg GLA-SE (delayed booster) | | | | | | | | | | | |
| Study Day 187 | 30 μg Sm-p80 + 5 μg GLA-SE (delayed booster) | | | | | | | | | | | |
| Max Severity Post<br>Baseline | 100 μg Sm-p80 (unadjuvanted) | | | | | | | | | | | |
| | 10 μg Sm-p80 + 5 μg GLA-SE | | | | | | | | | | | |
| | 30 μg Sm-p80 + 5 μg GLA-SE (delayed booster) | | | | | | | | | | | |
| | 30 μg Sm-p80 + 5 μg GLA-SE | | | | | | | | | | | |
| | 100 μg Sm-p80 + 5 μg GLA-SE | | | | | | | | | | | |

Note: The "Max Post Baseline" rows indicate the maximum severity experienced by each subject at any time point post baseline, including unscheduled assessments.

Note: N = Number of subjects in the Safety Population with lab results at the specified visit.

#### Tables with similar format to Table 78:

[Implementation Note: For systolic blood pressure, columns will be separated into increase and decrease severity. For example, "Mild/Grade 1" will be "Mild/Grade 1 Decrease" and "Mild/Grade 1 Increase".]

- Table 79: Vital Signs by Assessment, Maximum Severity, Time Point, and Treatment Group Systolic Blood Pressure
- Table 80: Vital Signs by Assessment, Maximum Severity, Time Point, and Treatment Group Diastolic Blood Pressure
- Table 81: Vital Signs by Assessment, Maximum Severity, Time Point, and Treatment Group Heart Rate
- Table 82: Vital Signs by Assessment, Maximum Severity, Time Point, and Treatment Group Oral Temperature

# 14.4 Summary of Concomitant Medications

Table 83: Number and Percentage of Subjects with Prior and Concurrent Medications by WHO Drug Classification and Treatment Group

| WHO Drug Code | WHO Drug Code<br>Level 2, Therapeutic | 100 μg<br>(unadji | up A:<br>Sm-p80<br>uvanted)<br>=X) | 10 μg Sτ<br>μg Gl | up A:<br>n-p80 + 5<br>LA-SE<br>=X) | 30 μg Sr<br>μg Gl<br>(delayed | up C:<br>n-p80 + 5<br>LA-SE<br>l booster)<br>=X) | 30 μg Sr<br>μg Gl | up D:<br>n-p80 + 5<br>LA-SE<br>=X) | 100 μg Si<br>μg Gl | up E:<br>m-p80 + 5<br>LA-SE<br>=X) | | ubjects<br>=X) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Level 1, Anatomic Group | Subgroup | n | % | n | % | n | % | n | % | n | % | n | % |
| Any Level 1 Codes | Any Level 2 Codes | X | XX | х | xx | х | xx | х | xx | х | XX | x | XX |
| [ATC Level 1 - 1] | Any [ATC 1 – 1] | | | | | | | | | | | | |
| | [ATC 2 - 1] | | | | | | | | | | | | |
| | [ATC 2 - 2] | | | | | | | | | | | | |
| | [ATC 2 - 3] | | | | | | | | | | | | |
| [ATC Level 1 – 2] | [ATC 2 - 1] | | | | | | | | | | | | |
| | [ATC 2 - 2] | | | | | | | | | | | | |
| | [ATC 2 - 3] | | | | | | | | | | | | |

Note: N = Number of subjects in the Safety Population; n=Number of subjects reporting taking at least one medication in the specific WHO Drug Class. Subjects are counted once per WHO Drug Code Level 2, Therapeutic Subgroup.

# APPENDIX 2. FIGURE MOCK-UPS

# LIST OF FIGURES

| Figure 1: | CONSORT Flow Diagram | 134 |
|---|---|---|
| Figure 2: | Reverse Cumulative Distribution of Anti-Sm-p80 ELISA Total IgG Results by Time Point and Treatment Group, mITT Immunogenicity Population | 135 |
| Figure 3: | Geometric Mean Anti-Sm-p80 ELISA Total IgG Response Over Time by Treatment Group with 95% Confidence Intervals, mITT Immunogenicity Population | 138 |
| Figure 4: | Individual Time Trends of ELISA Total IgG Response by Treatment Group, mITT Immunogenicity Population | 139 |
| Figure 5: | Maximum Severity of Solicited Systemic Symptoms per Subject by Day Post-Vaccination – Post Dose 1 | 140 |
| Figure 6: | Maximum Severity of Solicited Systemic Symptoms per Subject by Day Post-Vaccination – Post Dose 2 | 141 |
| Figure 7: | Maximum Severity of Solicited Systemic Symptoms per Subject by Day Post-Vaccination – Post Dose 3 | 141 |
| Figure 8: | Number and Percentage of Subjects Experiencing Solicited Systemic Events by Event, Maximum Severity, and Treatment Group – Post Dose 1 | 142 |
| Figure 9: | Number and Percentage of Subjects Experiencing Solicited Systemic Events by Event, Maximum Severity, and Treatment Group – Post Dose 2 | 142 |
| Figure 10: | Number and Percentage of Subjects Experiencing Solicited Systemic Events by Event, Maximum Severity, and Treatment Group – Post Dose 3 | 142 |
| Figure 11: | Number and Percentage of Subjects Experiencing Solicited Systemic Events by Event, Maximum Severity, and Treatment Group – Post Any Dose | 142 |
| Figure 12: | Maximum Severity of Solicited Injection Site Symptoms per Subject by Day Post-Vaccination – Post Dose 1 | 143 |
| Figure 13: | Maximum Severity of Solicited Injection Site Symptoms per Subject by Day Post-Vaccination – Post Dose 2 | 143 |
| Figure 14: | Maximum Severity of Solicited Injection Site Symptoms per Subject by Day Post-Vaccination – Post Dose 3 | 143 |
| Figure 15: | Number and Percentage of Subjects Experiencing Solicited Injection Site Events by Event, Maximum Severity, and Treatment Group – Post Dose 1 | 144 |
| Figure 16: | Number and Percentage of Subjects Experiencing Solicited Injection Site Events by Event, Maximum Severity, and Treatment Group – Post Dose 2 | 144 |
| Figure 17: | Number and Percentage of Subjects Experiencing Solicited Injection Site Events by Event, Maximum Severity, and Treatment Group – Post Dose 3 | 144 |
| Figure 18: | Number and Percentage of Subjects Experiencing Solicited Injection Site Events by Event, Maximum Severity, and Treatment Group – Post Any Dose | |
| | Duse | 1 77 |

| Figure 19: | Frequency of Related Adverse Events by MedDRA System Organ Class and Severity | 145 |
|---|---|---|
| Figure 20: | Incidence of Related Adverse Events by MedDRA® System Organ Class and Maximum Severity | 146 |
| Figure 21: | Laboratory Results by Scheduled Visits: Mean Changes from Baseline by Laboratory Parameter, and Treatment Group – Creatinine | 147 |
| Figure 22: | Laboratory Results by Scheduled Visits: Mean Changes from Baseline by Laboratory Parameter, and Treatment Group – Alanine Aminotransferase | 147 |
| Figure 23: | Laboratory Results by Scheduled Visits: Mean Changes from Baseline by Laboratory Parameter, and Treatment Group – White Blood Cells | 147 |
| Figure 24: | Laboratory Results by Scheduled Visits: Mean Changes from Baseline by Laboratory Parameter, Sex, and Treatment Group – Hemoglobin | 147 |
| Figure 25: | Laboratory Results by Scheduled Visits: Mean Changes from Baseline by Laboratory Parameter, and Treatment Group – Platelets | 148 |

# 10.1 Disposition of Subjects

Figure 1: CONSORT Flow Diagram



## 14.2 Efficacy/Immunogenicity Data

- 14.2.2 Efficacy/Immunogenicity Response Figures by Measure, Treatment/Vaccination, and Time Point
- Figure 2: Reverse Cumulative Distribution of Anti-Sm-p80 ELISA Total IgG Results by Time Point and Treatment Group, mITT Immunogenicity Population

[Implementation Note: Figure will be paneled by scheduled time point: 7 and 28 days after each vaccination, and 124 days after the last vaccination. The y-axis will be the "Percent of Subjects (%)" with a max of 100 and the x-axis will be "Baseline-Adjusted Concentrations (OD<sub>450</sub>)". Each treatment group will have its own marker type and color. A legend will be included containing each treatment group and dosage if enough space available, e.g. Group A would be displayed as "Group A: 100 µg Sm-p80 (unadjuvanted)". Otherwise treatment group only will be shown.]

Figure 2: Reverse Cumulative Distribution of Anti-Sm-p80 ELISA Total IgG Results by Time Point and Treatment Group, mITT Immunogenicity Population (continued)



#### Pseudo Code:

Figure 2: Reverse Cumulative Distribution of Anti-Sm-p80 ELISA Total IgG Results by Time Point and Treatment Group, mITT Immunogenicity Population (continued)

Figure 3: Geometric Mean Anti-Sm-p80 ELISA Total IgG Response Over Time by Treatment Group with 95% Confidence Intervals, mITT Immunogenicity Population

[Implementation Note: The y-axis will be "Baseline-Adjusted Concentrations (OD<sub>450</sub>)", and the x-axis will be actual study day labelled as "Study Day" with tick marks on 7-days post vaccination, 28-days post vaccination, and 124-days post last vaccination. Each treatment group will have its own marker type and color consistent across all figures. A legend will be included containing each treatment group and dosage if enough space available, e.g. Group A would be displayed as "Group A: 100 µg Sm-p80 (unadjuvanted)". Otherwise treatment group only will be shown.]



Figure 4: Individual Time Trends of ELISA Total IgG Response by Treatment Group, mITT Immunogenicity Population

[Implementation Note: Figure will be paneled (3 rows and 2 columns) by treatment group. The y-a xis should be labelled "Anti-CSP Total IgG Titers" and range from minimum to maximum values. If titer range exceeds 150, then scale y-axis by log base 2. The x-axis will be labelled "Study Day" with tick marks on 7-days post vaccination, 28-days post vaccination, and 124-days post last vaccination. A dashed black line will be added to show the geometric mean time trend. Add a legend for the dashed black line labelled "Geometric Mean". Panel labels will include treatment group and dose if enough space available, e.g. "Group A: 100 µg Sm-p80 (unadjuvanted)". Otherwise, treatment group only will be shown.]



#### 14.3 Safety Data

#### 14.3.1 Adverse Events

#### 14.3.1.1 Solicited Adverse Events

Figure 5: Maximum Severity of Solicited Systemic Symptoms per Subject by Day Post-Vaccination

- Post Dose 1

[Implementation Note: This figure will have 3 columns and 2 rows and will be paneled by treatment group and "All Subjects". The y-axis will be "Post Dose Day" and the x-axis will be "Percent of Subjects (%)". This figure will be annotated with the fraction of subjects who experienced the symptom (n/N). Panel labels will include treatment group and dose if enough space available, e.g. "Group A: 100 µg Sm-p80 (unadjuvanted)". Otherwise, treatment group only will be shown.]



Figures with similar format to Figure 5:

- Figure 6: Maximum Severity of Solicited Systemic Symptoms per Subject by Day Post-Vaccination Post Dose 2
- Figure 7: Maximum Severity of Solicited Systemic Symptoms per Subject by Day Post-Vaccination Post Dose 3

Figure 8: Number and Percentage of Subjects Experiencing Solicited Systemic Events by Event, Maximum Severity, and Treatment Group – Post Dose 1

[Implementation Note: The symptoms should start with "Any Symptom" and then in alphabetical order. This figure will have 3 columns and 2 rows and will be paneled by treatment group and "All Subjects". The y-axis will be "Symptom" and the x-axis will be "Percent of Subjects (%)". This figure will be annotated with the fraction of subjects who experienced the symptom (n/N). Panel labels will include treatment group and dose if enough space available, e.g. "Group A:  $100 \mu g$  Sm-p80 (unadjuvanted)". Otherwise, treatment group only will be shown.]



Figures with similar format to Figure 8:

- Figure 9: Number and Percentage of Subjects Experiencing Solicited Systemic Events by Event, Maximum Severity, and Treatment Group Post Dose 2
- Figure 10: Number and Percentage of Subjects Experiencing Solicited Systemic Events by Event, Maximum Severity, and Treatment Group Post Dose 3
- Figure 11: Number and Percentage of Subjects Experiencing Solicited Systemic Events by Event, Maximum Severity, and Treatment Group Post Any Dose

Figure 12: Maximum Severity of Solicited Injection Site Symptoms per Subject by Day Post-Vaccination – Post Dose 1

[Implementation Note: This figure will have 3 columns and 2 rows and will be paneled by treatment group and "All Subjects". The y-axis will be "Post Dose Day" and the x-axis will be "Percent of Subjects (%)". This figure will be annotated with the fraction of subjects who experienced the symptom (n/N). Panel labels will include treatment group and dose if enough space available, e.g. "Group A: 100 µg Sm-p80 (unadjuvanted)". Otherwise, treatment group only will be shown.]



Figures with similar format to Figure 12:

Figure 13: Maximum Severity of Solicited Injection Site Symptoms per Subject by Day Post-Vaccination – Post Dose 2

Figure 14: Maximum Severity of Solicited Injection Site Symptoms per Subject by Day Post-Vaccination – Post Dose 3

Figure 15: Number and Percentage of Subjects Experiencing Solicited Injection Site Events by Event, Maximum Severity, and Treatment Group – Post Dose 1

[Implementation Note: The symptoms should start with "Any Symptom" and then in alphabetical order. This figure will have 3 columns and 2 rows and will be paneled by treatment group and "All Subjects". The y-axis will be "Symptom" and the x-axis will be "Percent of Subjects (%)". This figure will be annotated with the fraction of subjects who experienced the symptom (n/N). Panel labels will include treatment group and dose if enough space available, e.g. "Group A:  $100 \mu g$  Sm-p80 (unadjuvanted)". Otherwise, treatment group only will be shown.]



Figures with similar format to Figure 15:

- Figure 16: Number and Percentage of Subjects Experiencing Solicited Injection Site Events by Event, Maximum Severity, and Treatment Group Post Dose 2
- Figure 17: Number and Percentage of Subjects Experiencing Solicited Injection Site Events by Event, Maximum Severity, and Treatment Group Post Dose 3
- Figure 18: Number and Percentage of Subjects Experiencing Solicited Injection Site Events by Event, Maximum Severity, and Treatment Group Post Any Dose
#### 14.3.1.2 Unsolicited Adverse Events

### Figure 19: Frequency of Related Adverse Events by MedDRA System Organ Class and Severity

[Implementation Note: This figure will include serious and non-serious unsolicited adverse events deemed related to the study product. The SOCs should be sorted "Any SOC" first and then descending frequency. This figure will have 3 columns and 2 rows and will be paneled by treatment group and "All Subjects". The y-axis will be "System Organ Class" and the x-axis will be "Number of Events". This figure will be annotated with the number of events (n). Panel labels will include treatment group and dose if enough space available, e.g. "Group A: 100 µg Sm-p80 (unadjuvanted)". Otherwise, treatment group only will be shown.]



Figure 20: Incidence of Related Adverse Events by MedDRA® System Organ Class and Maximum Severity

[Implementation Note: This figure will include serious and non-serious unsolicited adverse events deemed related to the study product. The SOCs should be sorted "Any SOC" first and then descending frequency. This figure will have 3 columns and 2 rows and will be paneled by treatment group and "All Subjects". The y-axis will be "System Organ Class" and the x-axis will be "Percent of Subjects (%)". This figure will be annotated with the fraction of subjects who experienced the symptom (n/N). Panel labels will include treatment group and dose if enough space available, e.g. "Group A: 100 µg Sm-p80 (unadjuvanted)". Otherwise, treatment group only will be shown.]



#### 14.3.5 Displays of Laboratory Results

Figure 21: Laboratory Results by Scheduled Visits: Mean Changes from Baseline by Laboratory Parameter, and Treatment Group – Creatinine

[Implementation Note: The x-axis will be actual study day labelled as "Study Day" with tick marks on vaccination days, 7-days post vaccination, and 28-days post vaccination. The y-axis will be the "Mean Change from Baseline"; include relevant units. For example, creatinine would be "Mean Change from Baseline (mg/dL)". A reference line will be added at Y=0. A legend will be included containing each treatment group and dosage if enough space available, e.g. Group A would be displayed as "Group A: 100 µg Sm-p80 (unadjuvanted)". Otherwise treatment group only will be shown.]



Figures with similar format to Figure 21:

- Figure 22: Laboratory Results by Scheduled Visits: Mean Changes from Baseline by Laboratory Parameter, and Treatment Group Alanine Aminotransferase
- Figure 23: Laboratory Results by Scheduled Visits: Mean Changes from Baseline by Laboratory Parameter, and Treatment Group White Blood Cells
- Figure 24: Laboratory Results by Scheduled Visits: Mean Changes from Baseline by Laboratory Parameter, Sex, and Treatment Group Hemoglobin

[Implementation Note: Panel by sex.]

Figure 25: Laboratory Results by Scheduled Visits: Mean Changes from Baseline by Laboratory Parameter, and Treatment Group – Platelets

# APPENDIX 3. LISTINGS MOCK-UPS

# LISTINGS

| Listing 1: | 16.1.6: Listing of Subjects Receiving Investigational Product | 151 |
|---|---|---|
| Listing 2: | 16.2.1: Early Terminations or Discontinued Subjects | 152 |
| Listing 3: | 16.2.2.1: Subject-Specific Protocol Deviations | 153 |
| Listing 4: | 16.2.2.2: Non-Subject-Specific Protocol Deviations | 154 |
| Listing 5: | 16.2.3: Subjects Excluded from Analysis Populations | 155 |
| Listing 6: | 16.2.4.1: Demographic Data | 156 |
| Listing 7: | 16.2.4.2: Pre-Existing and Concurrent Medical Conditions | 157 |
| Listing 8: | 16.2.5: Compliance and/or Drug Concentration Data | 158 |
| Listing 9: | 16.2.6: Individual Efficacy/Immunogenicity Response Data | 159 |
| Listing 10: | 16.2.7.1: Solicited Events – Systemic Symptoms | 160 |
| Listing 11: | 16.2.7.2: Solicited Events – Injection Site Symptoms | 161 |
| Listing 12: | 16.2.7.3: Unsolicited Adverse Events | 162 |
| Listing 13: | 16.2.8.1: Clinical Laboratory Results – Chemistry | 163 |
| Listing 14: | 16.2.8.2: Clinical Laboratory Results – Hematology | 164 |
| Listing 15: | 16.2.9.1: Vital Signs | 165 |
| Listing 16: | 16.2.9.2: Physical Exam Findings | 166 |
| Listing 17: | 16.2.10: Concomitant Medications | 167 |
| Listing 18: | 16.2.11.1: Pregnancy Reports – Maternal Information | 168 |
| Listing 19: | 16.2.11.2: Pregnancy Reports – Gravida and Para | 168 |
| Listing 20: | 16.2.11.3: Pregnancy Reports – Live Birth Outcomes | 169 |
| Listing 21: | 16.2.11.4: Pregnancy Reports – Still Birth Outcomes | 169 |
| Listing 22: | 16.2.11.5: Pregnancy Reports – Spontaneous, Elective, or Therapeutic Abortion Outcomes | 169 |

# Listing 1: 16.1.6: Listing of Subjects Receiving Investigational Product

(not included in SAP, but this is a placeholder for the CSR)

# 16.2 Database Listings by Subject

# 16.2.1 Discontinued Subjects

# **Listing 2:** 16.2.1: Early Terminations or Discontinued Subjects

[Implementation Note: Category will either by "Early Termination" or "Treatment Discontinuation". Sort by Treatment Group, Subject ID, alphabetically by Category.]

| Treatment Group | Subject ID | Category | Reason for Early Termination or Treatment Discontinuation | Study Day |
|---|---|---|---|---|

### **16.2.2 Protocol Deviations**

# **Listing 3:** 16.2.2.1: Subject-Specific Protocol Deviations

[Implementation Note: Sort by Treatment Group, Subject ID, DV Number.]

| Treatment<br>Group | Subject ID | DV Number | Deviation | Deviation<br>Category | Study Day | Reason for<br>Deviation | Deviation<br>Resulted<br>in AE? | Deviation Resulted<br>in Subject<br>Termination? | Deviation<br>Affected<br>Product<br>Stability? | Deviation<br>Resolution | Comments |
|---|---|---|---|---|---|---|---|---|---|---|---|

# Listing 4: 16.2.2.2: Non-Subject-Specific Protocol Deviations

[Implementation Note: Sort by Start Date. Use DATE9 format for all dates.]

| Start Date | Deviation | End Date | Reason for<br>Deviation | Deviation<br>Resulted in<br>Subject<br>Termination? | Deviation<br>Affected<br>Product<br>Stability? | Deviation<br>Category | Deviation<br>Resolution | Comments |
|---|---|---|---|---|---|---|---|---|

### 16.2.3 Subjects Excluded from the Efficacy Analysis

# **Listing 5:** 16.2.3: Subjects Excluded from Analysis Populations

[Implementation Note: Exclusion reasons should match the SAP text that describes who will be excluded from analyses. Sort by Treatment Group and Subject ID.]

| Treatment Group | Subject ID | Analyses in which<br>Subject is Included | Analyses from which<br>Subject is Excluded | Results Available? | Reason Subject Excluded |
|---|---|---|---|---|---|
| | | [e.g., Safety, ITT, PP] | [e.g., Safety, ITT, PP, Day x] | | |

Note: "Yes" in the "Results available" column indicates that available data were removed from the analysis. "No" indicates that no data were available for inclusion in the analysis.

# 16.2.4 Demographic Data

# Listing 6: 16.2.4.1: Demographic Data

[Implementation Note: Sort by Treatment Group and Subject ID.]

| Treatment Group | Subject ID | Sex | Age at Enrollment (years) | Ethnicity | Race |
|---|---|---|---|---|---|

# Listing 7: 16.2.4.2: Pre-Existing and Concurrent Medical Conditions

[Implementation Note: "Condition Start Day" and "Condition End Day" are relative to enrollment. Sort by Treatment Group, Subject ID, MH Number.]

| Treatment<br>Group | Subject ID | MH Number | Medical History Term | Condition Start Day | Condition End Day | MedDRA System Organ Class | MedDRA Preferred Term |
|---|---|---|---|---|---|---|---|

# 16.2.5 Compliance and/or Drug Concentration Data (if available)

# Listing 8: 16.2.5: Compliance and/or Drug Concentration Data

[Implementation Note: Sort by Treatment Group, Subject ID, and Dose Number.]

### Scenario 2

| Treatment Group | Subject ID | Dose(s) Missed |
|-----------------|------------|-------------------------------|
| | | [e.g., Day 3, Day 3 AM, etc.] |

# 16.2.6 Individual Efficacy/Immunogenicity Response Data

# Listing 9: 16.2.6: Individual Efficacy/Immunogenicity Response Data

[Implementation Note: Sort by Treatment Group, Subject ID, Planned Time Point.]

| Treatment Group | Subject ID | Planned Time Point | Actual Study Day | ELISA Total IgG |
|---|---|---|---|---|

#### 16.2.7 Adverse Events

#### **Listing 10:** 16.2.7.1: Solicited Events – Systemic Symptoms

[Implementation Note: To indicate severity for quantitative symptoms (*e.g.*, temperature, measurements), include the grade in parentheses after the number, *e.g.*, 100.7 (Mild). This listing will include baseline assessments and post-vaccination assessments. Sort by Subject ID, Dose Number, Post Dose Day, Symptom.]

| Treatment<br>Group | Subject ID | Dose Number | Post Dose Day | Assessmenta | Symptom | Severity | Attributed to<br>Alternate<br>Etiology? <sup>b</sup> | Alternate Etiology |
|---|---|---|---|---|---|---|---|---|
| | | | | MA | | | | |
| | | | | Clinic | | | | |

<sup>&</sup>lt;sup>a</sup> MA = Data reported by subject on the Memory Aid and reviewed by clinic staff and reported in Solicited Events eCRF.

Note: Clinic = Data collected by clinic staff during physical exam or symptom assessment (treatment administration record, in-clinic assessment, etc.)

<sup>&</sup>lt;sup>b</sup> Grade 3 events only.

### **Listing 11:** 16.2.7.2: Solicited Events – Injection Site Symptoms

[Implementation Note: To indicate severity for quantitative symptoms (*e.g.*, temperature, measurements), include the grade in parentheses after the number, *e.g.*, 100.7 (Mild). This listing will include baseline assessments and post-vaccination assessments. Sort by Subject ID, Dose Number, Post Dose Day, Symptom.]

| Treatment Group | Subject ID | Dose Number | Post Dose Day | Assessmenta | Symptom | Severity |
|---|---|---|---|---|---|---|
| | | | | MA | | |
| | | | | Clinic | | |

<sup>&</sup>lt;sup>a</sup> MA = Data reported by subject on the Memory Aid and reviewed by clinic staff and reported in Solicited Events eCRF.

Note: Clinic = Data collected by clinic staff during physical exam or symptom assessment (treatment administration record, in-clinic assessment, etc.)

# **Listing 12:** 16.2.7.3: Unsolicited Adverse Events

[Implementation Note: Sort by Treatment Group, Subject ID, Associated with Dose No., and No. of Days Post Associated Dose. If the table will be multi-page, move the footnote/explanation to the footer so that it repeats for each page of the table.]

| Adverse<br>Event | Associated with Dose No. | No. of Days Post Associated Dose (Duration) | Severity | SAE? | Relationship<br>to Study<br>Treatment | In Not<br>Related,<br>Alternative<br>Etiology | Action<br>Taken with<br>Study<br>Treatment | Subject<br>Discontinued<br>Due to AE | Outcome | MedDRA<br>System<br>Organ Class | MedDRA<br>Preferred<br>Term |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Treatment ( | Group: , Subject | ID: , AE Numbe | r: | | <b>-</b> | | | | | | |
| | | | | | 1 | | | | | | |
| Comments: | I. | | | | | | | | | | |
| | <u> </u> | 1 1 | 1 | | | | | | | | |
| Treatment ( | Group: , Subject | ID: , AE Numbe | r: | | | | | | | | |
| | T | 1 | | | | | | 1 | | 1 | |
| Comments: | <u> </u> | <u> </u> | | | | | | | | 1 | |
| Note: For a | dditional details | s about SAEs, se | e Table: xx. | | | | | | | | |

# 16.2.8 Individual Laboratory Measurements

# **Listing 13:** 16.2.8.1: Clinical Laboratory Results – Chemistry

[Implementation Note: Severity should be included in parentheses after the result for abnormal results, *e.g.*, 16.2 (Mild). Sort by Treatment Group, Subject ID, and Planned Time Point.]

| Treatment<br>Group | Subject ID | Planned Time<br>Point | Actual<br>Study Day | Sex | Age (years) | Laboratory Parameter (Units) | Result (Severity<br>Grade) | Reference Range<br>Low | Reference Range<br>High |
|---|---|---|---|---|---|---|---|---|---|

# **Listing 14:** 16.2.8.2: Clinical Laboratory Results – Hematology

[Implementation Note: Sort by Treatment Group, Subject ID, and Planned Time Point.]

| Treatment<br>Group | Subject ID | Planned Time<br>Point | Actual<br>Study<br>Day | Sex | Age<br>(years) | Laboratory Parameter<br>(Units) | Result (Severity<br>Grade) | Reference Range<br>Low | Reference Range<br>High |
|---|---|---|---|---|---|---|---|---|---|

# 16.2.9 Vital Signs and Physical Exam Findings

# Listing 15: 16.2.9.1: Vital Signs

[Implementation Note: Severity should be included in parentheses after the result for abnormal results, *e.g.*, 16.2 (Mild). Sort by Treatment Group, Subject ID, and Planned Time Point.]

| Treatment<br>Group | Subject ID | Planned Time<br>Point | Actual<br>Study Day | Temperature<br>(°C) | Systolic Blood<br>Pressure<br>(mmHg) | Diastolic Blood<br>Pressure<br>(mmHg) | Heart Rate (beats/min) | Weight<br>(kg) | Height (cm) |
|---|---|---|---|---|---|---|---|---|---|

# Listing 16: 16.2.9.2: Physical Exam Findings

[Implementation Note: If the subject does not have any findings upon examination, they will not be included in this listing. If reported as an AE, display "Yes" with the AE number in parentheses, *e.g.*, "Yes (7)". Sort by Treatment Group, Subject ID, Planned Time Point.]

| Treatment<br>Group | Subject ID | Planned Time<br>Point | Actual Study<br>Day | Body System | Abnormal Finding | Reported as an AE?<br>(AE Description; Number) |
|---|---|---|---|---|---|---|

#### **16.2.10** Concomitant Medications

### **Listing 17: 16.2.10: Concomitant Medications**

[Implementation Note: If ongoing, display "Ongoing" in the "Medication End Day" column. If taken for an AE or MH, display "Yes" with the AE or MH Number in parentheses, *e.g.*, "Yes (7)". Sort by Treatment Group, Subject ID, and CM Number.]

| Treatment<br>Group | Subject ID | CM<br>Number | Medication | Medication Start<br>Day | Medication End<br>Day | Indication | Taken for an AE?<br>(AE Description;<br>Number) | Taken for a condition<br>on Medical History?<br>(MH Description;<br>Number) | ATC Level 1<br>(ATC Level 2) |
|---|---|---|---|---|---|---|---|---|---|

### 16.2.11 Pregnancy Reports

# **Listing 18:** 16.2.11.1: Pregnancy Reports – Maternal Information

[Implementation Note: Sort by Treatment Group, Subject ID, Pregnancy Number.]

| Treatment<br>Group | Subject<br>ID | Pregnancy<br>Number | Study Day<br>Corresponding<br>to Estimated<br>Date of<br>Conception | Source of<br>Maternal<br>Information | Pregnancy<br>Status | Mother's<br>Pre-<br>Pregnancy<br>BMI | Mother's<br>Weight<br>Gain<br>During<br>Pregnancy | Tobacco, Alcohol, or Drug Use During Pregnancy? | Medications<br>During<br>Pregnancy? | Maternal<br>Complications<br>During<br>Pregnancy? | Maternal<br>Complications<br>During Labor,<br>Delivery, or<br>Post-Partum? |
|---|---|---|---|---|---|---|---|---|---|---|---|

Note: Maternal Complications are included in the Adverse Event listing. Medications taken during pregnancy are included in the Concomitant Medications Listing.

# Listing 19: 16.2.11.2: Pregnancy Reports – Gravida and Para

| | | | Live Births | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject<br>ID | Pregnancy<br>Number | Gravida | Extremely<br>PB <sup>a</sup> | Very<br>Early<br>PB <sup>a</sup> | Early<br>PB <sup>a</sup> | Late<br>PB <sup>a</sup> | Early<br>TB <sup>b</sup> | Full<br>TB <sup>b</sup> | Late<br>TB <sup>b</sup> | Post<br>TB <sup>b</sup> | Still<br>Births | Spontaneous<br>Abortion/<br>Miscarriage | Elective<br>Abortions | Therapeutic<br>Abortions | Major<br>Congenital<br>Anomaly<br>with<br>Previous<br>Pregnancy? |

Note: Gravida includes the current pregnancy, para events do not.

<sup>&</sup>lt;sup>a</sup> Preterm Birth

<sup>&</sup>lt;sup>b</sup> Term Birth

# **Listing 20:** 16.2.11.3: Pregnancy Reports – Live Birth Outcomes

| Subject<br>ID | Pregnancy<br>Number | Fetus<br>Number | Pregnancy<br>Outcome<br>(for this<br>Fetus) | Fetal Distress During Labor and Delivery? | Delivery<br>Method | Gestational<br>Age at Live<br>Birth | Size for<br>Gestational<br>Age | Apgar<br>Score, 1<br>minute | Apgar<br>Score, 5<br>minutes | Cord<br>pH | Congenital<br>Anomalies? | Illnesses/<br>Hospitalizations<br>within 1 Month<br>of Birth? |
|---|---|---|---|---|---|---|---|---|---|---|---|---|

Note: Congenital Anomalies are included in the Adverse Event listing.

# **Listing 21:** 16.2.11.4: Pregnancy Reports – Still Birth Outcomes

| Subje<br>ID | Date of<br>Initial<br>Report | Fetus<br>Number | Pregnancy<br>Outcome<br>(for this<br>Fetus) | Fetal Distress During Labor and Delivery? | Delivery<br>Method | Gestational<br>Age at Still<br>Birth | Size for<br>Gestational<br>Age | Cord pH | Congenital<br>Anomalies? | Autopsy<br>Performed? | If Autopsy,<br>Etiology for Still<br>Birth Identified? |
|---|---|---|---|---|---|---|---|---|---|---|---|

# **Listing 22:** 16.2.11.5: Pregnancy Reports – Spontaneous, Elective, or Therapeutic Abortion Outcomes

| Subject<br>ID | Date of<br>Initial<br>Report | Fetus<br>Number | Pregnancy<br>Outcome<br>(for this<br>Fetus) | Gestational<br>Age at<br>Termination | Abnormality in Product of Conception? | Reason for<br>Therapeutic<br>Abortion |
|---|---|---|---|---|---|---|

# APPENDIX 4. NCA TEMPLATE

See separate document, if applicable.